#### **COVER LETTER**

Official Title of Study: Nenunkumbi/Edahiyedo ("We Are Here Now"): A Mult-level, Multi-component Sexual and Reproductive Health Intervention for American Indian Youth

NCT number: 03694418.

This manual of operations was created on February 1, 2019.

Nenunkumbi/Edahiyedo ("We Are Here Now"): A Mult-level, Multi-component Sexual and Reproductive Health Intervention for American Indian Youth was funded by the National Institute of Minority Health and Health Disparities, Grant Number R01MD01271. Our NCT number is: 03694418.

This document contains the following: 1) study summary; 2) study protocol; 3) analysis plan; 4) study intervention administration of data collection; 5) selection and enrollment of participants; 6) human subjects; 7) data safety monitoring plan; 8) revision history; and 9) appendices.

Institutional Review Board Approval was received from Montana State University on February 5, 2018 and from the Fort Peck Tribes on October 29, 2018. These IRB approvals as well as subsequent IRB modification requests due to the COVID 19 pandemic are in the appendices. Updated IRB approvals from Montana State University (11.06.20- 5-year renewal timeline) and the Fort Peck Tribes (11.02.23 - yearly renewal timeline) were included in the appendices on 9.25.24.

# Nenunkumbi/Edahiyedo ("We Are Here Now"): A Mult-level, Multicomponent Sexual and Reproductive Health Intervention for American Indian Youth

## **Principal Investigator**

Elizabeth Rink PhD, MSW
Associate Professor
Department of Health and Health Development
Montana State University
Bozeman, Montana
Email: elizabeth.rink@montana.edu

#### Supported by:

The National Institute of Minority Health and Health Disparities

National Institute of Health

Grant Number: R01 MD012701

# Study Intervention Provided by:

Nenunkumbi/Edahiyedo ("We Are Here Now") is an equitable collaborative community-academic partnership grounded in trust, respect, mutual understanding and a commitment to improving the lives of young people and their families on the Fort Peck Indian Reservation. Nenunkumbi/Edahiyedo ("We Are Here Now") is implemented by: Fort Peck Community College, the Fort Peck Tribes Language and Cultural Department, the Fort Peck Tribal Health Department, the school districts of Frazer, Wolf Point, Poplar, Brockton and Culbertson and Montana State University.

# TABLE OF CONTENTS

| SECTION 1: STUDY SUMMARY | Page 2 |
|-----------------------------------------------------------------|---------|
| SECTION 2: STUDY PROTOCOL | Page 2 |
| SECTION 3: ANALYSIS PLAN | Page 8 |
| SECTION 4: STUDY INTERVENTION ADMINISTRATION OF DATA COLLECTION | Page 10 |
| SECTION 5: SELECTION AND ENROLLMENT OF PARTICIPANTS | Page 13 |
| SECTION 6: HUMAN SUBJECTS | Page 14 |
| SECTION 7: DATA SAFETY MONITORING PLAN | Page 20 |
| SECTION 8: TOOL REVISION HISTORY | Page 25 |
| SECTION 9: APPENDICES | Page 26 |

#### **SECTION 1: STUDY SUMMARY**

American Indian (AI) communities in the United States (US) are disproportionately affected by sexual and reproductive health disparities, compared to other populations, placing current and future generations of AI societies in jeopardy. Our study, "Nen OnkUmbi/EdaHiYedo (NIE - "We are Here Now")", utilizes a culturally tailored ecological intervention in which the prevention of sexual-risk behaviors among AI youth that lead to STIs, HIV, HCV, and teen pregnancy are addressed. N/E takes place on the Fort Peck Reservation in northeastern Montana. N/E is a community-based participatory research sexual and reproductive health (SRH) intervention, constructed on Ecological Systems Theory. Based on Fort Peck tribal members' desire to implement a holistic SRH intervention for the tribes' youth, N/E includes: 1) A school-based SRH curriculum called Native Stand, designed to address individual-level factors that lead to risky behaviors; 2) a family-level curriculum called Native Voices, tailored to increase communication between adult family members and youth about SRH topics; 3) a cultural mentoring component at the community-level that pairs AI youth with adults and elders to discuss traditional AI beliefs and practices about SRH; and 4) a systems-level strategy to activate a multi-sectoral network of local youth servicing organizations to coordinate SRH services. The overarching aim of this proposal is to refine and tailor the components of N/E and evaluate its efficacy. N/E is a 5-year study involving 456 15- to 18-year-old AI youth and their parent/legal guardian.

#### **SECTION 2: STUDY PROTOCOL**

- **2.1 Study Team Roster.** *NIE's* tribal community and academic study team combines Indigenous expertise in traditional knowledge, contemporary reservation culture, and local tribal resources and skills with Westernized research experience in SRH interventions among Indigenous populations and qualitative and quantitative research methodologies. The study team members are listed below.
  - *Elizabeth Rink*, Ph.D., MSW, at Montana State University (MSU) is the principal investigator (PI) for *NIE*. Dr. Rink will be responsible for the overall research and fiscal administration, implementation, and evaluation of *NIE*.

Email: elizabeth.rink@montana.edu

• **Paula FireMoon** (Sioux), M.A., is *NIE's* Fort Peck-based Project Director. Ms. FireMoon will oversee community participation, including implementation of *NIE*, and coordination of *NIE's* research activities with tribal schools, health care facilities, and other youth-servicing agencies on the Fort Peck Reservation.

Email: PFiremoon@fpcc.edu.

• **Ramey Growing Thunder** (Sioux/Navajo), M.Ed., is director of the Fort Peck Tribes' Language and Culture Department. Mrs. Growing Thunder will lead the implementation of *NIE's* cultural mentoring program.

Email: <a href="mailto:rgrowingthunder@gmail.com">rgrowingthunder@gmail.com</a>.

• Adriann Ricker (Assiniboine), MPH, CHES, is associate director of the Fort Peck Tribes' Health Promotion and Disease Prevention Program. Ms. Ricker will increase coordination among, and access to, SRH services for Al youth in schools, health care facilities, and youth-servicing agencies at Fort Peck.

Email: adricker@gmail.com.

- Community Advisory Board (CAB) that includes five tribal members. CAB members are: Ingrid FireMoon Email: IFiremoon@fortpecktribes.net, Bruce Bauer- Email: bwbauer@yahoo.com, Olivia Johnson Email: ojohnson@brockton.k12.mt.us; Martel Reum Email: MReum@fpcc.edu; and Alexandria Herrald Email: alexandria.herrald26@gmail.com.
- **Julie Baldwin** (Cherokee), Ph.D., director of The Center for Health Equity Research at Northern Arizona University, with over 20 years of research expertise in the design, implementation, and

evaluation of HIV and substance abuse prevention interventions for AI youth is the study's Co-Investigator and senior research mentor to Dr. Rink.

Email: Julie.Baldwin@nau.edu.

• *Mike Anastario*, Ph.D., is Co-Investigator and statistician for the study.

Email: manastar@fiu.edu.

• **Rachel Hallum-Montes,** Ph.D., an independent contractor who has worked on a variety of national teen pregnancy-prevention studies with the CDC will consult on the assessment of the coordination and implementation of SRH services for Al youth.

Email: rhallum.montes@gmail.com.

• Genevieve Cox, Ph.D., NIE's MSU-based research program manager.

Email: <a href="mailto:genevieve.cox@montana.edu">genevieve.cox@montana.edu</a>.

**2.2 Study Sites.** NIE is implemented on the Fort Peck Reservation in Northeastern Montana. Fort Peck is located in a Northern Plains frontier environment and spans 2.1 million acres. It borders the  $47\frac{1}{2}$  parallel to the north Uust south of the border with Canada), with Big Muddy Creek to the east, the Missouri River to the south, and Big Porcupine Creek to the west. Approximately 8,000 enrolled tribal members, predominately from the Assiniboine and Sioux Nations, live on the reservation. The Assiniboine and Sioux are descendants of the Nakada, Nakata, Nakona, Lakota, and Dakota Nations. The Assiniboine comprise Wadopana (Canoe Paddlers Who Live on the Prairie) and Hudashana (Red Bottom) bands, and the Sioux comprise Sisseton/Wahpetons, the Yanktonais, and the Teton Hunkpapa bands. NIE will be implemented in the communities of Frazer, Wolf Point, Poplar, Brockton, and Culbertson. These 5 communities have public high schools that serve Al students. Frazer, Wolf Point, Poplar, and Brockton are on the reservation, and Culbertson is a border town on the east end of the reservation that Al youth from the reservation community of Fort Kipp attend (See Figure 1 for map of reservation and high schools).

Collaborating entities in *NIE* are:

- Montana State University, 318 Herrick Hall, Bozeman, MT. 59715, phone: 406.994.3833, Fax: 406.994.2013
- Fort Peck Community College. PO Box 398
  Poplar, MT. 59255, phone: (406) 768-6300, Fax: 768.6301
- The Fort Peck Tribes Language and Cultural Department, 603 Court Avenue, PO Box 1027, Poplar, MT. 59255, phone: 406.768.3520, Fax: 406.768.3531.

Frazer (45)
Wolf Point (228)
Wolf Point (228)
Wolf Point (219)
Brockton (47)
Culbertson (78)

Figure 1. Study sites on or near the Fort Peck Reservation.

High school enrollment shown in parentheses.

- <u>The Fort Peck Tribal Health Department.</u> 107 H Street East, PO Box 1027, Poplar, MT. 59255, Phone: 406, 653,1191, Fax: 406, 768,5780.
- Frazer Public School, 325 6th Street, Frazer, MT, 59225, Phone: 406.695,2241, Fax: 406.695,2243.
- Wolf Point School District, 213 6<sup>th</sup> Ave. South, Wolf Point, MT. 59201, Phone: 406.653.2361, Fax: 406. 653.3405.
- <u>Poplar School District</u>, 400 4<sup>th</sup> Avenue West, Poplar, MT. 59255, Phone: 406.768.6600, Fax: 406.768.6800.
- Brockton School District, 215 North 5<sup>th</sup> Street, Brockton, MT. 59213, Phone: 406.768.3311, Fax: 406. 786.3377.
- <u>Culbertson School.</u> 423 1st Avenue West, P.O. Box 459, Culbertson, MT. 59218, Phone:

406.787.6241, Fax: 406.787.62

#### 2.3 RESEARCH DESIGN OVERVIEW

**2.3.1 Study Title.** Nenunkumbi/Edahiyedo ("We Are Here Now"): A Mult-level, Multi-component Sexual and Reproductive Health Intervention for American Indian Youth

# 2.3.2 Study\_ Aims.

- <u>AIM 1</u> begins with a year of formative work to refine and tailor the components of N/E. Our community advisory board and the Fort Peck-based and MSU-based research team will design culturally appropriate adaptations for N/E's 4 levels.
- <u>AIM 2</u> tests the efficacy of N/E using a cluster-randomized stepped-wedge design (SWD), in which the 5 high schools that Fort Peck youth attend are randomized into the intervention 1 at a time. N/E's primary outcome is increased condom use during sexual intercourse. Secondary outcomes are delayed onset of sexual intercourse, number of sex partners, frequency of sexual intercourse, pregnancy history, consistent use of birth control during sexual intercourse, and whether alcohol and/or other drugs are used during sexual intercourse. Tertiary outcomes are increased parent/legal guardian-child communication about SRH topics, increased understanding of cultural values related to traditional Al beliefs regarding SRH, and increased use of SRH services. Quantitative data collection includes: student surveys at baseline, 3, 9 and 12 months; parent/legal guardian surveys at baseline, 9 and 12 months. Qualitative data collection includes SRH service provider discussion groups at baseline and thereafter once a year over the 5-year study, with logs to track coordination and implementation at baseline and 3, 6, 9 and 12 months.
- <u>AIM 3</u> will evaluate the fidelity and acceptability of N/E with focus groups, activity logs, and staff meeting notes and staff field notes.

Our **long-term goal** is to produce a toolkit, including curriculum manuals, an SRH cultural mentoring program, and specific systems-level actions suitable for replication in other tribal communities. The **public health impact** is the prevention of STIs, HIV, HCV, and teen pregnancies in Al youth resulting in reduced sexual and reproductive health disparities and improved health in Al families and communities.

**2.3.3 Design Overview.** NIE is a community-based participatory research (CBPR) multi-level, multi-component sexual and reproductive health (SRH) intervention, constructed on Ecological Systems Theory. NIE is based on Fort Peck tribal members' desire to implement a holistic SRH intervention for Al youth. NIE includes: 1) A school-based SRH curriculum called  $Native\ Stand$ , designed to address **individual-level** factors that lead to sexual risk behaviors; 2) a **family-level** curriculum called  $Native\ Voices$ , tailored to increase communication between adult family members and youth about SRH topics; 3) a cultural mentoring component at the **community level** that pairs Al youth with adults and elders to discuss traditional Al beliefs and practices about SRH; and 4) a mobilizing strategy to activate a multi-sectoral network of youth-servicing organizations at the **systems level** in Fort Peck to coordinate SRH services for Al youth. The overarching aim of this study is to refine, tailor, and finalize the components of NIE and evaluate its efficacy. We will use a cluster-randomized stepped-wedge design (SWD), in which 5 schools that Al youth from Fort Peck attend are the clusters to be randomized into the intervention 1 at a time, with all schools eventually being randomized to the intervention. The 5 schools are located in separate communities, mitigating the potential for cross-contamination. NIE is a 5-year study involving 456 15- to 18-year-old Al youth.

**2.3.4 Intervention Design.** NIE is a 5-year CBPR ecological intervention for 456 15- to 18-year-old Al youth living on the Fort Peck Reservation. Nen OnkUmbilEdaHiYedo ("We Are Here Now") derives from the Assiniboine (Nen OnkUmbt) and Sioux (EdaHiYedo) names for their traditional coming-of-age ceremonies, when, at the age of 15 and over, young tribal members are believed to be ready for integrated education and training on sex, what it means to be a man or a woman, relationships, having children, and being a parent. NIE is guided by a 5-member CAB. The primary institutional partners responsible for the implementation of NIE are Fort Peck Community College (FPCC), the Fort Peck Tribes Language and Culture Program, the Fort Peck Tribal Health Department (Epi Team)¹, and MSU.

NIE will be implemented simultaneously over the 9-month school year (Table 1). Components include: 1) Individual Level. Native Stand is a school-based, 27-module STI-, HIV-, and teen pregnancy-prevention curriculum, originally developed for rural white youth and adapted in 2008 as a stand-alone SRH curriculum for Al youth. For NIE, an adaptation of Native Stand will be implemented in the study's 5 high schools to educate Al youth on sexual risk behavior prevention strategies. The tailoring of *Native Stand* will reduce its 27 modules to 18 modules and will include specific community-relevant traditional and contemporary cultural lesson plans. Native Stand will be integrated into each of the 5 schools' established curriculum and will be delivered by the NIE School Coordinator in a classroom setting as part of the students' regular class schedule. 2) Family Level. Native Voices is a video-based HIV/STI-prevention intervention designed for AI youth to address condom use, negotiation skills, group discussion, and role playing. Native Voices will be adapted from 1 module into 4 modules to involve parents/legal guardians, as recommended by the CDC. Our adaptation of Native Voices involves students with one of their parents/legal guardians to promote parent/legal guardian/youth discussions about preventing STIs, HIV, HCV, and teen pregnancy. The NIE School Coordinator will present Native Voices to groups of students and their parents/legal guardians at the study's high schools for 2 hours in the evening. 3) Community Level. The third level of NIE is a cultural mentoring component that pairs Al youth with older adults and elders to discuss traditional Al beliefs and practices about reproductive health. The mentoring program is based on Assiniboine and Sioux traditional knowledge and the National Mentoring Partnership standards for mentoring. The mentoring program was designed specifically for Fort Peck youth by the Fort Peck Tribes' Language and Culture Department and has been in existence for 5 years. NIE integrates this cultural mentoring program into NIE's overall framework with an emphasis on addressing traditional topics related to SRH, such as overall information on cultural beliefs, values, and ceremonies, and more specific information on cultural beliefs and values regarding sex, having children, parenting, and relationships. Our cultural mentoring program will include older male and female tribal members who will be paired with the youth by gender and tribal affiliation. Al youth will meet one-on-one with their mentors each month and also monthly in mentor-mentee small groups. Depending on the purpose of the cultural mentoring sessions, the sessions will take place at either the study's high schools, the Fort Peck Language and Culture Department's main office in Poplar, community centers on the reservation, or at the Buffalo Ranch. Ramey Growing Thunder will oversee the implementation of the cultural mentoring program. 4) **Systems Level.** The fourth level of NIE mobilizes the existing Epi Team to enhance the coordination and implementation of SRH services at Fort Peck. The members of the Epi Team will utilize the recommendations in the CDC's Contraceptive and Reproductive Health Services for Teens: Evidence-based Clinical Best Practices Guide to enhance the coordination and implementation of SRH services for Al youth. This enhancement process will take place during the Epi Team's monthly meetings at the Fort Peck Tribal Headquarters in Poplar by developing a coordination and monitoring plan that can be tracked over time to address the barriers, facilitators, and solutions to increase access to SRH

-

<sup>&</sup>lt;sup>1</sup> Fort Peck Tribal Epidemiology Team (Epi Team), which is a local committee that has been in existence for 15 years to monitor diseases on the reservation and the health status of tribal members. The Epi Team is comprised of the Fort Peck Tribal Health Department; the Indian Health Service (Poplar Service Unit and Wolf Point Service Unit); the Roosevelt County Health Department; school nurses from the Fort Peck Health Promotion and Disease Prevention Program; the high schools of Frazer, Wolf Point, Poplar, Brockton, and Culbertson; and the Fort Peck Tribal Executive Board.

services for Al youth at Fort Peck. Dr. Rink, Ms. FireMoon, Ms. Ricker and Dr. Cox will attend the Epi Team's monthly meetings to work in partnership to implement *NIE's* systems-level component.

Table 1. Overview of N/E's 9-month multi-level, multi-component intervention plan.

| INDIVIDUAL | FAMILY | COMMUNITY | SYSTEMS |
|---|---|---|---|
| Native Stand (NS): 18-session school-based curriculum delivered twice a month over 9 months in N/E's 5 participating schools. NS will be integrated into the schools' existing class schedules. | Native Voices (NV): 4 sessions delivered once every other month to students and parents/legal guardians after school hours at N/E's 5 participating schools. | Cultural Mentoring Program (CMP):<br>9 mentoring sessions delivered twice<br>a month over 9 months that include<br>one group activity with CMP mentors<br>and mentees and one 1:1 meeting.<br>CMP activities will take place at<br>varying locations on the Reservation<br>depending on the activity. | SRH Services: Monthly meetings<br>over 12 months with Epi Team at the<br>Fort Peck Tribes Headquarters offices<br>in Poplar, Montana. |
| NS 1: Introduction to an overview of<br>N/E and Native Stand<br>NS 2: Culture & Tradition – Part 1 | NV 1: Introduction to an overview of<br>N/E and Native Voices | CMP 1: Assiniboine/Sioux kinship<br>networks and concepts of family and<br>genealogy | Epi Team meetings will take place<br>monthly over 9 months to enhance<br>coordination and implementation of |
| NS 3: Culture & Tradition – Part 2 | | CMP 2: Traditional male/female roles and cultural beliefs about healthy | SRH services for AI youth. |
| NS 4: Healthy Relationships – Part 1 | | relationships | |
| NS 5: Healthy Relationships - Part 2 | NV 2: Talking with youth about topics related to sex | CMP 3: Cultural beliefs about sex and how to make decisions about sex that | |
| NS 6: Reproductive Health - Part 1 | | integrate cultural values | |
| NS 7: Reproductive Health - Part 2 | | CMP 4: Cultural beliefs about parent-<br>ing and the role of family | |
| NS 8: Pregnancy & Parenting | | | |
| NS 9: Preventing Pregnancy | NV 3: Prevention of STIs, HIV/AIDS, and HCV | CMP 5: The role of ceremony in tradi-<br>tional Assiniboine/Sioux culture | |
| NS 10: Condoms & Birth Control | | | |
| NS 11: Sexually Transmitted Diseases | | CMP 6: The role of sweat lodges in Al spirituality | 1 |
| NS 12: HIV/AIDS & HCV | | | |
| NS 13: Drugs, Alcohol, & Sex | NV 4: Strategies for fostering healthy relationships in your child's intimate | CMP 7: Honoring ceremonies in the lives of young men and women | |
| NS 14: Mental Health & Sex | relationships | | |
| NS 15: Negotiation & Refusal Skills | | CMP 8: Understanding the sacredness of the land | |
| NS 16: Decision-Making | | P471 (0.000) (0.000) | |
| NS 17: Effective Communication | | CMP 9: Buffalo Harvest | |
| NS 18: Putting It All Together | | | |

Trial Design. **2.3.5** Our selection of an SWD to evaluate *NIE* is consistent with tribal members' desires that all 15- to 18-year-old Al vouth receive the intervention. The SWD is a cluster-randomized trial. which involves random and sequential crossover of clusters from control to intervention until all clusters are exposed to the intervention. <sup>5 29</sup>. The first observation period corresponds to a baseline measurement observation, in which none of the clusters have been randomized to NIE. Clusters are randomized to *NIE* at subsequent steps until all clusters have

completed treatment. *Following randomization of the schools to the intervention, there will be three waves of implementation: Wave 1 (1school in 2019), Wave 2 (2schools in 2019-2020), and Wave 3 (2 schools in 2020-2021).* The 5 schools on the Fort Peck Reservation will be the clusters that are randomized to *NIE. NIE* will take approximately 40 weeks, or 3 quarters, to implement. The first observation period (Q4 of Year 2) provides baseline measurements for all respondents drawn from every cluster. The cluster is then surveyed at 3, 9, and 12 months for the students in the cluster once they have begun participation in the intervention, and at 9 and 12 months for the parents/legal guardians in the cluster once they have begun participation in the intervention. Following completion of the intervention across all clusters, we will conduct the quantitative analysis. The SWD allows us to control for the effect of time and ensure that the full Al population of schools at Fort Peck receives *NIE*. The systems-level component of *NIE* will be implemented reservation-wide rather than school-wide during Years 2 to 4 of NIE as the SWD is rolled out. The systems level component will be measured and analyzed qualitatively.

**2.3.6 Trial Timeline.** The timeline for NIE is: <u>Year 1-Refine</u>, tailor, and finalize the components of NIE with the CAB by reviewing our current quantitative and qualitative data from Fort Peck and by talking with elders

Figure 4. Trial design and timeline for implementing N/E relative to grant and sites/schools.

| Y | EAR 1 | (201 | 18) | YE | AR 2 | 2 (201 | 19) | YEAR 3 (2020) | | | 2020) YEAR 4 (2021) | | | | | YEAR 5 (2022) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Q1 | Q2 | Q3 | Q4 | Q1 | Q2 | Q3 | Q4 | Q1 Q2 Q3 Q4 Q1 Q2 Q3 Q4 Q1 Q2 Q3 Q4 | | | | | Q3 Q4 Q1 Q2 Q3 Q4 | | | | Q4 | | | |
| of ME | Site 1 | | | 3mf 9mf 12mf | | | | | | | | | | | | ning | | lion | | Cluster unexposed to N/E |
| components | Site | | bsln | | | | 3mf | N/E | 9mf | 12mf | | | | | bility Plar | | and Dissemination | | Intervention cluster | |
| tailor comp | Site 3 bsln | | | | 3mf N/E 9mf | | | | | 12mf | | | | | stainabi | | and Dis | | Post-intervention cluster | |
| aug | Site | e 4<br>bsln | | | | 3mf | | | | | 3mf 9mf 12mf | | | | | sis / Su | | ▼<br>Publication | bsl | n = baseline data collection; |
| Refine | Site | | bsln | | | | | | | 3mf | N/E | 9mf | 12m | f | | Analysis | | Pub | mf | = 3, 9, or 12 months |

and community stakeholders. We will have monthly team meetings and quarterly CAB meetings. When necessary, we will meet with CAB members individually. We will also recruit, hire, and train staff in *Native Stand* and *Native Voices*; identify the cultural mentors; purchase all necessary materials and supplies; finalize research protocols and IRB approvals. <u>Years 2, 3, and 4-</u> Collect baseline data; Implement *NIE*; conduct quantitative and qualitative data collection; conduct ongoing fidelity and acceptability data collection; and continue monthly team meetings and quarterly CAB meetings. <u>Year 5-Finish</u> data collection; conduct data analysis; work with CAB on interpretation of data analysis; develop sustainability plan; develop intervention toolkit; and disseminate results to scientific, professional, and Fort Peck communities. See Appendices for *NIE* timeline.

**2.3.7** Sample Size and Population. NIE's sample size is 456 Al male and female youth ages 15 to 18 years old. The population of Al youth 15 to 18-year-old attending the five schools participating in the study is approximately 617.

2.3.8 Study Background and Rationale. Comprehensive national surveillance data on SRH among Als is difficult to assess due to the underrepresentation of Als in national surveys. The data on Al SRH in the United States that are available demonstrate that Als are disproportionately affected by adverse conditions attributable to SRH, compared to other populations. Al youth report earlier onset of sexual intercourse than other adolescent populations in the U.S. The teen birth rate among Als is 2 to 3 times higher than that among Caucasians. In addition, the rates of pre-term birth and low birth weight are much higher in Als compared to Caucasians. STIs are up to 4.6 times higher for AI males and females compared to Caucasians, with young AI males having the highest chlamydia rates of any racial- and age-specific population in the U.S. As a result, Al females have higher rates of miscarriages and ectopic pregnancies than Caucasian females and are at risk for infertility. For Al males, STIs can lead to urethritis, epididymitis, and prostate cancer, which is higher in Al men than all other racial and ethnic males in the U.S. In addition, the costly and burdensome health consequences of Al youths' high STI rates include infection with HIV and HCV. The incidence of HIV in Al males and females is 30% higher than in Caucasian males and females, and in recent years Als are the only racial and ethnic group in which the incidence of HIV continues to rise. Furthermore, of all population subgroups in the U.S., the incidence of HCV is highest in Als. At present no extant multi-level, multi-component intervention has been shown to be efficacious in addressing SRH among Al youth. The majority of Al interventions appearing in the peer-reviewed literature instead focus on alcohol and substance use reduction. Thus, a critical need exists to address the SRH disparities among Al youth, which place current and future generations of Al societies in jeopardy.

The literature related to SRH among Al youth identifies poverty, isolation, alcohol and other drug use, physical and sexual victimization, and lack of comprehensive and coordinated SRH education and clinical services as factors that influence unintended pregnancies and STIs. Evidence also suggests that ambivalence toward sex, social pressures, depression, anxiety, and experiences of historical trauma and loss influences sexual risk behavior among Als. Mistrust of research and researchers continues in Al communities due to a legacy of neglect and betrayal by the U.S. government and by researchers from outside their communities. This mistrust impedes the cooperation between tribal communities and academics to design, implement, and evaluate effective interventions to address SRH disparities among Al youth.

The complex factors that influence sexual risk behaviors among Al youth warrant novel Al community-specific interventions. Previous research with Al youth on SRH has lacked an ecological design and implementation, and it has neither addressed nor leveraged the interconnectedness of the individual, family, community, and larger systems in preventing STIs, HIV, HCV, and teen pregnancy. Furthermore, CBPR, which has become an established methodological framework for partnering with Al communities to conduct research, has been sparsely applied to understanding and addressing Indigenous SRH. CBPR has the potential to facilitate the

implementation and evaluation of an ecological intervention in Al communities, particularly given its amenability to multi-sectoral and multi-level stakeholder involvement in the research process.

#### **SECTION 3: ANALYSIS PLAN**

<u>3.1.1</u> <u>Power analysis.</u> Sample size requirements were calculated taking into account a unique design effect for the SWD,<sup>2</sup> such that  $Nsw = Nu \times DEsw$  (where Nu is the total number of students needed to detect the treatment effect with a power of 80% and a significance level of 0.05, uncorrected for cluster and repeated measurements). The design effect was calculated as:

$$DE_{sw} = \frac{1 + \rho(ktn + bn - 1)}{1 + \rho(\frac{1}{2}ktn + bn - 1)} \times \frac{3(1 - \rho)}{2t(k - \frac{1}{k})}$$

where k is the number of steps, n is the expected number of students per cluster, b is the number of baseline measurements, t is the number of measurements after each step, and p is the intra-class correlation coefficient, estimated to be 0.016 based on findings reported by Kaufman et al.<sup>3</sup> With an  $\rho$  of 0.05, power of 0.8, Nu = 292, DEsw = 1.3273, and the expectation of 15% attrition during the study, a sample size of 456 will allow the detection of a 0.14 increase in the proportion of condom use relative to the frequency of sexual intercourse from baseline to the 12-month observation period hypothesized under Aim 2.

**3.1.2 Missing data.** Attrition is likely to covary with truancy, suggesting a missing data mechanism that is not missing at random (NMAR). To address this, a dropout variable Di will be developed for each individual across the 4 observation periods, where Di=k for dropout between the (k-1/hand k<sup>th</sup> occasion. A model of th probability of dropout, where

log  $\left\{\frac{(\Pr(D_i=k)}{(\Pr(D_i>k)} \middle| \frac{D_i\geq k, Y_{i_1},...,Y_{i_k}}{D_i>k, Y_{i_1},...,Y_{i_k}}\right\} = \theta_1 + \theta_2 Y_{i_{k-1}} + \theta_3 Y_{i_k}$  presumes that  $\theta_3 \neq 0$  for the NMAR mechanism. Missing data will be examined using multiple imputation, where missing values are replaced by a set of m plausible values using a propensity scoring sequence to generate a single estimate of the parameters of interest. Observations will first be grouped on the basis of propensity score similarity, then individuals with missing values will be randomly matched to those with observed values, and finally missing values will be randomly selected with replacement from the random sample of observed values. This sequence will be repeated sequentially starting at the 3-month follow-up observation through the 12-month follow-up observation, and the entire propensity scoring and time imputation sequence(s) will be repeated at minimum across 2::5 datasets (m) to estimate  $\bar{\beta} = \frac{1}{m} \sum_{k=1}^{m} \hat{\beta}^{(k)}$ . Sensitivity analyses will also be used to assess the robustness of primary results attributable to missing data by examining imputed and nonimputed data.

**3.1.3 Dose.** The treatment dose is the number of intervention components delivered to the individual student, accounting for individual students' attendance and participation. This will be tracked using the fidelity log, staff field notes, and the CAB meeting. A count, nominal, or weighted percentage will be used to represent dose pending analysis of the dose frequency distribution.

<u>3.1.4</u> <u>Baseline data analysis.</u> Baseline data will first be analyzed to determine whether demographic and SRH variables vary relative to school (cluster). The psychometric properties of scales will be explored, and confirmatory factor analyses (CFA) for scales will be conducted. Finally, structural equation models (SEM) will

be developed based on the multi-level components derived from the Ecological Systems Theory model

10

<sup>&</sup>lt;sup>2</sup>Woertman W et al. Stepped wedge designs could reduce the required sample size in cluster randomized trials. J Clin Epidemiol. July 2013;66(7):752-758.

<sup>3</sup> Kaufman C et al. Effectiveness of Circle of Life, an HIV-preventive interventive intervention for American Indian middle school youths. Am J Public Health. June 2014; 104(6):e106-e112.

<sup>&</sup>lt;sup>4</sup> Fitzmaurice G, Laird N, Ware J. Generalized Linear mixed effects Models in Applied Longitudinal Analysis. Hoboken, NJ: John Wiley & Sons Inc.; 2004.

upon with the N/E was built. CFAs and SEMs will be conducted using Mplus software.

**3.1.5 Randomization of schools.** The 5 schools that Al youth from Fort Peck attend are the clusters to be randomized into the intervention, with all schools eventually being randomized to the intervention. Students and their parents/legal guardians will be recruited for baseline participation prior to randomization of the sites. Schools will be randomized to the intervention following baseline data collection using a single sequence random assignment to clusters that will determine order of intervention receipt.<sup>5</sup>

3.1.5 Generalized linear mixed-effects models. To test for effectiveness of the NIE intervention across all hypotheses under Aim 2, the generalized linear mixed-effects models (GLMM) will be used to model binary primary and secondary outcomes (condom use under H1, condom use and other sexual risks under H2) and continuous tertiary outcomes (H3) in the data. The GLMM allows for individual-level binary and continuous responses to be modeled, key covariates to be controlled for, the specification of autocorrelation within individuals, and clustering by school. The GLMM is also the most frequently employed analytic method to adjust for the longitudinal nature of SWDs,<sup>6</sup> and it was chosen over the Generalized Estimating Equations (GEEs) because GEEs show inflated Type 1 error rates when the number of clusters is small, as is the case with the number of schools at Fort Peck. Hussey and Hughes proposed a mixed-effects regression approach for the SWD-CRT design,<sup>7</sup> where:

 $Y_{ijl} = \mu + \beta_j + \theta X_{ij} + u_i + e_{ijl}$ , and where  $u_i \sim N(0, \sigma_u^2)$ ;  $e_{ijl} \sim N(0, \sigma_e^2)$ , with  $\beta_j$ =the fixed effect of time,  $X_{ij}$ =intervention (0,1 or dose representation),  $\theta$  =intervention effect,  $u_i$ =random effect for cluster, and  $e_{ijl}$ =residual for i clusters, j time periods, and l adolescents.  $Y_{ijl}$  will be modeled for SRH outcomes and interpreted in terms of a contrast of the log odds of response relative to Al youths with similar values for unobserved random effects. In order to test for changes in the tertiary outcomes, we will specify  $Y_{ijl}$  as continuous response outcomes. STATA statistical software will be used to conduct GLMMs. However, SAS will be used if more complex specification of the intraclass correlation becomes necessary.

<u>3.1.6</u> 7 Analysis of focus group data. Focus group data will be transcribed and coded using a partially inductive procedure. First, all transcript data will be open coded (line-by-line coding). The open codes will be pre-sorted based on whether participants are responding to acceptability or fidelity prompts. Within each implementation domain, axial codes will be developed to group the open codes, and the team will meet to discuss how axial codes saturate the pre-defined acceptability and fidelity categories. Transcripts will be coded using Atlas.ti software.

<u>3.2 Qualitative Data Analysis.</u> The systems level component and the FAS evaluation component of N/E will be analyzed using content analysis. Common themes will be identified from the two respective sets of data collection instruments. Coding will proceed in stages. A topical indexing scheme will be developed with input from the community advisory board members to identify the text pertaining to particular topics relevant to the systems level and FAS components of N/E. The software program, Atlis.ti will be used to construct and organize a topical indexing system of codes identifying sections of text that capture the central concepts of interests. Then, content coding will be developed by the research team with advice from the community

<sup>&</sup>lt;sup>5</sup> Esserman D, Allore HG, Travison TG. The Method of Randomization for Cluster-Randomized Trials: Challenges of Including Patients with Multiple Chronic Conditions. International journal of statistics in medical research. 2016;5(1):2-7. doi:10.6000/1929-6029.2016.05.01.1.

<sup>6</sup> Barker D, McElduff P, D'Este C, Campbell MJ. Stepped wedge cluster randomized trials: A review of the statistical methodology used and available. *BMC Med Res Methodol.* 2016;16:69.

<sup>&</sup>lt;sup>7</sup> Hussey M, Hughes J. Design and analysis of stepped wedge cluster randomized trials. Contemp Clin Trials. February 2007;28(2):182-191

advisory board to capture the content, themes, or sentiment of responses within topics. The community advisory board members will receive copies of the content coding and the content, themes, and sentiment of responses for each of the themes identified in the qualitative data collection forms. Members of the research team, including the community advisory board, will individually identify themes from all text pertaining to a specific topic are related to N/E's AIMS 2 and 3 in order to then assist the research team in developing codes to be analyzed using Atlis.ti. The codes will be reviewed and approved of by the community advisory board prior to analysis. The coding reliability for the content coding will be determined through check coding of at least 20% of the randomly chosen text within major topical categories. Once the data are coded, the themes and patterns will be summarized and interpreted. Coded text will be used to identify illustrative quotes from the qualitative data collection materials.

#### SECTION 4: STUDY INTERVENTION ADMINISTRATION OF DATA COLLECTION

 $N\!I\!E$  is a mixed methods study involving quantitative and qualitative methodology. There are four data collection components to  $N\!I\!E$ : 1) student survey (quantitative); 2) parent survey (quantitative); 3) systems level tracking (qualitative); and 4) fidelity, acceptability and sustainability evaluation (qualitative). The student survey, parent survey and systems level tracking data collection are described in section 4.1. The fidelity, acceptability and sustainability evaluation data collection is described in section 4.2.

**4.1. NIE** Intervention Components: The intervention components and corresponding modes of data collection to test efficacy of the four aspects of our intervention are shown in the table below. The left column indicates the intervention component, while the right column indicates the type of data collection and the timeline of data collection.

| Intervention Component | Types of Data Collection and Timeline |
|---|---|
| Individual level: Native Stand Family level: Native Voices | Student Surveys: baseline, 3 months, 9 months, 12 months |
| Community level: Cultural Mentoring | Parent Surveys: baseline, 9 months, 12 months |
| Systems level: Enhancement of the coordination and implementation of SRH services at Fort with the Fort Peck Epi Team | Barriers and Facilitators Discussion<br>Group: yearly |
| ' | Coordination & Implementing Monitoring<br>Plan Tracking Loq: quarterly |

Subsequent to randomization of the 5 area schools to the intervention, there will be a baseline data collection from the middle of March to June 2019, followed by three waves of implementation and concurrent data collection over the next 3 years. For a visual picture of how these intervention components and methods of data collection fit into an overall Timeline, please see our Trial Timeline in the appendix.

For the student and parent/legal guardian participating in NIE, there are 2 forms of data collection: a student survey and a parent/legal guardian survey. Ms. FireMoon, a part-time assistant, and the N/E school outreach coordinator will oversee both surveys' administration. The student surveys and parent/legal guardian surveys will be completed using Research Electronic Data Capture or "REDCap." REDCap is a secure web application for building and managing surveys and databases.

The students and parents will take the survey on iPads that have the mobile application version of REDCap installed on the tablets. The mobile app version of REDCap collects data offline to be uploaded to an online, secure database once a secure wifi location is reached. Deidentified data will be stored virtually on the REDCap server and available for download to Genevieve Cox, Paula Firemoon, Michael Anastario, Rachel Hallum-Montes and Beth Rink. Only Paula Firemoon, the NIE outreach coordinator, and Genevieve Cox will have access to names linking students and parents to their records during data collection and intervention implementation. These files will be kept in a locked file cabinet by Genevieve Cox at MSU after data collection.

From Years 2-4, 456 students and one of their parents/legal guardians will participate in NIE's data collection. Student surveys for baseline, 3, and 9 months will be administered during regularly scheduled classes in an assigned classroom by Ms. FireMoon, the assistant, and N/E's outreach coordinator. Baseline data collection will begin in March 2019 for all schools and parents included in the intervention. Groups of 20 students at a time will be appropriately spaced in the classroom in order to ensure privacy, and survey instructions will be presented to students prior to REDCap administration. Ms. FireMoon, the assistant, and the NIE outreach coordinator will thoroughly review the assent form with the students, which will include a description of NIE, types of questions that will be asked, and potential risks and benefits of participating in NIE. All students will be reminded that they can withdraw at any time without consequences. Prior similar procedures have been successfully used by Dr. Rink and Ms. FireMoon for data collection in the Fort Peck schools with Al youth. For students who graduate from high school prior to the 12-month follow-up, they and their parent/legal guardian will be contacted by Ms. FireMoon to complete the 12-month follow-up (during evening hours) at the high school from which they graduated following the same procedure described above. Although data collection for the students has been designed to coincide with the school year, the same procedures will be followed if the data collection occurs when school is not in session.

Wave 1 data collection will commence in December 2019 with 1 school after students have begun receiving the Native Stand and Cultural Mentoring components of the intervention during the school year.

Wave 1 9- month follow-up will take place at the end of the school year in May/June 2020 as the intervention is completed. The Wave 1 12-month follow-up will take place at the beginning of the next school year in September 2020.

Wave 2 (2 schools) and Wave 3 (schools) will follow the same procedures and pattern of timeline of data collection. The parent survey will be administered during evening hours at the high school by Ms. FireMoon, the assistant, and N/E's outreach coordinator. All baseline parent data will be collected in Fall 2019. We will use the same REDCap administration procedures for parents/legal guardians that are described for students above. Ms. FireMoon, the assistant, and the N/E outreach coordinator will review the consent forms with the parents/legal guardians to ensure their understanding of the purpose of N/E, types of questions they will be asked, and the study's potential risks and benefits. All parents/legal guardians will be reminded that they can withdraw themselves and/or their child at any time without consequences.

Wave 1 (parents of first school) parent 9- month follow up will take place in spring of 2020. Wave 1 parent 12-month follow-up will take place in Fall 2020. Wave 2 (parents of schools 2 and 3) and Wave 3 (parents of schools 4 and 5) will follow the same procedures and pattern of timeline of data collection. Data Safety & Monitoring Plan describes participant safety and support plans

# 4.1.2 For the systems-level component of N/E, there are 2 forms of data collection: a barriers/ facilitators discussion quide, and a coordination and implementation monitoring plan tracking log.

These 2 forms of data collection span the 8 service domains relative to improving SRH services for adolescents as outlined by the CDC. The barriers/facilitators discussion guide will be administered in a group discussion format to the Epi Team at baseline and at 12 months during a standing monthly meeting held at the Fort Peck Tribal Headquarters to assess the factors that impede or strengthen the provision of SRH services for Al youth at Fort Peck. The Epi Team's discussion of the barriers/facilitators will be recorded and transcribed. Based on findings from the barriers/facilitators guide, a coordination and implementation monitoring plan will be developed in the form of a tracking log, in order to monitor improved coordination and provision of SRH services. The coordination and implementation monitoring plan tracking log will be completed as part of the baseline data collection and tracked quarterly during a regular monthly meeting of the Epi Team. Dr. Rink and Ms. FireMoon will be the primary research staff-with assistance from two of N/E's consultants, Ms. Adriann Ricker and Dr. Rachel Hallum-Montes-to collaborate with the Epi Team in completing the barriers/facilitators discussion guide, developing the implementation monitoring plan, and tracking the plan's progress toward increasing access to SRH services for Al youth. No identifying data or participants will be collected.

**4.1.3** Incentives: Incentives for the students and parents/legal guardians are based on discussions with N/E's Community Advisory Board and members of the FPCC research team, as well as Dr. Rink's prior experience with research studies involving Indigenous communities. Students will receive \$10 at the baseline, 3-month, and 9-month data collections and \$20 at the 12-month data collection. Parents/legal guardians will receive \$10 at the baseline and 9-month data collections and at each of the 4 sessions of Native Voices, plus \$20 at the 12-month data collection. Similar incentives for students and parents have been previously successful. Epi Team members will not receive incentives for participation in N/E, as it is part of their tribal employment responsibilities.

**4.2 Fidelity. Acceptability and Sustainability Data Collection.** Fidelity recommendations from the National Institutes of Health Behavior Change Consortium will be implemented across the 5 areas of study design, component leader training, delivery of treatment, receipt of treatment, and enactment of treatment skills. The Fidelity, Acceptability, and Sustainability (FAS) of the N/E intervention will be emphasized with a variety of internal processes and data collection methods. The left column describes the FAS component, while the right column describes the corresponding type of data collection and timeline of data collection.

| Fidelity, Acceptability, and Sustainability Component | Types of Data Collection and Timeline |
|---|---|
| Community Advisory Board (CAB) meetings | CAB FAS Meeting Form: quarterly CAB meeting notes: quarterly |
| Team-wide meetings | Team-wide meetings FAS Form: bi-<br>monthly |
| Consistency of staff training | Staff training evaluation log: yearly |
| FAS of coordination/implementation enhancement of Epi Team | Fidelity Reach Log/Staff Field notes:<br>monthly |
| Intervention implementation of Native Stand, Native Voice, and Cultural Mentoring | Fidelity Reach Log/Staff Field notes: each day of intervention |
| Community level FAS | 8 Focus Groups (2 youth, 2 parent, 2 regarding Cultural mentoring, 2 professionals): yearly beginning in Year 3 (Total of 24 Focus Groups) |

**4.2.1 FAS Data Collection:** In consultation with Dr. Hallum-Montes, Dr. Rink, Dr. Cox, and Ms. Firemoon developed four forms to collect FAS data during the implementation of the intervention.

#### Forms:

- 1.) The "Community Advisory Board Meeting Form" will be collected once per quarter after each meeting of the CAB. It will document the barriers and facilitators to intervention implementation discussed at CAB meetings, any social, environmental, political, or bureaucratic contextual factors such as the death of an elder or Tribal Council election year, that may have inhibited or facilitated intervention implementation, and any suggestions to mitigate these barriers the CAB discusses. CAB meeting notes will also be taken during each meeting.
- 2.) The "Whole Team Meeting Form" will document bi-monthly meetings that include Paula Firemoon, Beth Rink, Adriann Ricker, Ramey Growing Thunder, the N/E outreach coordinator, the Cultural Mentor outreach coordinator, and Genevieve Cox. This form will include any barriers and facilitators to intervention implementation discussed, contextual factors (social, environmental, political, or bureaucratic) discussed, suggestions, and who will be responsible for implementing these suggestions.
- <u>3.) The "Staff Training Evaluation Log"</u> will be collected yearly and documents who has been trained, what procedures were followed during training, problems encountered during trainings, and any feedback from the trainings.
- <u>4.) The "Fidelity Reach Log and Field Notes"</u> form includes documenting the delivery of the intervention and any field observations study staff note. It will document the date of the intervention, the length of time the intervention was delivered, specific modules delivered, and any barriers and facilitators to the delivery of the intervention.

The outreach coordinator will also document any environmental, social, political, or bureaucratic barriers or facilitators and suggested solutions to the intervention delivery. With the exception of names of staff trained, no identifying data will be collected. These files will be kept in a locked file cabinet by Genevieve Cox at MSU after data collection.

In addition to the 4 FAS forms, we will implement 8 focus groups at 12 months from inception of the intervention for each year of the 3 years of planned intervention implementation (a total of 24 focus groups). The focus groups will include 6 to 8 individuals per group. The 8 focus groups will consist of 2 focus groups with youth, 2 focus groups with parents, 2 focus groups with the cultural mentors, and 2 focus groups with professionals from schools, agencies, and health care organizations that a re involved in N/E. The focus groups will be recorded and transcribed. Written consent will be obtained from the adults participating in the fidelity and acceptability focus groups. Written consent and assent will be obtained from the parents/legal guardians and their child, respectively, in order for the child to participate in the focus groups. Focus group participants will receive a \$20 incentive. No identifying data will be collected.

#### **SECTION 5: SELECTION AND ENROLLMENT OF PARTICIPANTS**

**4.1 Inclusion Criteria.** To be eligible for inclusion in *NIE*, students must be: 1) 15 to 18 years old; 2) a registered member of a federally recognized tribe or an associate tribal member; and 3) a resident of Fort Peck with a parent/legal guardian. For inclusion in the systems-level component of *NIE*, only those staff members who sit on the Epi Team as representatives of their respective agencies are eligible. Written informed consent will be obtained from the head of each agency represented on the Epi Team and the staff member participating in the Epi Team.

<u>4.2 Exclusion Criteria</u>. Exclusion criteria are minimal due to the CAB's value of inclusion in *NIE*. Exclusion criteria include: 1) not meeting the aforementioned inclusion criteria; and 2) having a medically identified physical or cognitive impairment that would impede their understanding of and participation in the educational content and activities of *Native Stand*. *Native Voices*, and the cultural mentoring program.

**4.3 Study Enrollment Procedures.** Students and their parent/legal guardian will be recruited from each of the study's 5 schools. Based on discussions with school personnel and our previously successful recruitment strategies, recruitment will occur via flyers posted in the schools, letters to the parents, parent-teacher meetings, and word of mouth. Additionally, a parent/legal guardian session that provides an overview of *NIE*, the content and format of the intervention components, and risks and benefits of participation will be held at each of the study's 5 schools. Students and their parents/legal guardians, and students from each cluster, will be recruited for participation at baseline. Students and their parents/legal guardians will be recruited for baseline participation **prior to randomization of the sites.** Students and parents/legal guardians will be assigned unique study identification numbers. No persons who refuse to participate in the study, in whole or in part, will be coerced to engage in any study activity. After written consent and assent is obtained from the parent/legal guardian and child, respectively, they will be enrolled in the study.

#### **SECTION 6: HUMAN SUBJECTS**

- **6.1 Institutional Review Board Approvals.** The study has approval from the Fort Peck Institutional Review Board and the Montana State University Institutional Review Board. In addition, the study has been registered with ClinicalTrials.gov. These aforementioned approvals are in agreement with the conditions for approval to conduct human subjects research as outlined in our Notice of Grant Award from the National Institute of Minority Health & Health Disparities. See Appendices for research approvals.
- <u>5.2. Human Subjects' Characteristics</u>. There three groups participating in the study in which data will be collected include: 1) 15 to 18-year-old youth; 2) a parent/legal guardian; and 3) members of the Fort Peck Epi Team.
- <u>6.3. Data Sources for Human Subjects Based on Intervention Levels.</u> Our study includes four levels of intervention:
- 1) Individual Level. Native Stand is a school-based, 27-module STI-, HIV-, and teen pregnancy-prevention curriculum, originally developed for rural white youth and adapted for Native youth in 2008. For our study, an adaptation of Native Stand will be implemented over 9 months in the 5 tribal high schools to educate Fort Peck tribal youth on sexual risk behavior prevention strategies by tailoring and reducing the 27 modules into 18 modules, as well as including specific community-relevant traditional and contemporary cultural lesson plans. Trained project staff will deliver Native Stand in school classroom settings during the school year as part of each school's curriculum. American Indian students only will be recruited for Levels 2 and 3 and for data collection.
- 2) Family Level. Native Voices is a video-based HIV/STI prevention intervention designed for Al adolescents, which includes condom use, negotiation skills, group discussion, and role playing. Native Voices will be adapted from 1 module into 4 modules, as recommended by the creators of Native Voices for curriculum adaptations involving family members, and will involve students and one of their parents/legal guardians. Our adaptation of Native Voices promotes discussions between the students and their parent/legal guardian regarding STI, HIV, HCV, and pregnancy prevention relevant to the Fort Peck tribal community. Ms. FireMoon will implement Native Voices to groups of 10 students and their parents/legal guardians at one time at the local high school for 2 hours in the evening. Native Voices' 4 modules will be implemented over 9 months.
- 3) Community Level. The third level of our study is a cultural mentoring component that pairs Al youth with older adults and elders to discuss traditional American Indian beliefs and practices about reproductive health. To our knowledge, no mentoring programs have been designed for Al youth that specifically address sexual and reproductive health issues. The mentoring program is based on Assiniboine and Sioux traditional knowledge and the National Mentoring Partnership standards for mentoring. The mentoring program was designed specifically for Fort Peck youth by the Fort Peck Tribes' Language and Cultural Department and has been in existence for 5 years. Our study integrates this cultural mentoring program into our study's overall framework. Our cultural mentoring program will include older male and female tribal members from the Assiniboine and Sioux tribes. The older adults will be paired with the youth participating in the intervention by gender and tribal affiliation. Students participating in Native Stand and Native Voices with their parent/legal guardian will meet monthly over the course of 9 months one-on-one with their mentor and monthly in mentor mentee small groups. Topics addressed in the cultural mentoring program include overall information on Assiniboine and Sioux cultural beliefs, values, and ceremonies, as well as more specific information on Assiniboine and Sioux cultural beliefs and values regarding sex, having children, parenting, and relationships.

4) Systems Level. The fourth level of our study is a community-level strategy that involves mobilizing a network of education, health care, and social service agencies at Fort Peck to coordinate reproductive health services for 15- to 18-year-old Al youth over a 12-month period. The systems-level approach will utilize existing tribal infrastructure by enhancing the work of the established Fort Peck Tribal Epidemiology Team (Epi Team). The Epi Team is a local committee made up of the Fort Peck Tribal Health Department; Indian Health Service (Poplar Service Unit and Wolf Point Service Unit); the Roosevelt County Health Department; and school nurses from the Fort Peck Health Promotion and Disease Prevention Program. The Epi Team meets monthly and has been in existence for 15 years with the purpose of monitoring diseases on the reservation and the health status of the Assiniboine and Sioux tribes. As part of N/E, the Epi Team is tasked with improving the coordination and implementation of STI, HIV, and HCV screening, condom distribution, contraceptive services, and pregnancy testing on the Fort Peck Reservation.

5.3.1. Data Collection Materials for Human Subjects. For the individual-, family-, and community-level components of N/E, there are two forms of data collection: a student survey administered at baseline and at 3, 9, and 12 months after intervention inception, and a parent/legal guardian survey administered at baseline and at 9 and 12 months after intervention inception. The student survey will assess participation in Native Stand, Native Voices, and the cultural mentoring program. The parent survey will assess participation in Native Voices. Ms. FireMoon and the study's outreach coordinator will oversee the administration of the student surveys and the parent/legal guardian surveys. The student surveys and parent/legal guardian surveys will be completed utilizing REDCap. Between Years 2-4, 456 students and one of their parents or legal guardians will participate in N/E's data collection. Student surveys for baseline, 3 months, and 9 months will be administered to groups of 20 students at a time during regularly scheduled classes in an assigned classroom by Ms. FireMoon and the study's outreach coordinator. During data collection, groups of 20 students will be appropriately spaced in the classroom in order to ensure privacy, and survey instructions will be presented to students prior to REDCap administration. Ms. FireMoon and the study's outreach coordinator will thoroughly review the assent form with the students at the baseline data collection, which will include a description of N/E, types of questions that will be asked, and potential risks and benefits of participating in N/E. All students will be reminded that they can withdraw at any time without consequences. For students that graduate from high school prior to the 12 months data collection, they will be contacted by Ms. FireMoon directly to complete the 12 months data collection (during evening hours) at the high school they graduated from following the same procedure described above. This same procedure will be followed if the data collection time point occurs for some reason when school is not in session. The parent survey will be administered during evening hours at the high school in an assigned classroom by Ms. FireMoon and the study's outreach coordinator. We will use the same REDCap procedures for parents/legal quardians that are described for youth above. In addition, written consent will be obtained from the parents/legal guardians prior to their participation in the study. Ms. Firemoon and the study's outreach coordinator will review the informed consent with the parents/legal guardians at the time of data collection.

For the systems-level component of N/E, there are two forms of data collection: a barriers/facilitators discussion guide and a coordination and implementation monitoring plan tracking log. These two forms of data collection span the 8 service domains relative to improving SRH services for adolescents as outlined by the Centers for Disease Control and Prevention (CDC). The barriers/facilitators discussion guide will be administered in a group discussion format to the Epi Team at baseline and at 12 months during a standing monthly meeting held at the Fort Peck Tribal Headquarters to assess the factors that impede or strengthen the provision of SRH services for Al youth on the Fort Peck Reservation. The Epi Team's discussion of the barriers/facilitators will be recorded and transcribed. Based on findings from the barriers/facilitators guide, a coordination and implementation monitoring plan will be developed in the form of a tracking log in order to

monitor improved coordination and provision of SRH services. The coordination and implementation monitoring plan tracking log will be completed as part of the baseline data collection and tracked at 3, 6, 9, and 12 months during a regular monthly meeting of the Epi Team. In collaboration with the Epi Team, Ms. FireMoon, Ms. Adriann Ricker, and Dr. Rink will complete the barriers/facilitators discussion guide, develop the implementation monitoring plan, and track the plan's progress toward increasing access to sexual and reproductive health services for American Indian youth on the Fort Peck Reservation.

All students attending each school will be eligible to participate in the individual-level Native Stand curriculum, as it will be incorporated into that school's regular curriculum. In order to be eligible for inclusion in the family and community-level components of N/E and the data collections, students must be: 1) 15 to 18 years old; 2) a registered member of a federally recognized tribe or an associate member; 3) a resident of the Fort Peck Reservation with a parent/legal guardian; and 4) enrolled at one of the five schools participating in N/E.

Exclusion criteria are minimal due to the value the CAB places on inclusion in N/E's program implementation. Exclusion criteria include 1) not meeting the aforementioned inclusion criteria, and 2) having a physical or cognitive impairment that would impede the student's understanding of and participation in the content of Native Stand, Native Voices, and the cultural mentoring program. Study-enrolled students must agree at the outset to participate in Native Stand, Native Voices, and the cultural mentoring program, and agree to complete the survey at baseline and at 3, 9, and 12 months during and shortly after their cluster's program. Parents/legal guardians must also agree to participate in Native Voices and complete the parent/legal guardian survey at baseline and at 9 and 12 months. No persons will be coerced to engage in any study activity, and anyone may refuse to participate at any time. After written consent and assent are obtained from the parents/legal guardians and their children, respectively, they will be enrolled in the study. For inclusion in the systems-level component of the study, only those staff members who sit on the Epi Team as representatives of their respective agencies are eligible. Written informed consent will be obtained from the head of each agency represented on the Epi Team and the staff member participating in the Epi Team.

If at any point in the study a student discloses abuse, they will be referred to the appropriate person or organization. For example, a research participant who is under the age of 18 and in school who discloses that he or she is being abused at home will be referred to the counselors in the school for assistance, with the possibility of joint reporting to Child Protective Services. Students will be informed during the informed consent process that any abuse they may disclose will be reported, since the members of the research team and the interviewers are mandated reporters.

Another form of data collection that involves human subjects is related to Aim 3 of our study, which is to evaluate the fidelity and acceptability of N/E. As part of Aim 3 we will conduct focus groups. We will implement 8 focus groups at 12 months from inception of the intervention's curricular components for each year of the 3 years of planned intervention implementation (a total of 24 focus groups). The focus groups will include 6 to 8 individuals per group. The 8 focus groups will consist of 2 focus groups with youth, 2 focus groups with parents, 2 focus groups with the cultural mentors, and 2 focus groups with professionals from schools, agencies, and health care organizations that are involved in N/E. Written consent and assent will be obtained from adults, parents/legal guardians, and youth, respectively. Focus groups will be recorded and transcribed. No names or other identifying information, such as an address, will be included on the transcripts. However, age and gender will be recorded. After each focus group, the focus group facilitator will check the audiotapes for clarity. Clear audiotapes will be transcribed. Audiotapes that are not sufficiently clear, or do not have adequate volume to transcribe, will not be transcribed. Instead, responses typed or directly written down by the focus group guide during the interview will be used as the transcript for content analysis. Names of students or others identified in the transcripts will be blacked out in order to ensure confidentiality.

Student Survey: To assess students' participation in N/E, we draw from several existing measurements that have been implemented and validated in research studies with Al youth. Primary outcome measure: Condom use will measure frequency of condom use relative to frequency of sex during sexual intercourse using questions derived from the Risk Behavior Assessment. Secondary outcome measures: These will include the number of sex partners; age of onset of sexual intercourse; frequency of sexual intercourse; pregnancy history; frequency and type of birth control used during sexual intercourse relative to the frequency of sexual intercourse; and frequency and types of substance use (cigarettes, marijuana, alcohol, and methamphetamine). Tertiary outcome measures: Parent/legal guardian communication is measured by the frequency and types of SRH topics that parent/legal guardian and child discussed. Cultural identity is measured using two established measurements: One measure assesses the extent to which a student identifies with his or her American Indian culture and feels cultural pride, and the other measure assesses frequency and type of participation in cultural activities. Access to SRH services is measured by frequency and type of SRH service used (ever been tested for STIs and follow-up, ever been tested for HIV and follow-up, ever been tested for HCV and follow-up, ever been pregnant/gotten someone pregnant and follow-up). Other variables to be measured in N/E that assess attitudes, intentions, skills, and mental health are: Motivation to avoid STIs, HIV, HCV, and pregnancy, as measured by asking students how important it is to them to keep themselves (or someone else) from getting an STI, HIV, and HCV, and how important it is to them to keep from getting pregnant or getting someone pregnant. Intention to use condoms and/or birth control is measured by asking students how likely it is they will use condoms and/or birth control the next time they have sexual intercourse. Intention to abstain from sex is measured by asking students how likely it is that they will not participate in sexual intercourse. Condom and birth control use self-efficacy is measured by assessing confidence in one's ability to use condoms and birth control. Refusal skills regarding sex are assessed by how strongly students believe they can say no to sex. Knowledge about STIs, HIV, HCV, pregnancy, and healthy relationship characteristics are measured using true/false/don't know questions. Mental health is assessed using two established measures: One measure assesses depression using the C-ESD, and the other measurement assesses exposures to stressful life events by assessing lifetime occurrences of a series of negative events. Standard demographic measures in the student survey are age, gender, sexual orientation, school, and highest grade completed.

<u>Parent/Legal Guardian Survey.</u> The parent/legal guardian survey is based on parents'/legal guardians' participation in Native Voices. It includes a list of SRH topics about which the parent/legal guardian has spoken to the child and the frequency of times discussed. The parent/legal guardian measures have been validated in previous studies evaluating parent/child SRH communication and have been used by Dr. Rink in her Greenland studies. The SRH topic list and frequency is the same as in the student survey, only adapted for parents/legal guardians. Standard demographic measures included in the parent/legal guardian survey are age, gender, marital status, highest grade completed, and occupation.

<u>Barriers/Facilitators Discussion Guide.</u> The barriers/facilitators discussion guide is a qualitative assessment using open-ended questions that address the factors impeding and facilitating SRH services for Al youth on the Fort Peck Reservation. The guide is based on the 8 service domains for evidence-based clinical practices outlined in the CDC's Contraceptive and Reproductive Health Services for Teens: Evidence-based Clinical Best Practices Guide(80-82)-namely, contraceptive access; provision of hormonal contraception/IUD; emergency contraception; cervical cancer screening; STI/HIV/HCV testing and treatment; cost, confidentiality, consent; health center infrastructure; and health center environment.

<u>Coordination and Implementation Monitoring Plan Tracking Log</u>. The tracking log will monitor the progress toward completion of the 8 SRH service domains identified from the barriers/facilitators discussion

guide and corresponding evidence-based clinical practice elements.

**Focus Groups.** Data collection related to Aim 3 of our study, which is to evaluate the fidelity and acceptability of N/E, includes a focus group guide, as described above. The Aim 3 focus groups will include questions such as what experiences/activities they liked and/or did not like about the intervention, what educational information they did and/or did not like about the intervention, and what recommendations they have for improving the intervention.

#### Table 2. NIE Measures.

Table 2. N/E Measures.

| Data Collection Instruments and Measures | Data<br>Base | | llectio | | Description of Measures |
|---|---|---|---|---|---|
| Student Survey | | 3 | 9 | 12 | Number of Items; Scale Anchors; Benchmark Values |
| Primary Outcome Variable | *** | | | | Al Si |
| Proportion of condom use during sexual intercourse (SI) | X | Х | X | X | 2 items; number of times condom used relative to number of times had SI |
| Secondary Outcome Variables | | | | | |
| Age of onset of sexual intercourse | X | X | X | X | 2 items; ever had SI & age at first SI |
| Number of sex partners | X | X | X | X | 2 items; lifetime & past-month sex partners |
| Frequency of sexual intercourse | X | X | Х | X | 1 item; frequency of SI in past month |
| Pregnancy history | X | X | X | X | 1 item; number of pregnancies |
| Type & frequency of birth control (BC) during sexual intercourse | X | X | X | X | 3 items; type of BC use and number of times BC used during SI |
| Type & frequency of substance use (SU) during sexual intercourse | X | X | X | X | 1 item measures SU with SI; 5 items measure lifetime and past month SU |
| Tertiary Outcome Variables | | | | | |
| Type & frequency of parent/legal guardian–child SRH communication | X | Х | X | Х | 24 items Likert scale; higher score = higher communication |
| Cultural identity & participation in cultural activities | Х | Х | X | X | 3 items cultural identity ( $\alpha$ = .75); 2 items cultural activities engagement ( $\alpha$ = .46) |
| Type & frequency of SRH services | X | X | X | X | 9 items; frequency, type, and follow-up of SRH services used |
| Other Variables | 7.7011 | | | | |
| Motivation to avoid STIs, HIV, HCV, & pregnancy | × | X | X | X | Up to 9 items; 1 (very true) to 5 (very untrue); 1 = more positive attitude/motivation |
| Condom & birth control use intention & self-efficacy | X | X | X | X | 4 items per intention; 1 (very true) to 5 (very untrue); 1 = higher intention; 6 self-efficacy items; 1 (very easy) to 4 (very hard); 1 = high self-efficacy |
| Abstinence | X | X | X | X | 3 items; 1 (strongly disagree) to 4 (strongly agree); 4 = more supportive of teen abstinence |
| Refusal skills regarding sex | Х | Х | X | Х | 7 items; 1 (I definitely can say no) to 5 (I definitely can't); 1 = stronger refusal skills |
| Knowledge of STIs, HIV, HCV, pregnancy, & health relationships | X | Х | X | Х | Range of 4 to 10 items per topic; True/False/DK; Average proportion of guestions correct |
| Depression (CES-D) & exposure to stressful life events | Х | Х | X | Х | CES-D — 7 items ( $\alpha$ = .80); Life Events — 24 items; Yes/No; number of events observed |
| Student Demographics | | 45 0 | | N N | |
| Age, gender, sexual orientation, school, highest grade completed | X | X | X | Х | 4 items |
| Parent/Legal Guardian Survey | 2 | | | | |
| Type & frequency of parent/legal guardian–child SRH communication | X | | X | Х | 24 items Likert scale; higher score = higher communication |
| Parent/Legal Guardian Demographics | | | | | |
| Age, gender, marital status, highest grade completed, occupation | X | | X | X | 5 items |
| Barriers/Facilitators Discussion Guide | 22. | 10.00 | | | |
| 8 Service Domains for Evidence-Based Clinical Best Practices | X | | | Х | Open-ended questions about barriers/facilitators for: contraceptive access, provision of hormonal contraception/IUD, emergency contraception, cervical cancer screening, STI/HIV/HCV testing and treatment, cost confidentiality, consent, health center infrastructure, & health center environment. |
| Coordination & Implementation Monitoring Plan Tracking Log | Base | 3 | 6 9 | 12 | |
| 8 Service Domain Elements | X | X | XX | X | Tracks action steps, timeline, and responsible party |

#### 6.4 Potential Risks

There may be minor risks to agreeing to participate in N/E. Student and parent/legal guardian participants may be asked some questions that make them feel uncomfortable, sad, or confused (e.g., questions about sexual risk behaviors). For participants in the systems-level component of the study that evaluates the enhancement of the coordination of SRH services, we anticipate low to no risks, since none of the data being collected will be of a personal nature. For Aim 3, which uses focus groups as one method of data collection to evaluate the fidelity and acceptability of N/E, we also anticipate low to no risk, since none of the data being collected will be of a personal nature. All study participants will be informed that they may choose to stop their participation in N/E at any time or decline to answer a particular question asked of them on a data collection instrument or during a data collection process. We will inform study participants that the study is voluntary and that they can withdraw from the study, by stating that they want to do so, at any time over the course of the study.

#### 6.4.1. Adequacy of Protection Against Risks

Nenunkumbi/Edahiyedo ("We Are Here Now'?: A Mult-level, Multi-component Sexual and Reproductive Health Intervention for American Indian Youth

#### A. Recruitment and Informed Consent

The high schools in Frazer, Wolf Point, Poplar, Brockton, and Culbertson will serve as the primary recruitment sites for our study. Based on discussions with school personnel and our previously successful recruitment strategies, recruitment will occur via flyers posted in the schools, letters to the parents, parent-teacher meetings, and word of mouth. Additionally, a parent/legal guardian session that provides an overview of N/E, the content and format of the intervention components, and risk and benefits of participation will be held at each of the study's 5 schools. Students and their parents/legal guardians from each cluster will be recruited for participation at baseline (Q2 of Year 2). At the time of the student data collection at baseline, Paula FireMoon and the study's outreach coordinator will thoroughly review the assent form with the students, which will include a description of the N/E curricular components, types of questions that will be asked in the data collection, and potential risks and benefits of participating in N/E. All attempts will be made to help the students understand the nature of the study. Paula FireMoon and the study's outreach coordinator will thoroughly review the consent forms with the parents, which will include a description of N/E, types of questions that will be asked, and potential risks and benefits of participating in N/E. Parents will provide informed consent for their child as well as for themselves prior to their participation in the Native Voices curriculum. For the systems-level component, Epi Team members will complete an informed consent at the time of the first barriers and facilitators discussions in Year 2. If members change from one such discussion to the next, new informed consents will be collected as needed. For the Aim 3 focus groups, informed consent will be obtained from the mentors or the professionals representing agencies prior to their participation in the focus groups as key stakeholders. Consent and assent will be obtained from parents/legal guardians for their participation in a parent group, and from parents/legal guardians and their children, respectively, for the children's participation in a children's focus group. All study participants, both adults and children, will be reminded that they can withdraw at any time without consequences. No study participant will be coerced to participate in the study, in whole or in part. Human subjects approval has been received from the Fort Peck IRB for the Year/Aim 1 refining, tailoring, and finalizing the intervention design. At that point, new applications to the Fort Peck IRB and the MSU IRB will receive approvals prior to study start.

# B. Protection Against Risk

Because N/E involves children ages 15 to 18 years old, we will ensure that parents/legal guardians understand the research protocol and are able to provide informed consent for themselves and their participating children in this minimal-risk intervention study. To preserve confidentiality, all data collection forms will be coded with a unique identifier. All of the project data, including the audiotapes and transcripts, will be labeled with study identification numbers and stored separately from the informed consent forms. Consent forms will be kept in a locked file cabinet in Paula FireMoon's office at Fort Peck Community College, which has a combination lock on the door that only Paula FireMoon knows. All survey data will be stored in a password-protected file on a password-protected computer at Fort Peck Community College in Paula FireMoon's office. Focus group documents will be uploaded onto MSU's Box server, a password-protected cloud data storage system. All of the project data-including the audiotapes, transcripts, and interview summaries with study identification numbers-will be stored separately from the informed consent forms in a locked file cabinet in Dr. Rink's locked office at Montana State University, to which only Dr. Rink and the MSU-based research program manager, Genevieve Cox, will have access. Once the focus groups have been transcribed and checked for validation against the audiotapes, the audiotapes will be destroyed in order to ensure no voice recognition. At the end of the project, all of the deidentified data files (though not individual surveys) will be returned to Fort Peck Community College and stored in the Fort Peck research archives in Poplar, Montana, as is required by the Fort Peck IRB. Please note that none of the data returned to Fort Peck Community College will contain a study participant's name or contact information to ensure that personal information collected during the study is not associated with a study participant's name. Data files at Fort Peck Community College will be kept in

accordance with federal law regarding research material. Also, the study participants (completing surveys or participating in focus groups) will be informed of where the data will be stored during the informed consent process. All data will be kept in accordance with federal law requirements regarding research material.

#### **SECTION 7: DATA SAFETY MONITORING PLAN**

This plan describes the general data and safety monitoring procedures for the proposed research activities, including the responsibilities of the PI, Co-Investigators, and the Community Advisory Board, as well as the reporting of adverse events. This data safety monitoring plan was submitted with our R01 proposal and approved by the review panel, project officer and grants management officer at NIH. Protocols for data safety have also been reviewed and approved by the Fort Peck and Montana State University Institutional Review Boards.

The principal investigator, Elizabeth Rink, Ph.D., the Fort Peck-based project director Paula FireMoon, M.Ed. (co-investigator), and the Fort Peck Tribes' Language and Culture Department director Ramey Growing Thunder, MA (co-investigator), will be responsible for knowing and adhering to the cultural protocols and official policies of the Fort Peck Tribes and the five participating high schools; the Fort Peck IRB policies and procedures; and the MSU IRB policies and procedures. Dr. Rink will be the lead on the Fort Peck and MSU IRB correspondences and reports. She will maintain accurate documentation of the Fort Peck and MSU IRB correspondences and reports on her password-protected desktop computer in her locked office at MSU. The PI and the local Fort Peck co-investigators (FireMoon and Growing Thunder), who together will oversee the intervention at Fort Peck, are responsible for documentation and handling of all possible study-related adverse events. They all are experienced in conducting research and implementing and evaluating community based programs with American Indian youth. Rink and FireMoon have experience conducting such research related to sexual and reproductive health. All will assure that data collection and safety monitoring systems are in place and implemented-Mrs. Growing Thunder for the mentoring program and Ms. FireMoon for the other intervention components.

#### The Data and Safety Monitoring Plan includes the following descriptions:

- 1. Potential adverse events resulting from participation;
- 2. Procedures to safeguard against those events;
- 3. Response procedures for adverse events;
- 4. Reporting procedures foradverse events;
- 5. Oversight.

#### 1. Potential Adverse Events Resulting from Participation

- A. Possible violation of confidentiality;
- B. Possible violation of cultural protocols or official policies;
- C. Possible discomfort due to completing data collection tools:
- D. Possible embarrassment in disclosing personal sensitive information;
- E. Possible disclosure of information about intended physical harm to victims, or abuse of children, that would need to be reported to the child welfare agency, and an investigation of the allegations(s) and further action, as indicated, that could ensue;
- F. Possible dissatisfaction with completing the data collection tools:
- G. Possible dissatisfaction with the intervention activities.

#### 2. Procedures to Safeguard Against Adverse Events

All data collection protocols include a form on which the research team will record any problems with the data collection, concerns about the adolescents, or unusual occurrences during the conduct of the intervention or the collection of data. These forms allow the team to quickly review and respond to any possible concerns or adverse effects. The form includes contact information for Rink, FireMoon, and Growing Thunder. One or more of them will always be available during data collection. During phone conferences and meetings (weekly during the intervention periods and monthly otherwise), all problems and concerns will be discussed and processed among themselves, and with other project personnel as needed.

- A. <u>Informed Consent:</u> Ms. FireMoon and the N/E outreach coordinator will review the consent forms with the parents/legal guardians at baseline to ensure their understanding of the purpose of N/E, types of questions they will be asked, and the study's potential risks and benefits. They will be reminded that they can withdraw themselves or their child at any time without consequences. Likewise, Ms. FireMoon and the study's outreach coordinator will thoroughly review the assent form with the 456 students to be enrolled, which will include a description of N/E, types of questions that will be asked, and potential risks and benefits of participating in N/E. All students will be reminded that they can withdraw at any time without consequences. After written consent and assent are obtained from the parents/legal guardians and their child, respectively, they will be enrolled in the study. For inclusion in the systems level component of the study, only those staff members who sit on the Epi Team as representatives of their respective agencies are eligible. Written informed consent will be obtained from the head of each agency represented on the Epi Team and the staff member participating in the Epi Team. Written consent and assent will be obtained from the maximum of 192 adult professionals, parents/legal guardians, and youth, respectively, for participation in the 24 planned focus groups. All study participants will be informed of where and how the data will be stored during the informed consent process.
- B. Confidentiality and Data Safeguards: To ensure confidentiality, all information will be coded using a unique identification number so that it cannot be associated with any individual. All of the survey data will be labeled with study identification numbers and stored separately from the informed consent forms in a locked file cabinet in Paula FireMoon's locked office at Fort Peck Community College. A master sheet, with individual names and their respective unique study identification numbers, will be kept in a separate locked file that can be accessed only under supervision of the PI or Project Director. The data collection from the student surveys and parent/legal guardian surveys will be downloaded using the RedCap software into the MSU Box server, a file-sharing cloud server, for storage. This is a password protected virtual storage system for de-identified research materials that only specified invited individuals (members of the research team) may view. The audiotapes of the focus groups will be stored separately from the informed consent forms in a locked file cabinet in Dr. Rink's locked office at Montana State University. All other focus group data including the deidentified transcripts, interview summaries, and the results of the content analysis will be stored on the MSU Box server. All data entered into Box as part of the project's computerized database will be identified by unique identification number only. The entire research team and all other project personnel who come in contact with data or with the human subjects of the intervention will sign a formal oath of confidentiality. The information gathered will be used only for scientific, program evaluation, or instructional purposes. No information about the identities of study participants will be published or presented at conferences.
- C. <u>Cultural Protocols and Tribal/Schoo/ Policy Safeguards:</u> Dr. Rink and Ms. FireMoon will be responsible for working with the study's CAB, other investigators, and consultants to ensure that the intervention adheres to the cultural protocols and official policies of the Fort Peck Tribes; the Fort Peck IRB policies and procedures; and the MSU IRB policies and procedures. Tribal elders will be consulted on traditional topics and protocols that cannot otherwise be addressed by Ms. FireMoon, the study's CAB members, and Mrs. Growing Thunder. Dr. Rink and Ms. FireMoon will hold quarterly meetings with the study's CAB. All documents related to N/E will be developed, reviewed, and vetted by the study's CAB members as necessary during the quarterly CAB

meetings. Similarly, all data resulting from N/E will be reviewed, interpreted, and approved by the CAB. If necessary, Dr. Rink and Ms. FireMoon will also meet individually with CAB members to discuss the study's research protocols, data collection instruments, and findings. In addition to the CAB-related meetings, Dr. Rink, Ms. FireMoon, and Mrs. Growing Thunder will hold monthly team meetings to discuss the study's research protocols, implementation strategies and progress, research-related documents, data collection procedures, and analysis. Any concerns brought up by the CAB or other members of the research team will be discussed until a resolution is reached.

As part of N/E we will use fidelity and acceptability recommendations from the National Institutes of Health Behavior Change Consortium. These recommendations address study design, component leader training, delivery of treatment, receipt of treatment, and enactment of treatment skills. In order to assess the fidelity and acceptability of N/E, data sources will include: staff training logs, fidelity reach logs, staff field notes, notes from discussions at monthly team meetings, and notes from discussions with CAB members and at CAB meetings. Focus groups are an additional qualitative measure to assess fidelity and acceptability. These fidelity and acceptability data sources will assist the MSU based and FPCC-based research teams and the CAB to monitor the enrollment of students and parents/legal guardians into the study, monitor the data submission, quality-check the data being reported, avoid potential study related bias or inconsistencies, and prepare interim reports when necessary.

- D. <u>Mandatory Reporting Safeguards:</u> Procedures to prevent the violation of confidentiality will be limited by mandatory reporting requirements. Subjects will be informed in the consent document that the research team must report to authorities: (1) physical injury to any child caused by other than accidental means; and (2) information from a study participant that leads the research team to believe a person is in imminent danger of physical harm. The project personnel will inform parents or guardians if, in the judgment of the research team/project personnel, their child (under 18) is in imminent danger of trying to harm him/herself.
- E. Research Team Safeguards: All research team/project personnel who interface in any way with intervention protocols, data collection, or data analysis are required to complete and be up-to-date with the extensive Collaborative Institutional Training Initiative (CITI) training and testing program and the NIH Good Clinical Practice Training. Weekly or monthly meetings or phone conferences will occur among the key personnel for ongoing training, monitoring of protocols, and problem solving. Questions concerning data collection will be processed during this time. The Project Director (Ms. FireMoon) will coordinate and oversee all activities at the data collection sites and will report all activities, concerns, and questions to the PI on an ongoing basis. Prior to the start of the intervention cycle, the entire team on the ground in the Fort Peck communities, including personnel to be hired, will be trained to identify events that would fall under mandatory reporting guidelines. These include physical injury to any child caused by other than accidental means, or information from a student participant that leads staff to believe a person is in imminent danger of physical harm.
- F. <u>Discomfort with Completing Intetvention Data Collection Instruments or Disclosure Safeguards:</u> During the course of participation in the research, a participant may have questions concerning the data collection tools. Either the Project Director (Ms. FireMoon) or the Outreach Coordinator (to-be-hired) will be available at each school data collection event to answer questions. Likewise, the mentoring program Director (Mrs. Growing Thunder) and her Community Mentorship Coordinator (to-be-hiredDo you want to add name?) will be available at each group mentoring meeting to answer questions. To prevent discomfort or embarrassment, the Project Director (Ms. FireMoon) is trained in counseling and has experience in therapeutic interaction. The PI has training and previous work experience in clinical social work and will be available to all participants via cell phone, email, or in person when she is at Fort Peck to address any concerns regarding the data collection instruments. The remaining staff will receive specialized training in sexual and reproductive health and will also be available to participants.

G. <u>Dissatisfaction Safeguards:</u> Participants will be encouraged to discuss with the PI or Fort Peck-based project personnel any possible dissatisfaction with the data collection tools or intervention activities.

# 3. Response Procedures for Adverse Events

- A. <u>Discomfort with Disclosure:</u> All project personnel working in the reservation communities are under the supervision of the PI, who is highly trained in counseling. Any participant experiencing embarrassment or discomfort when completing data collection tools will be responded to in a compassionate and professional manner. If a participant experiences any other adverse reactions to the data collection tools or intervention activities/sessions, the participant will be referred to IHS Poplar Service Unit, HIS Wolf Point Service Unit, or the Fort Peck Tribes Health Promotion and Disease Prevention Program (HPDP) on the Fort Peck reservation, which all have trained psychotherapists available to tribal members. Participants will also be encouraged to contact the research team/project personnel in the event of a late adverse reaction and will receive specific written and verbal instructions during the project consent procedures about how to do so if the need arises.
- B. <u>Mandatory Reporting</u>: Serious adversities shared by subjects that need to be reported by the research team/project personnel include physical abuse and neglect or threat of physical harm to self or others. To anticipate these concerns, the research team/project personnel have established procedures and guidelines to respond to risk disclosures among participants.

Four types of situations require special procedures:

- Suicide thoughts or attempts: Two types of risks will be addressed in the project: (a) ideation or presentation of thoughts or interest in suicide, and (b) action, which includes both thoughts of suicide as well as the presence of a plan and means to accomplish a suicide act. As participants complete the data collection instruments, key personnel will review instruments and items for response values that indicate concern. Based on the response values, these key personnel will collectively review disclosed information and, if deemed necessary, conduct follow-up inquiry with the participant to further determine level of risk. If the participant is determined to present immediate risk, a referral will be made to one of the following, depending on which is most appropriate for the situation: IHS Poplar Service Unit, IHS Wolf Point Service Unit, or Fort Peck Tribes' Health Promotion and Disease Prevention Program, which offers mental health services to youth in schools. If the disclosure is the result of one of the written items on the data collection tools, Ms. FireMoon will contact the participant by telephone. If the disclosure occurs during an on-site session, the session leader will follow through with an in-depth interview to clarify the presence of suicidal risk and develop a plan of action. Session leaders and mentors will be trained and required to identify suicidal risks in both the domains of ideation and action. Session leaders will follow up in the same way and inform the PI. In the most extreme cases of risk, the PI then assumes follow-up responsibility for the plan of action.
- <u>Abuse:</u> Child abuse concerns may arise from any or a combination of the following sources: (a) the youth verbally indicates that abuse has occurred or is occurring; (b) the youth answers one or more data collection tool items suggesting the possibility of abuse; (c) the youth is observed being treated in an abusive manner; (d) the youth is observed with bodily injury (e.g., bruise, burns, black eyes) whose origin appears to differ from the explanation given of the injury. At any time during the completion of the data collection instruments, or during intervention sessions, if any of the above information leads key personnel or mentors to suspect abuse or neglect of children, documented steps will be followed to obtain additional information and personnel will contact the Pl. Based on the information, the team will determine appropriate further inquiry and follow-up. Based on the information, the team will develop a safety plan that may include a participatory report to the Fort Peck Tribes/BIA Child Protective Services

agency, and/or possible referral to the Fort Peck Tribes' Family Violence Resource Center based in Wolf Point.

- <u>Threat of danger to others:</u> The threat of danger to others includes disclosure of potential physical harm by a participant to others, including members of the participant's family or other individuals in the school or community. At any time during completion of data collection tools or during intervention sessions, if any information emerges suggesting the threat of harm to others, the team will review the information and determine next steps in accordance with the law, school policies, and the guidance of the CAB and project partners.
- <u>Addiction:</u> Addiction to substances is a condition characterized by compulsive substance intake, craving, and seeking, despite negative consequences associated with the substance(s) used. This project does not directly address substance abuse and addiction. However, the student survey asks about substance use, and some intervention sessions related to substance use occur outside of school settings. A situation may occur where a participant reveals information or exhibits characteristics that suggest addiction to substances. The key personnel and mentors will be trained to recognize signs and symptoms of addiction. Together with the PI they will determine the best response and plan for referral to Spotted Bull Addiction Services based in Poplar on the reservation.
- C. <u>SRH Health Risks and Needs:</u> Due to the intervention and research subject matter of sexual and reproductive health, participants may reveal information during data collection or intervention sessions that suggests either sexually transmitted infections, HIV, HCV, or suspected pregnancy. Key personnel and mentors will have received training on the services available through the local IHS Service Units to test and treat STIs, HIV, HCV, and/or to provide pregnancy testing and prenatal care. Participants who present these issues will be referred to the appropriate health practitioners for care, and project personnel will follow up with participants as needed to ensure action was taken to address health risks. The intervention program itself will encourage youth to access services for disease and pregnancy prevention.

# D. Reporting Procedures for Adverse Events

The anticipated potential adversity inherent in the completion of the student survey is limited and will be addressed by the timely intervention of the key personnel and mentors, as appropriate-all with prior skills and/or training in risk assessment and mandatory reporting requirements. The occurrence of adverse events will be reported to the MSU and Fort Peck IRBs, the Data and Safety Monitoring Committee, and others as appropriate including the participating schools.

- E. <u>Reporting Procedure for Serious Unanticipated Adverse Events:</u> In the event of an unanticipated serious adverse event, the PI and Project Director will ensure that these events are reported to the NIH Program Official within hours by phone, fax, and/or email and will submit a written report to the Program Official no more than two days later. Project personnel will also utilize the following reporting procedures:
  - 1) When the research team/project personnel become aware of a serious adverse event, reporting requirements must be implemented in a timely manner.
  - 2) The PI completes an Adverse Event Report and submits it to the MSU and Fort Peck IRB Chairs, to the project's Data and Safety Monitoring Committee, and to the project Community Advisory Board. The CAB will help identify culturally and socially appropriate ways of remedying adverse events.
  - 3) The Chairs will convene expedited meetings of their respective IRBs. First the Fort Peck IRB and then the MSU IRB, with input from the PI and the Data and Safety Monitoring Committee, will review the study protocol and determine what further action to take based on the best interests of the participants and of the research.

#### F. Oversight

The boards that provide oversight to *NIE* are:

- · Community Advisory Board
- The Fort Peck Institutional Review Board
- · The Fort Peck Tribal Executive Board
- Montana State University Office of Research Compliance
- Montana State University Office of Sponsored Programs
- The Montana State University Institutional Review Board
- Data Safety and Monitoring Board

For the purposes of the Data Safety and Monitoring Plan, the Data Safety and Monitoring Board (DSMB) will be chaired by Dr. Jared Jobe, retired NIH program officer, Dr. David Huh, a researcher and statistician, Dr. William Lambert, a researcher, and Dr. Cynthia Pearson, a researcher. Meetings of the Committee will occur semi-annually by telephone or Zoom, and unless closed by the Chair, will be joined by the PI (Rink), the Project Director (Paula FireMoon), Ramey Growing Thunder, the Director of the Fort Peck Tribes Language and Culture Program, the study statistician (Mike Anastario), Dr. Julie Baldwin, the study co-Investigator, and the study's research program manager (Genevieve Cox). The DSMB will: a) review the research protocol and plans for data and safety monitoring; b) evaluate study progress, including data quality, participant recruitment rates, retention rates, outcome and adverse experience data, and risk versus benefit profile; and c) review the protocols to protect the confidentiality of the study data and the results of monitoring.

The study's community advisory aboard is updated quarterly on the study progress. The Fort Peck Tribal Executive Board, the Fort Peck IRS, the MSU IRB, and MSU's Office of Research Compliance and MSU's Office of Sponsored Programs are updated once a year on the study. The DSMB committee also will annually review the project's Data and Safety Monitoring Plan regarding: a) Reassessment of the risks and benefits to study participants; b) Participant recruitment, accrual, and retention; c) Data quality and confidentiality; d) Consideration of external scientific or therapeutic developments with impact on the safety of participants or the ethics of the study; e) Any adverse events.

The research team will update the general Data and Safety Monitoring Plan as well as the research protocols as needed. Adverse events will be reported to the Tribes, the participating schools, and the IRBs on an annual basis. Serious adverse events will be reported immediately to these entities as well as NIH and the DSMB. A written report will follow within 3 days of the event. The written report will be in the format required by the Tribes, schools, and the IRBs, and will contain information regarding the date of the event, description of the event, assessment of cause, whether the event indicates an increased risk for current or future subjects, and whether changes to the informed consent are necessary.

# **SECTION 8: APPENDICES**

The Appendices includes the following documents:

- IRB Approvals
- •

Fort Peck Tribal Institutional Review Board For the Protection of Human Subjects

FWA00019355

Chair: Robert McAnally 406-768-8377

bmcassin.@gma il.com

om FORT PECI

Fort Peck Community College Box 398 Poplar, MT 59255 406-768-5555

Administrator:

Joy Toavs 406-768-5555 <u>itoavs@fpcc.edu</u>

#### **MEMORANDUM**

TO: Elizabeth Rink, PhD. MSW

FROM: Robert McAnally

Chair, Institutional Review Board for the Protection of Human Subjects

**DATE:** October 26, 2018

SUBJECT: Nen UnkUmbi/EdaHiYedo ("We Are Here Now")

The above proposal was reviewed on October 4, 2018 by the Fort Peck Tribal Institutional Review Board. This proposal is now approved for a period of one-year.

Please keep track of the number of subjects who participate in the study and of any unexpected or adverse consequences of the research. If there are any adverse consequences, please report them to the committee as soon as possible. If there are serious adverse consequences, please suspend the research until the situation has been reviewed by the Institutional Review Board.

Any changes in the human subjects' aspects of the research should be approved by the committee before they are implemented.

It is the investigator's responsibility to inform subjects about the risks and benefits of the research. Although the subject's signing of the consent form, documents this process, you, as the investigator should be sure that the subject understands it. Please remember that subjects should receive a copy of the consent form and that you should keep a signed copy for your records.

In one year, you will be sent a questionnaire asking for information about the progress of the research. The information that you provide will be used to determine whether the committee will give continuing approval for another year. If the research is still in progress in 5 years, a complete new application will be required.

The Fort Peck IRB requests that when you have a manuscript, thesis, or presentation prepared for public consumption, that you provide the Fort Peck IRB with an opportunity to review the document prior to publication and to make recommendations to ensure that the document appropriately respects the Fort Peck peoples.



# INSTITUTIONAL REVIEW BOARD

#### For the Protection of Human Subjects FWA 00000165

960 Technology Blvd. Room 127 c/ o Microbiology & Immunology Montana State University Bozeman, MT 59718 Telephone: 406-994-6783

FAX: 406-994-4303

E-mail: cherylj@montana.edu

Chair: Mark Quinn 406-994-4707 mquinn@montana.edu

Administrator:

Cheryl Johnson 406-994-4706 cherylj@montana.edu

#### **MEMORANDUM**

TO: Elizabeth Rink

FROM: Mark Quinn

Chair, Institutional R view Board for the Protection of Human Subjects

DATE: February 5, 2018

SUBJECT: "Nen Onk?umbi/Edahiyedo ("We Are Here Now'J - a Multi-level, Multi-component

sexual and Reproductive Health Intervention for American Indian Youth" [ER020518]

The above proposal was reviewed by expedited review by the Institutional Review Board. This proposal is now approved for a period of one-year.

Please keep track of the number of subjects who participate in the study and of any unexpected or adverse consequences of the research. If there are any adverse consequences, please report them to the committee as soon as possible. If there are serious adverse consequences, please suspend the research until the situation has been reviewed by the Institutional Review Board.

Any changes in the human subjects' aspects of the research should be approved by the committee before they are implemented.

It is the investigator's responsibility to inform subjects about the risks and benefits of the research. Although the subject's signing of the consent form, documents this process, you, as the investigator should be sure that the subject understands it. Please remember that subjects should receive a copy of the consent form and that you should keep a signed copy for your records.

In one year, you will be sent a questionnaire asking for information about the progress of the research. The information that you provide will be used to determine whether the committee will give continuing approval for another year. If the research is still in progress in 5 years, a complete new application will be required.

# Nen OnkUmbi/EdaHiYedo ("We Are Here Now") Informed Consent to Participate in Human Subjects Research with Montana State University in Partnership with Fort Peck Community College

#### What is this project about?

We Are Here Now is an intervention project with Fort Peck Community College and Montana State University. The purpose of this intervention is to teach youth at Fort Peck important things they need to know about sex so that they can stay healthy and not get a sexually transmitted disease, HIV, or Hepatitis C, and so that they can make healthy decisions about having children, getting pregnant, or getting someone pregnant. We Are Here Now teaches parents about how to speak with their child about sensitive topics related to sex. We Are Here Now also teaches Assiniboine and Sioux youth about their culture and traditional beliefs and practices about what it means to be a young Native person who will soon be an adult.

#### Why me?

You have been selected to participate in this focus group because you participated in *We Are Here Now.* You may choose to participate or not participate in this focus group at any time.

# What happens to me if I decide to participate?

If you decide to be in this focus group we will be asking you questions about what you liked and did not like about *We Are Here Now.* The focus group will be about 1 hour. We will ask you questions about what you thought was good about We Are Here Now and what you did not like so much. We will also ask you what you think we need to change to make the program better the next time we do the program here at Fort Peck. We will record the focus group and we will not keep track of who is saying what. This means that nothing you say will be associated with you. Your responses are anonymous. If you agree to participate in this focus group, you will receive a \$10 gift card that you can use here at Fort Peck.

#### What are the risks?

There may be very minimal risks to participating in the focus group. We are going to ask you questions about what you liked and did not like about *We Are Here Now*. Maybe you might feel uncomfortable sharing with us what you thought about the program. That is okay. It is important that we hear for you about what you liked and did not like about *We Are Here Now* so that we can make it better the next time we implement the program here. If there is something you would really like us to know and do not feel comfortable talking about it in the focus group you can contact Paula Firemoon at Fort Peck Community College and speak with her.

# What are the benefits?

The information gathered in this focus group will help the We Are Here Now's research team and members of the Fort Peck community to understand how to make this program better for young people on the reservation.

# Who gets access to information from this interview?

The research team has access to the data collected for this project. The *We Are Here Now* community advisory board will also have access to the data collected for this intervention. All responses in this focus group are confidential amongst the other people in the focus group. It is important that what we say in the focus group stays here. So that we respect what everyone has to say. In the transcripts created from the focus group recording none of the responses will be associated with your name. This means that your responses in the focus group transcripts are anonymous. Neither the research team nor the community advisory board will know who you are in the focus group transcripts.





# How am I informed about the results of the project, and when will they be released and presented to someone else?

We will publish the intervention results and make presentations on the results from *We Are Here Now.* Your identity will never appear in a publication or in print or be discussed at a presentation. In addition, you will have the opportunity to learn about the intervention results by contacting members of the research team, attending community meetings where we share the results of the project, and through local (Fort Peck Reservation) media.

#### Who is involved in We Are Here Now?

If you have any questions regarding this survey please contact:

Paula Firemoon, Fort Peck Community College - Email: PFiremoon@fpcc,edu; Phone: 406.768.6300

## Ramey Growing Thunder, Fort Peck Tribes Language and Culture Department

Email:rgrowingthunder@gm ail.com; Phone: 406.768-3520

Elizabeth Rink, Montana State University- Email: elizabeth.rink@montana.edu; Phone: 406.994.3833

#### **CONSENT STATEMENT**

focus group.

#### If the research participant is a minor:

Focus Group Administrator Signature:

If you are 18 years or younger and you agree to participate in this focus group, please read, complete, and sign the statement below. By signing this consent form you are giving your verbal and written consent to complete this focus group.

Minor: I have read the above and understand the discomfort, inconvenience, and risks associated with this

| I, | , agree to participate in this focus group. |
|---|---|
| Name of Minor | |
| Minor Participant Signature: | |
| Parent/Legal Guardian agreement for minor | <u>:</u> |
| If as a parent or guardian you <b>do want</b> your chi sign the statement below. | ild to participate in this focus group, please read, complete, and |
| Parent/Legal Guardian for Minor: I have read risks associated with this focus group. | I the above and understand the discomfort, inconvenience, and |
| I,, do | o agree to have my child participate in this focus group. |
| Name of Parent/Guardian: | Date: |
| Parent/Guardian Signature: | Date: |



Date:
## Nen OnkUmbi/EdaHiYedo ("We Are Here Now") Informed Consent to Participate in Human Subjects Research with Montana State University in Partnership with Fort Peck Community College

### What is this project about?

We Are Here Now is an intervention project with Fort Peck Community College and Montana State University. The purpose of this intervention is to teach youth at Fort Peck important things they need to know about sex so that they can stay healthy and not get a sexually transmitted disease, HIV, or Hepatitis C, and so that they can make healthy decisions about having children, getting pregnant, or getting someone pregnant. We Are Here Now teaches parents about how to speak with their child about sensitive topics related to sex. We Are Here Now also teaches Assiniboine and Sioux youth about their culture and traditional beliefs and practices about what it means to be a young Native person who will soon be an adult.

### Why me?

You have been selected to participate in this focus group because you participated in *Native Voices* which is part of a larger intervention called *We Are Here Now.* You may choose to participate or not participate in this focus group at any time.

### What happens to me if I decide to participate?

If you decide to be in this focus group we will be asking you questions about what you liked and did not like about *Native Voices*. The focus group will be about 1 hour. We will ask you questions about what you thought was good about *Native Voices* and what you did not like so much. We will also ask you what you think we need to change to make the program better the next time we do the program here at Fort Peck. We will record the focus group and we will not keep track of who is saying what. This means that nothing you say will be associated with you. Your responses are anonymous. If you agree to participate in this focus group, you will receive a \$20 gift card that you can use here at Fort Peck.

### What are the risks?

There may be very minimal risks to participating in the focus group. We are going to ask you questions about what you liked and did not like about *Native Voices*. Maybe you might feel uncomfortable sharing with us what you thought about the program. That is okay. It is important that we hear for you about what you liked and did not like about *Native Voices* so that we can make it better the next time we implement the program here. We will also ask you questions about what you may have changed about the what and how you speak with your child about sex or relationships as a result of participating in *Native Voices*. If there is something you would really like us to know and do not feel comfortable talking about it in the focus group you can contact Paula Firemoon at Fort Peck Community College and speak with her.

### What are the benefits?

The information gathered in this focus group will help the *We Are Here Now's* research team and members of the Fort Peck community to understand how to make this program better for young people and their parents and families on the reservation.



### Who gets access to information from this interview?

The research team has access to the data collected for this project. The *We Are Here Now* community advisory board will also have access to the data collected for this intervention. All responses in this focus group are confidential amongst the other people in the focus group. It is important that what we say in the focus group stays here. So that we respect what everyone has to say. In the transcripts created from the focus group recording none of the responses will be associated with your name. This means that your responses in the focus group transcripts are anonymous. Neither the research team nor the community advisory board will know who you are in the focus group transcripts.

### How am I informed about the results of the project, and when will they be released and presented to someone else?

We will publish the intervention results and make presentations on the results from *We Are Here Now.* Your identity will never appear in a publication or in print or be discussed at a presentation. In addition, you will have the opportunity to learn about the intervention results by contacting members of the research team, attending community meetings where we share the results of the project, and through local (Fort Peck Reservation) media.

### Who is involved in We Are Here Now?

If you have any questions regarding this focus group please contact:

### Paula Firemoon, Fort Peck Community College

Email: PFiremoon@fpcc,edu; Phone: 406.768.6300

### Ramey Growing Thunder, Fort Peck Tribes Language and Culture Department

Email:rgrowingthunder@gmail.com; Phone: 406.768-3520

### Elizabeth Rink, Montana State University

Email: elizabeth.rink@montana.edu; Phone: 406.994.3833



### **CONSENT STATEMENT**

| Parent/Legal Guardian: I have read the and risks associated with this focus group | above and understand the discomfort, inconvenience, |
|---|---|
| 1, | , <b>do agree</b> to participate in this focus group. |
| Name of Parent/Guardian: | |
| Parent/Guardian Signature- | Date: |
| Focus Group Administrator Signature: | |



### INSTITUTIONAL REVIEW BOARD





2155 Analysis Drive c/o Microbiology & Immunology Montana State University Bozeman, MT 59718 Telephone: 406,994-6783 FAX: 406-994-4303

E-mail: cherylj@montana.edu

Chair: Mark Quinn
406-994-4707
mquinn@montana.edu
Administrator:

Cheryl Johnson 406-994-4706 cherylj@montana.edu

### **MEMORANDUM**

TO: Elizabeth Rink, Genevieve Cox, Paula Firemoon, Mike Anastario

FROM: Mark Quinn

Chair, Institutional Review Board for the Protection of Human Subjects

DATE: October 3, 2018

**SUBJECT:** "Nen unk?umbi/Edahiyedo ("We Are Here Now'? - a Multi-level, Mu/ti-component

Sexual and Reproductive Health Intervention for American Indian Youth" [ER100318-

FC]

The above proposal was reviewed by the Institutional Review Board. This proposal is now approved for a period of one-year.

Please keep track of the number of subjects who participate in the study and of any unexpected or adverse consequences of the research. *If there are any adverse consequences, please report them to the committee within 3 calendar days.* If there are serious adverse consequences, please suspend the research until the situation has been reviewed by the Institutional Review Board.

Any changes in the human subjects' aspects of the research should be approved by the committee before they are implemented.

It is the investigator's responsibility to inform subjects about the risks and benefits of the research. Although the subject's signing of the consent form, documents this process, you, as the investigator should be sure that the subject understands it. Please remember that subjects should receive a copy of the consent form and that you should keep a signed copy for your records.

In one year, you will be sent a questionnaire asking for information about the progress of the research. The information that you provide will be used to determine whether the committee will give continuing approval for another year. If the research is still in progress in 5 years, a complete new application will be required.

## NenUnkUmbi/EdaHiYedo ("We Are Here Now") Waiver of Consent to Participate in Human Subjects Research with Montana State University in Partnership with Fort Peck Community College

We Are Here Now is an intervention project with Fort Peck Community College and Montana State University. NenUnkUmbi/EdaHiYedo ("We are Here Now," or NIE) derives from the Assiniboine (NenUnkUmbi) and Sioux (EdaHiYedo) names for their traditional coming-of-age ceremonies. The purpose of this program is to teach youth at Fort Peck important things they need to know about sex so that they can stay healthy and not get a sexually transmitted disease, HIV, or Hepatitis C, and so that they can make healthy decisions about having children, getting pregnant, or getting someone pregnant. We Are Here Now also includes tribal elders and leaders teaching Assiniboine and Sioux youth about their culture and traditional beliefs and practices about what it means to be a young Native person who will soon be an adult. In addition to working with youth, We Are Here Now also is offering education to parents/legal guardians about how to speak with their children about sensitive topics related to sex.

As part of N/E will be working with the Fort Peck Epi Team to evaluate the reproductive health services available to youth on the Fort Peck Indian Reservation. Members of the Montana State University and Fort Peck based research team will be attending Epi team meetings to assess the reproductive health services available for youth on the reservation. These meetings will include discussions of the barriers and facilitators of reproductive health and tracking any changes that the agency you work for makes as result of our discussions. The Montana State University and Fort Peck based research team will provide regular feedback to the Epi Team of the monitoring we are conducting related to the barriers and facilitators of reproductive health services for tribal youth.

Our discussions will be audiotaped and transcribed in order to conduct content analysis of the primary themes that emerge related to the barriers and facilitators of our discussions. There is no risk associated with your involvement in the discussions; and there is no cost or compensation to you for participation in our discussions.

If you have any questions regarding N/E please contact:

Paula FireMoon, Fort Peck Community College Email: PFiremoon@fpcc.edu; Phone: 406.768.6300

Elizabeth Rink, Montana State University

Email: elizabeth.rink@montana.edu: Phone: 406.994.3833

Mark Quinn, Montana State University Institutional Review Board Chair

Email: mguinn@montana.edu; Phone: 406.994. 4707

### CONSENT STATEMENT

| I have read the purpose of N/E and the role of the Epi Team in this study. | |
|---|---|
| I, | |
| assessing the barriers and facility | ators of reproductive health services of youth on the Fort Peck Indian |
| Reservation. | · |
| G· | D. 4 |
| Signature: | Date: |



## NenUnkUmbi/EdaHiYedo ("We Are HereNow") Informed Consent to Participate in Human Subjects Research with Montana State University in Partnership with Fort Peck Community College

### What is this project about?

We Are Here Now is an intervention project with Fort Peck Community College and Montana State University. The purpose of this intervention is to teach youth at Fort Peck important things they need to know about sex so that they can stay healthy and not get a sexually transmitted disease, HIV, or Hepatitis C, and so that they can make healthy decisions about having children, getting pregnant, or getting someone pregnant. We Are Here Now also teaches Assiniboine and Sioux youth about their culture and traditional beliefs and practices about what it means to be a young Native person who will soon be an adult.

### Why me?

You have been selected to participate in *We Are Here Now* because you are a young person at Fort Peck. You may choose to participate or not participate at any time.

### What happens to me if I decide to participate?

If you decide to be in *We Are Here Now,* you will participate in a survey that will take 50 to 60 minutes. You will be asked to complete this survey three more times during the next year so that we can keep track of any changes you may have in your beliefs and behaviors as a result of participating in *We Are Here Now.* You will be asked several questions about different topics related to sex, having children, and sexually transmitted diseases in order to learn about what you think about having children and what you know about sexually transmitted diseases. You will also be asked questions about your sexual behavior and experiences with drugs and alcohol. You will also be asked questions about your feelings and emotions and your traditional culture. It is important that you know that all of your responses on this survey are anonymous. This means that no one will know that it is you who answered these questions. Your responses will be kept track of in the computer that you are taking the survey on. Your name will be nowhere in the computer or on the survey. There is no cost to you if you agree to participate in this study. If you agree to participate in this survey, you will receive a \$10 gift card that you can use here at Fort Peck. Also by agreeing to participate in *We Are Here Now*, your parent/legal guardian is agreeing to participate in an educational program called *Native Voices*, and you are agreeing to be part of a cultural mentoring program with the Fort Peck Tribes' Language and Culture Department.

### What are the risks?

There may be minor risks to agreeing to participate in the survey. Some of the questions may make you feel uncomfortable, sad, or confused. You may choose to stop the survey at any time or decline to answer a particular question. The questions will be about your life experiences as they relate to sex, drug and alcohol use, having children, sexually transmitted diseases, your feelings and emotions, and your understanding of your traditional culture. A list of resources are provided in this consent form if you feel that you would like to speak with someone further about your life experiences. None of the things that you say on the survey will be connected to your name.

### What are the benefits?

The information gathered in this survey will help the intervention's research team and members of the Fort Peck community to understand what kind of impact your participation in *We Are Here Now* is having on your decisions to avoid getting a sexually transmitted disease and your decisions about having children when you feel you are ready. We would also like you to know that if you tell us about any abusive situation you are experiencing or have experienced, we will need to report that to the appropriate services here at Fort Peck so that you can receive assistance.

### Who gets access to information from this interview?

All responses on this survey will be confidential. Only one person, Paula FireMoon, will know that you participated. Your personal information such as your name, telephone number and address will be linked to a study identification number to track your participation in the study. Your personal information will only be kept in order to contact you to participate in the follow up data collection for this study. Your personal information will be kept in a locked file cabinet at the Fort Peck Community College Institutional Review Board administration office in Poplar. Neither Paula nor the rest of the research team, nor the community advisory

board, will know what your individual responses to the survey are. The data collected in this study will not be associated with your name. The research team and the community advisory board will have access to the data collected for this project with no identifying information on it that can be associated with your name.

### <u>How am I informed about the results of the project, and when will they be released and presented</u> to <u>someone else?</u>

We will publish the intervention results and make presentations on the results from *We Are Here Now.* Your identity will never appear in a publication or in print or be discussed at a presentation. In addition, you will have the opportunity to learn about the intervention results by contacting members of the research team, attending community meetings where we share the results of the project, and through local (Fort Peck Reservation) media.

### Who is involved in We Are Here Now?

If you have any questions regarding this survey please contact:

### Paula FireMoon, Fort Peck Community College

Email: PFiremoon@fpcc,edu; Phone: 406.768.6300

Elizabeth Rink, Montana State University

Email: elizabeth.rink@montana.edu; Phone: 406.994.3833

Mark Quinn, Montana State University Institutional Review Board Chair

Email: mguinn@montana.edu; Phone: 406.994. 4707

### **CONSENT STATEMENT**

### If the research <u>participant</u> is a minor:

If you are 18 years or younger and you agree to participate in this survey, please read, complete, and sign the statement below. By signing this consent form you are giving your verbal and written consent to complete this survey.

| survey. | connort, inconvenience, and risks associated with this |
|---|---|
| I,,agr | ee to participate in this survey. |
| Name of Minor | |
| Minor Participant Signature: | Date: |
| Parent/Legal Guardian agreement for Jnir 1 or: | |
| If as a parent or guardian you <b>do want</b> your child to the statement below. | participate in this survey, please read, complete, and sign |
| Parent/Legal Guardian for Minor: I have read the a risks associated with this survey. | above and understand the discomfort, inconvenience, and |
| Name of Parent/Guardian, do agr | •ee to have my child participate in this survey. |
| Parent/Guardian Signature: | Date: |
| Survey Administrator Signature: | Date: |



### NenUnkUmbi/EdaHiYedo ("We Are Here Now") Informed Consent to Participate in Human Subjects Research with Montana State University in Partnership with Fort Peck Community College

### What is this project about?

We Are Here Now is an intervention project with Fort Peck Community College and Montana State University. NenUnkUmbi/EdaHiYedo ("We are Here Now," or NIE) derives from the Assiniboine (NenUnkUmb1) and Sioux (EdaHiYedo) names for their traditional coming-of-age ceremonies. The purpose of this program is to teach youth at Fort Peck important things they need to know about sex so that they can stay healthy and not get a sexually transmitted disease, HIV, or Hepatitis C, and so that they can make healthy decisions about having children, getting pregnant, or getting someone pregnant. We Are Here Now also includes tribal elders and leaders teaching Assiniboine and Sioux youth about their culture and traditional beliefs and practices about what it means to be a young Native person who will soon be an adult. In addition to working with youth, We Are Here Now also is offering education to parents/legal guardians about how to speak with their children about sensitive topics related to sex.

### Why me?

You and your child have been invited to participate in *We Are Here Now* and to help gather information about the program and its effects. Your participation in this intervention is entirely voluntary. You can choose not to participate at any time. You and your child may withdraw from the intervention at any time without negative consequences. Your participation in *We Are Here Now* is your choice.

### What happens to me if I decide to participate?

If you agree to participate in *We Are Here Now,* you will be with other guardians or parents of young people who are participating in *We Are Here Now,* and you will learn about how to talk with your child about sex. *We Are Here Now* is a project that educates youth and their guardians/parents about sexual and reproductive health. As a participant in *We Are Here Now,* you will be talking with other guardians/parents about healthy sexual behaviors and about how to talk with your children about sex. You will be asked to complete a survey specifically for guardians/parents about how you talk to your child about sex and what kinds of things about sex you speak with them about. There is no cost to you if you agree to participate in this study. You will receive an incentive of \$20 for this first survey, and then \$10 each time you attend the four *Native Voices* sessions (at 2 of these sessions you will again fill out the survey). Finally, you will receive a \$25 incentive for completing the final survey after the end of the program.

### What are the risks?

Some of the questions may make you feel a bit uncomfortable. For example, we will ask you about what kinds of sexual topics you talk about with your child. A list of community resources is provided with this informed consent if you feel you would like to speak with someone further about feelings that may have been brought up as a result of your participation in this study.

### What are the benefits?

Through this program you will learn about ways to speak effectively with your child about sex and topics related to sexual health. The information gathered in this survey will help the intervention's research team and members of the Fort Peck community to understand what kind of impact your participation in *We Are Here Now* is having on your decisions to talk with your child about sensitive



topics related to sex.

### Who gets access to information from this interview?

All responses on this survey will be confidential. Only one person, Paula FireMoon, will know that you participated. Your personal information such as your name, telephone number and address will be linked to a study identification number to track your participation in the study. Your personal information will only be kept in order to contact you to participate in the follow up data collection for this study. Your personal information will be kept in a locked file cabinet at the Fort Peck Community College Institutional Review Board administration office in Poplar. Neither Paula nor the rest of the research team, nor the community advisory board, will know what your individual responses to the survey are. The data collected in this study will not be associated with your name. The research team and the community advisory board will have access to the data collected for this project with no identifying information on it that can be associated with your name.

### How am I informed about the results of the project, and when will they be released and presented to someone else?

We will publish the intervention results and make presentations on the results from *We Are Here Now.* Your identity will never appear in a publication or in print or be discussed at a presentation. In addition, you will have the opportunity to learn about the intervention results by contacting members of the research team, by attending community meetings where we share the results of the project, and through local (Fort Peck Reservation) media.

### Who is involved in We Are Here Now?

If you have any questions regarding this survey please contact:

### Paula FireMoon, Fort Peck Community College

Email: PFiremoon@fpcc.edu; Phone: 406.768.6300

### Elizabeth Rink, Montana State University

Email: elizabeth.rink@montana.edu; Phone: 406.994.3833

### Mark Quinn, Montana State University Institutional Review Board Chair

Email: mguinn@montana.edu; Phone: 406.994. 4707

### **CONSENT STATEMENT**

| Parent/Legal Guardian for Minor: I have read the above and understand the discomfort, inconvenience, and risks associated with this survey. | |
|---|---|
| I,<br>Name of Parent/Guardian | , do agree to participate in this survey. |
| Parent/Guardian Signature: | Date: |
| Survey Administrator Signature: | Date: |





### INSTITUTIONAL REVIEW BOARD

### For the Protection of Human Subjects FWA 00000165

96 0 T echn ology Blvd. Room 127 c/o Microb io logy & Immun ology Mont ana St ate University Bozeman, MT 597 18 Telephone: 406-99 4-678 3 FAX: 406-99 4-4303

E-mail: cherylj@montana.edu

Chair: Mark Quinn 406-994-4707

mquinn @montana .edu

Administrator:

Ch eryl Johnson 406-994-4706 che rylj@ montan a.edu

### **MEMORANDUM**

TO: Elizabeth Rink

FROM: Mark Quinn

Chair, Institutional Review Board for the Protection of Human Subjects

**DATE:** August 9, 2019

SUBJECT: "Nen Onk?umbi/Edahiyedo ("We Are Here Now'J - a Multi-level, Multi-component

sexual and Reproductive Health Intervention for American Indian Youth - Pilot

Study [ER020518]

This is to acknowledge receipt of the request dated August 8, 2019 for a minor modification to the above protocol. The request for the following modification is approved:

 Increase the incentive for parents to complete the final survey three months after finishing Native Voices.

## NenUnkUmbi/EdaHiYedo ("We Are Here Now") Informed Consent to Participate in Human Subjects Research with Montana State University in Partnership with Fort Peck Community College

### What is this project about?

We Are Here Now is an intervention project with Fort Peck Community College and Montana State University. NenUnkUmbi/EdaHiYedo ("We are Here Now," or NIE) derives from the Assiniboine (NenUnkUmb1) and Sioux (EdaHiYedo) names for their traditional coming-of-age ceremonies. The purpose of this program is to teach youth at Fort Peck important things they need to know about sex so that they can stay healthy and not get a sexually transmitted disease, HIV, or Hepatitis C, and so that they can make healthy decisions about having children, getting pregnant, or getting someone pregnant. We Are Here Now also includes tribal elders and leaders teaching Assiniboine and Sioux youth about their culture and traditional beliefs and practices about what it means to be a young Native person who will soon be an adult. In addition to working with youth, We Are Here Now also is offering education to parents/legal guardians about how to speak with their children about sensitive topics related to sex.

### Why me?

You and your child have been invited to participate in *We Are Here Now* and to help gather information about the program and its effects. Your participation in this intervention is entirely voluntary. You can choose not to participate at any time. You and your child may withdraw from the intervention at any time without negative consequences. Your participation in *We Are Here Now* is your choice.

### What happens to me if I decide to participate?

If you agree to participate in *We Are Here Now*, you will be with other guardians or parents of young people who are participating in *We Are Here Now*, and you will learn about how to talk with your child about sex. *We Are Here Now* is a project that educates youth and their guardians/parents about sexual and reproductive health. As a participant in *We Are Here Now*, you will be talking with other guardians/parents about healthy sexual behaviors and about how to talk with your children about sex. You will be asked to complete a survey specifically for guardians/parents about how you talk to your child about sex and what kinds of things about sex you speak with them about. There is no cost to you if you agree to participate in this study. You will receive an incentive of \$20 each time you attend the four *Native Voices* sessions. At 2 of these sessions you will fill out a survey. You will also receive a \$25 incentive for completing the final survey three months after finishing *Native Voices*.

### What are the risks?

Some of the questions may make you feel a bit uncomfortable. For example, we will ask you about what kinds of sexual topics you talk about with your child.

### What are the benefits?

Through this program you will learn about ways to speak effectively with your child about sex and topics related to sexual health. The information gathered in this survey will help the intervention's research team and members of the Fort Peck community to understand what kind of impact your participation in *We Are Here Now* is having on your decisions to talk with your child about sensitive topics related to sex.



### **MSU IRB**

### Who gets access to information from this interview?

All responses on this survey will be confidential. Only one person, Paula FireMoon, will know that you participated. Your personal information such as your name, telephone number and address will be linked to a study identification number to track your participation in the study. Your personal information will only be kept inorder to contact you to participate in the follow up data collection for this study. Your personal information will be kept in a locked file cabinet at theFort Peck Community College Institutional Review Board administration office in Poplar. NeitherPaula nor the rest of the research team, nor the community advisory board, will know what yourindividual responses to the survey are. The data collected in this study will not be associated with your name. The research team and the community advisory board will have access to the data collected for this project with no identifying information on it that can be associated with your name.

### <u>How am I informed about the results of the project, and when will they</u> be released and <u>presented to someone else?</u>

We will publish the intervention results and make presentations on the results from *We Are Here Now.* Your identity will never appear in a publication or in print or be discussed at a presentation. In addition, you will have the opportunity to learn about the intervention results by contacting members of the research team, by attending community meetings where we share

the results of the project, and through local (Fort Peck Reservation) media.

### Who is involved in We Are Here Now?

If you have any questions regarding this survey please contact:

### Paula FireMoon, Fort Peck Community College

Email: PFiremoon@fpcc,edu; Phone: 406.768.6300

### Elizabeth Rink, Montana State University

Email: elizabeth.rink@montana.edu; Phone: 406.994.3833

### Mark Quinn, Montana State University Institutional Review Board Chair

Email: mguinn@montana.edu: Phone: 406.994, 4707

### **CONSENT STATEMENT**

| Parent/Legal Guardian for Minor: I have read the above and understand the discomfort,inconvenience, and risks associated with this survey. | |
|---|---|
| I,<br>Name of Parent/Guardian | , <b>do agree</b> to participate in this survey. |
| Parent/Guardian Signature: | Date: |
| Survey Administrator Signature: | Date: |

**APPROVED** 

# MSU IRB o 8/o 9/2019 Date approved

### INSTITUTIONAL REVIEW BOARD





960 Tedmology Blvd. Room 127 c/o Microbiology & Imm unology Montana Srate University Bozeman, MT 597 18 Telephone: 406-994--6783 FAX: 406-994-4303

E-mail: cherylj@montana.edu

Chair: Mark Quinn 406-994-4707 mquinn@montana.edu

Administrator:

Cheryl .John so n 406-9 94-4706

cherylj@montanaedu

### **MEMORANDUM**

TO: Elizabeth Rink

FROM: Mark Quinn

Chair , Institutional Review Board for the Protection of Human Subjects

**DATE:** April 20, 2020

SUBJECT: "Nen Onk?umbi/Edahiyedo ("We Are Here Now'? - a Multi-level, Multi-component

Sexual and Reproductive Health Intervention for American Indian Youth-Pilot

Study" [ER020518]

This is to acknowledge receipt of the request dated April 20, 2020 for minor modifications to the above protocol. The request for the following modifications is approved:

- Protocol is being changed for parents to read and complete a parent educational packet of resources alongside one-on-one meetings with our Native implementors, rather than group educational sessions;
- Request to include Focus Groups focused on Fidelity, Acceptability, and Sustainability of
  the project implementation to be conducted in summer 2020. A total of 8 focus groups
  will be conducted including two focus groups with youth participants, two focus groups
  with parents of youth participants, 2 focus groups surrounding the cultural mentoring
  components of the intervention, and 2 focus groups with professionals involved in the
  intervention.

## NenUnkUmbi/EdaHiYedo ("We Are Here Now") Informed Consent to Participate in Human Subjects Research with Montana State University in Partnership with Fort Peck Community College

We Are Here Now is an intervention project with Fort Peck Community College and Montana State University. NenUnkUmbi/EdaHiYedo ("We are Here Now," or NIE) derives from the Assiniboine (NenUnkUmb1) and Sioux (EdaHiYedo) names for their traditional coming-of-age ceremonies. The purpose of this program is to teach youth at Fort Peck important things they need to know about sex so that they can stay healthy and not get a sexually transmitted disease, HIV, or Hepatitis C, and so that they can make healthy decisions about having children, getting pregnant, or getting someone pregnant. We Are Here Now also includes tribal elders and leaders teaching Assiniboine and Sioux youth about their culture and traditional beliefs and practices about what it means to be a young Native person who will soon be an adult. In addition to working with youth, We Are Here Now also is offering education to parents/legal guardians about how to speak with their children about sensitive topics related to sex.

You have been chosen to participate in a Focus Group to help us understand the value and effectiveness of *We Are Here Now* because you are involved in the intervention as a youth participant in the schools, as a parent of a participant, or as someone who has been helping to facilitate *We Are Here Now*. We would like to better understand your point of view on what has worked best so far with *We Are Here Now* and what might be improved. Specifically, we would like to understand what experiences and activities you have liked or did not like, what educational information you liked or did not like, and any recommendations you might have for improving *We Are Here Now*.

Our discussions will be audiotaped and transcribed. These transcriptions are anonymous and confidential, and we will ask all participants to maintain confidentiality of discussions. However, we cannot guarantee full confidentiality because we cannot guarantee that participants involved in this Focus Group will not share stories or discussions outside our group. However, in transcriptions, no names will be used. There is no risk associated with your involvement in the discussions; and there is no cost to you for your participation in our discussions. You will receive \$20 for your time.

We will publish the intervention results and make presentations on the results from *We Are Here Now.* Information from the project **will** also be posted on the U.S. website, https://ClinicalTrials.gov. Your identity will never appear in a publication or in print or be discussed at a presentation. In addition, you will have the opportunity to learn about the intervention results by contacting members of the research team, attending community meetings where we share the results of the project, and through your local community media.

If you have any questions regarding this Focus Group please contact:

Paula FireMoon, Fort Peck Community College

Email: PFiremoon@fpcc,edu; Phone: 406-768-6300

Olivia Johnson, Fort Peck Community College Email: OJohnson@fpcc.edu; Phone: 406-768-6300

Elizabeth Rink, Montana State University

Email: elizabeth.rink@montana.edu; Phone: 406-994-3833

Mark Quinn, Montana State University Institutional Review Board Chair

Email: mquinn@montana.edu; Phone: 406-994-4707



### **CONSENT STATEMENT:**

### If the research participant is a minor:

If you are 18 years or younger and you agree to participate in this focus group, please read, complete, and sign the statement below. By signing this consent form you are giving your verbal and written consent to complete this focus group.

| Minor: I have read the above and underst with this focus group. | and the discomfort, inconvenience, and risks associated |
|---|---|
| Name of Minor | , <b>agree</b> to participate in this focus group. |
| Minor Participant Signature: | Date: |
| Parent/Legal Guardian agreement for notified as a parent or guardian you do want you complete, and sign the statement below. | ur child to participate in this focus group, please read, |
| Parent/Legal Guardian for Minor: I have r inconvenience, and risks associated with the | ead the above and understand the discomfort, his focus group. |
| I,group. | _ , <b>do agree</b> to have my child participate in this focus |
| Name of Parent/Guardian: | |
| Parent/Guardian Signature: | Date: |
| Focus Group Administrator Signature: | Date |





### INSTITUTIONAL REVIEW BOARD

### For the Protection of Human Subjects FWA 00000165

960 Technology Blvd. Room 127 c/o Microbiology & Immunology Montana State University Bozeman, MT 59718 Telephone: 406-994-6783

FAX: 406-994-4303

E-mail: cherylj@montana.edu

Chair: Mark Quinn 406-994-4707 mquinn@montana.edu

Administrator:

Cheryl Johnson 406-994-4706 cherylj@montana.edu

### **MEMORANDUM**

**TO:** Elizabeth Rink, Genevieve Cox, Paula Firemoon, Mike Anastario

FROM: Mark Quinn

Chair, Institutional Review Board for the Protection of Human Subjects

DATE: September 30, 2020

SUBJECT: "Nen Onk?umbi/Edahiyedo ("We Are Here Now'J - a Multi-level, Multi-component

sexual and Reproductive Health Intervention for American Indian Youth

[ER100318-FCJ

This is to acknowledge receipt of the request dated September 29, 2020 for minor modifications to the above protocol. The request for the following modifications is approved:

- Will conduct a within scope data collection of the impact of COVID-19 on their primary outcome variables and the study's stepped wedge design.
- Will be collecting data from a subset of the study participants. The data collection will include: a chain referral network survey and in-depth interviews.
- Submitted the consent forms and data collection instruments for the two methods of data collection.

## Nen OnkUmbi/EdaHiYedo ("We Are Here Now") Informed Consent to Participate in Human Subjects Research with Montana State University in Partnership with Fort Peck Community College

### What is this project about?

We Are Here Now is an intervention project with Fort Peck Community College and Montana State University. The purpose of this intervention is to teach youth at Fort Peck important things they need to know about sex so that they can stay healthy and not get a sexually transmitted disease, HIV, or Hepatitis C, and so that they can make healthy decisions about having children, getting pregnant, or getting someone pregnant. We Are Here Now also teaches Assiniboine and Sioux youth about their culture and traditional beliefs and practices about what it means to be a young Native person who will soon be an adult. For the purpose of this interview we would like to learn from you how COVID-19 and the sheltering in place orders have impacted your behaviors.

### Why me?

You have been selected to participate in this survey because you participate in the original data collection for *We Are Here Now* in Spring 2019. You may choose to participate or not participate at any time.

### What happens to me if I decide to participate?

If you decide to participate in this interview we will ask you a series of questions about how COVID-19 and the sheltering in place orders impacted some of your behaviors and your feelings as well as your friends and family. The interview that will take about 45 minutes. You will be asked several questions about different topics related to sex, your feelings and what you did during the sheltering in place orders from March 2020 to May 2020 and then, you will also be asked questions about what has happened in your life more recently. It is important that you know that all of your responses are anonymous. his means that no one will know that it is you who answered these questions. We will audio-tape and transcribe your interview. Your name will be nowhere in the transcript of your interview. If you agree to participate in this interview, you will receive a \$10 gift card that you can use here at Fort Peck. If you would like a copy of your interview please let us know and we will make sure that you receive a copy of the transcript from our discussion.

### What are the risks?

There may be minor risks to agreeing to participate in the interview. Some of the questions may make you feel uncomfortable, sad, or confused. You may choose to stop the interview at any time or decline to answer a particular question. The questions will be about your perceptions of what was going on in your life during the sheltering place orders last Spring, from March 2020 to May 2020 and then now. None of the things that you say in the interview will be connected to your name. Although there are minor risks to agreeing to participate in the interview, if you feel sad or lonely or anxious you can talk to the person here today who is giving you this survey about how you are feeling and they are help you. You are also contact the names on this informed consent and we can assist you with finding someone to help you with how you are feeling.

### What are the benefits?

The information gathered in this interview will help us understand how COVID-19 has impacted young people at Fort Peck so that we can help the Tribes, schools and other resources at Fort Peck you and your family now and in the future. We would also like you to know that if you tell us about any abusive situation you are experiencing or have experienced, we will need to report that to the appropriate services here at Fort Peck so that you can receive assistance.

### Who gets access to information from this interview?

The research team has access to the data collected for this project. The *We Are Here Now* community advisory board will also have access to the data collected for this intervention. All responses on this survey will be anonymous. Neither the research team nor the community advisory board will know who you are and what your responses to the survey are.

### How am I informed about the results of the project, and when will they be released and presented to someone else?

We will publish the results and make presentations on the results from this survey. Your identity will never appear in a publication or in print or be discussed at a presentation. In addition, you will have the opportunity to learn about the intervention results by contacting members of the research team, attending



community meetings where we share the results of the project, and through local (Fort Peck Reservation) media.

### Who is involved in We Are Here Now?

If you have any questions regarding this survey please contact:

### Paula FireMoon, Fort Peck Community College

Email: PFiremoon@fpcc,edu; Phone: 406.768.6300

### Bob McAnnally, Fort Peck Institutional Review Board Chair

Email: bmcassin@gmail.co; Phone: 406.768.6300.

### **Elizabeth Rink, Montana State University**

Email: elizabeth.rink@montana.edu; Phone: 406.994.3833

### Mark Quinn, Montana State University Institutional Review Board Chair

Email: MQuinn@montana.edu; Phone: 406-994-4707

### **CONSENT STATEMENT**

### If the research participant is a minor:

If you are 18 years or younger and you agree to participate in this survey, please read, complete, and sign the statement below. By signing this consent form you are giving your verbal and written consent to complete this survey.

| <u>Minor:</u> I have read the above and understand th survey. | e discomfort, inconvenience, and risks associated with this |
|---|---|
| I, | agree to participate in this survey. |
| Name of Minor | |
| Minor Participant Signature: | Date: |
| Parent/Legal Guardian agreement for minor: | |
| If <b>as a</b> parent or guardian you <b>do want</b> your child sign the statement below. | d to participate in this survey, please read, complete, and |
| Parent/Legal Guardian for Minor: I have read tand risks associated with this survey. | the above and understand the discomfort, inconvenience, |
| l, <u>d</u> o a | gree to have my child participate in this survey. |
| Name of Parent/Guardian | |
| Parent/Guardian Signature: | Date: |
| Survey Administrator Signature: | Date |



## Nen UnkUmbi/EdaHiYedo ("We Are Here Now") Informed Consent to Participate in Human Subjects Research with Montana State University in Partnership with Fort Peck Community College

### What is this project about?

We Are Here Now is an intervention project with Fort Peck Community College and Montana State University. The purpose of this intervention is to teach youth at Fort Peck important things they need to know about sex so that they can stay healthy and not get a sexually transmitted disease, HIV, or Hepatitis C, and so that they can make healthy decisions about having children, getting pregnant, or getting someone pregnant. We Are Here Now also teaches Assiniboine and Sioux youth about their culture and traditional beliefs and practices about what it means to be a young Native person who will soon be an adult. For the purpose of this survey we would like to learn from you how COVID-19 and the sheltering in place orders have impacted your behaviors.

### Why me?

You have been selected to participate in this survey because you participate in the original data collection for *We Are Here Now* in Spring 2019. You may choose to participate or not participate at any time.

### What happens to me if I decide to participate?

If you decide to participate in this survey we will ask you a series of questions about how COVID-19 and the sheltering in place orders impacted some of your behaviors and your feelings. The survey that will take about 45 minutes. You will be asked several questions about different topics related to sex, your feelings and what you did during the sheltering in place orders from March 2020 to May 2020 and then, you will also be asked questions about what you have done over the past month. It is important that you know that all of your responses on this survey are anonymous. This means that no one will know that it is you who answered these questions. Your responses will be kept track of in the computer that you are taking the survey on. Your name will be nowhere in the computer or on the survey. If you agree to participate in this survey, you will receive a \$10 gift card that you can use here at Fort Peck. Once you have finished the survey, you will be given a coupon to give to 2 or 3 of the people that you socialize with so that they can participate in the survey .lso. For each person you tell to participate in the survey you will receive another \$10 gift card. You may also sk you to participate in an interview to talk with us further about what you think is important for us to know about how COVID 19 influenced your life.

### What are the risks?

There may be minor risks to agreeing to participate in the survey. Some of the questions may make you feel uncomfortable, sad, or confused. You may choose to stop the survey at any time or decline to answer a particular question. The questions will be about sex, drug and alcohol use, your feelings and emotions, and how your life has been impacted by COVID-19 and the sheltering in place orders. None of the things that you say on the survey will be connected to your name. Although there are minor risks to agreeing to participate in the survey, if you feel sad or lonely or anxious you can talk to the person here today who is giving you this survey about how you are feeling and they are help you. You are also contact the names on this informed consent and we can assist you with finding someone to help you with how you are feeling.

### What are the benefits?

The information gathered in this survey will help us understand how COVID-19 has impacted young people at Fort Peck so that we can help the Tribes, schools and other resources at Fort Peck you and your family now and in the future. We would also like you to know that if you tell us about any abusive situation you are experiencing or have experienced, we will need to report that to the appropriate services here at Fort Peck so that you can receive assistance.

### Who gets access to information from this interview?

The research team has access to the data collected for this project. The *We Are Here Now* community advisory board will also have access to the data collected for this intervention. All responses on this survey will be anonymous. Neither the research team nor the community advisory board will know who you are and what your responses to the survey are.



### INSTITUTIONAL REVIEW BOARD

### How am I informed about the results of the project, and when will they be released and presented to someone else?

We will publish the results and make presentations on the results from this survey. Your identity will never appear in a publication or in print or be discussed at a presentation. In addition, you will have the opportunity tolearn about the intervention results by contacting members of the research team, attending community meetings where we share the results of the project, and through local (Fort Peck Reservation) media.

### Who is involved in We Are Here Now?

If you have any questions regarding this survey please contact:

### Paula FireMoon, Fort Peck Community College

Email: PFiremoon@fpcc,edu; Phone: 406.768.6300

### Bob McAnnally, Fort Peck Institutional Review Board Chair

Email: bmcassin@gmail.co; Phone: 406.768.6300.

### Elizabeth Rink, Montana State University

Email: elizabeth.rink@montana.edu; Phone: 406.994.3833

### Mark Quinn, Montana State University Institutional Review Board Chair

Email: MQuinn@montana.edu; Phone: 406-994-4707

### **CONSENT STATEMENT**

### If the research participant is a minor:

If you are 18 years or younger and you agree to participate in this survey, please read, complete, and sign the statement below. By signing this consent form you are giving your verbal and written consent to complete this survey.

Minor: I have read the above and understand the discomfort, inconvenience, and risks associated with this

| survey. | |
|---|---|
| I, | , <b>agree</b> to participate in this survey. |
| Minor Participant Signature: | Date:· |
| Parent/Legal Guardian agreement for minor: | <u>.</u> |
| If as a parent or guardian you <b>do want</b> your chil statement below. | ld to participate in this survey, please read, complete, and signthe |
| Parent/Legal Guardian for Minor: I have read risks associated with this survey. | the above and understand the discomfort, inconvenience, and |
| I,, do | agree to have my child participate in this survey. |
| Parent/Guardian Signature: | Date: |
| Survey Administrator Signature | Date |

Supplemental Funding Request In-Depth Interview Guide 9-28-20

### Nen ŨnkUmbi/EdaHiYedo ("We Are Here Now")

# Informed Consent to Participate in Human Subjects Research with Montana State University in Partnership with Fort Peck Community College

### What is this project about?

We Are Here Now is an intervention project with Fort Peck Community College and Montana State University. The purpose of this intervention is to teach youth at Fort Peck important things they need to know about sex so that they can stay healthy and not get a sexually transmitted disease, HIV, or Hepatitis C, and so that they can make healthy decisions about having children, getting pregnant, or getting someonepregnant. We Are Here Now also teaches Assiniboine and Sioux youth about their culture and traditional beliefs and practices about what it means to be a young Native person who will soon be an adult. For the purpose of this interview we would like to learn from you how the COVID-19 pandemic over the past year impacted your behaviors.

### Why me?

You have been selected to participate in this interview because you participate in the original data collection for *We Are Here Now* in Spring 2019. You may choose to participate or not participate at any time.

### What happens to me if I decide to participate?

If you decide to participate in this interview, we will ask you a series of questions about how COVID-19 and the sheltering in place orders impacted some of your behaviors and your feelings as well as your friends and family. The interview that will take about 45 minutes. You will be asked several questions about different topics related to sex, your feelings and what you did during COVID-19 pandemic when you could not go to school because your school was shut down, you will also be asked questions about what has happened in your life more recently. It is important that you know that all of your responses are anonymous. This means that no one will know that it is you who answered these questions. We will audiotape and transcribe your interview. Your name will be nowhere in the transcript of your interview. If you agree to participate in this interview, you will receive a \$10 gift card that you can use here at Fort Peck. If you would like a copy of your interview please let us know and we will make sure that you receive a copy of the transcript from our discussion.

### What are the risks?

There may be minor risks to agreeing to participate in the interview. Some of the questions may make you feel uncomfortable, sad, or confused. You may choose to stop the interview at any time or decline to answera particular question. The questions will be about your perceptions of what was going on in your life over thepast year during the COVID-19 pandemic. None of the things that you say in the interview will be connected to your name. Although there are minor risks to agreeing to participate in the interview, if you feel sad or lonely or anxious you can talk to the person here today who is giving you this interview about how you are feeling, and they are help you. You are also contact the names on this informed consent and we can assist you with finding someone to help you with how you are feeling.

### What are the benefits?

The information gathered in this interview will help us understand how the COVID-19 pandemic has impacted young people at Fort Peck so that we can help the Tribes, schools and other resources at Fort Peck you and your family now and in the future. We would also like you to know that if you tell us about anyabusive situation you are experiencing or have experienced, we will need to report that to the appropriate services here at Fort Peck so that you can receive assistance.

### Who gets access to information from this interview?

The research team has access to the data collected for this project. The *We Are Here Now* community advisory board will also have access to the data collected for this intervention. All responses in this interview are anonymous. Neither the research team nor the community advisory board will know who you're and what your responses to the interview are.

### How am I informed about the results of the project, and when will they be released and presented to someone else?

We will publish the results and make presentations on the results from the interviews that we conduct to agencies at Fort Peck and the Fort Peck Tribal Executive Board. Your identity will never appear in a publication or in print or be discussed at a presentation. In addition, you will have the opportunity to learn

Supplemental Funding Request In-Depth Interview Guide

9-28-20

about the intervention results by contacting members of the research team, attending community meetingswhere we share the results of the project, and through local (Fort Peck Reservation) media.

### Who is involved in We Are Here Now?

If you have any questions regarding this interview, please contact:

### Paula FireMoon, Fort Peck Community College

Email: PFiremoon@fpcc,edu; Phone: 406.768.6300

### **Bob McAnnally, Fort Peck Institutional Review Board Chair**

Email: bmcassin@gmail.co; Phone: 406.768.6300.

### **Elizabeth Rink, Montana State University**

Email: elizabeth.rink@montana.edu; Phone: 406.994.3833

### Mark Quinn, Montana State University Institutional Review Board Chair

Email: MQuinn@montana.edu; Phone: 406-994-4707

### **CONSENT STATEMENT**

### If the research participant is a minor:

If you are 18 years or younger and you agree to participate in this interview, please read, complete, and sign the statement below. By signing this consent form, you are giving your verbal and written consent tocomplete this interview.

| <u>Minor</u> : I have read the above and und interview. | derstand the discomfort, inconvenience, and risks associated with this |
|---|---|
| I,<br>Name of Minor | , <b>agree</b> to participate in this interview. |
| Minor Participant Signature: | Date: |
| <u>Parent/Legal Guardian a</u> | greement for minor: |
| If as a parent or legal guardian you <b>d</b> ecomplete, and sign the statement below | owant your child to participate in this interview, please read, ow. |
| Parent/Legal Guardian for Minor: and risks associated with this interv | I have read the above and understand the discomfort, inconvenience, iew. |
| l, | , <b>do agree</b> to have my child participate in this interview. |
| Name of Parent/Legal Guardian | |
| Parent/Legal Guardian Signature:_ | Date: |
| Interview Administrator Signature:_ | Date |

Supplemental Funding Request In-Depth Interview Guide 9-28-20

### ClinicalTrials. gov PRS

### Protocol Registration and Results System

ClinicalTrials.gov Protocol Registration and Results System (PRS) Receipt Release Date: October 1, 2018

ClinicalTrials.gov ID: NCT03694418

### Study Identification

Unique Protocol ID: R01MD012761

Brief Title: We Are Here Now: a Multi-level, Multicomponent Sexual and Reproductive

Health Intervention for American Indian Youth (NE)

Official Title: We Are Here Now: a Multi-level, Multicomponent Sexual and Reproductive

Health Intervention for American Indian Youth

Secondary IDs:

### Study Status

Record Verification: October 2018

Overall Status: Not yet recruiting

Study Start: March 1, 2019 [Anticipated]

Primary Completion: November 30, 2021 [Anticipated]

Study Completion: November 30, 2022 [Anticipated]

### Sponsor/Collaborators

Sponsor: Montana State University

Responsible Party: Principal Investigator

Investigator: Elizabeth Rink [erink]
Official Title: Associate Professor
Affiliation: Montana State University

Collaborators:

### Oversight

U.S. FDA-regulated Drug: No

U.S. FDA-regulated Device: No

U.S. FDA IND/IDE: No

Human Subjects Review: Board Status: Pending

Board Name: Montana State University IRB

Board Affiliation: Mark Quinn

Phone: 994-4707

Email: mquinn@montana.edu

Address:

960 Technology Blvd. Room 127

### Montana State University Bozeman, Montana 59718

Data Monitoring: Yes

FDA Regulated Intervention: No

### Study Description

Brief Summary: N/E is a community-based participatory research (CBPR) multi-level, multicomponent sexual and reproductive health (SRH) intervention, constructed on Ecological Systems Theory. N/E is based on Fort Peck tribal members' desire to implement a holistic SRH intervention for Al youth. N/E includes: 1) A schoolbased SRH curriculum called Native Stand, designed to address individuallevel factors that lead to sexual risk behaviors; 2) a family-level curriculum called Native Voices, tailored to increase communication between adult family members and youth about SRH topics; 3) a cultural mentoring component at the community level that pairs Al youth with adults and elders to discuss traditional Al beliefs and practices about SRH; and 4) a mobilizing strategy to activate a multi-sectoral network of youth-servicing organizations at the systems level in Fort Peck to coordinate SRH services for Al youth. The overarching aim of this proposal is to refine, tailor, and finalize the components of N/E and evaluate its efficacy. We will use a cluster-randomized stepped-wedge design (SWD), in which 5 schools that Al youth from Fort Peck attend are the clusters to be randomized into the intervention 1 at a time, with all schools eventually being randomized to the intervention. The 5 schools are located in separate communities, mitigating the potential for cross-contamination. N/E is a 5-year study involving 456 15- to 18-year-old Al youth.

Detailed Description: N/E is a community-based participatory research (CBPR) multi-level, multicomponent sexual and reproductive health (SRH) intervention, constructed on Ecological Systems Theory. N/E is based on Fort Peck tribal members' desire to implement a holistic SRH intervention for Al youth. N/E includes: 1) A schoolbased SRH curriculum called Native Stand, designed to address individuallevel factors that lead to sexual risk behaviors; 2) a family-level curriculum called Native Voices, tailored to increase communication between adult family members and youth about SRH topics; 3) a cultural mentoring component at the community level that pairs Al youth with adults and elders to discuss traditional Al beliefs and practices about SRH; and 4) a mobilizing strategy to activate a multi-sectoral network of youth-servicing organizations at the systems level in Fort Peck to coordinate SRH services for Al youth. The overarching aim of this proposal is to refine, tailor, and finalize the components of N/E and evaluate its efficacy. We will use a cluster-randomized stepped-wedge design (SWD), in which 5 schools that Al youth from Fort Peck attend are the clusters to be randomized into the intervention 1 at a time, with all schools eventually being randomized to the intervention. The 5 schools are located in separate communities, mitigating the potential for cross-contamination. N/E is a 5-year study involving 456 15- to 18-year-old Al youth.

### Our specific aims are:

AIM 1: Refine, tailor, and finalize the components of N/E. Our community advisory board and the Fort Peck-based and MSU-based research team will design culturally appropriate adaptations for N/E's 4 levels during the first year of the study, based on the analysis of our recently completed qualitative and quantitative research (focus groups, interviews, and surveys), as well as discussions with elders and community stakeholders.

AIM 2: Test the efficacy of N/E for 15- to 18-year-old Al youth. Our hypotheses are:

H1: Al youth who participate in N/E will demonstrate increased condom use at 3, 9, and 12 months. (12 months will be used in the Primary Outcome analysis; 3 and 9 months will be used in the Secondary Outcomes analysis.) H2: Al youth who participate in N/E will demonstrate increased use of other birth control at 3, 9, and 12 months. They also will demonstrate a decrease in sexual risk behaviors as measured by reduced number of sex partners, delayed onset of sexual intercourse, and decreased substance use during sex, at 3, 9, and 12 months. (Secondary Outcomes) H3: N/E parents/legal guardians and youth will demonstrate significantly increased communication about topics related to SRH at 3, 9, and 12 months. Al youth who participate in the cultural mentoring program will demonstrate significantly increased understanding of cultural values related to traditional Al beliefs regarding SRH at 3, 9, and 12 months. And Al youth who participate in N/E will report significantly increased use of SRH services at 3, 9, and 12 months as a result of improved coordination among education, health care, and social service agencies on the Fort Peck Reservation. (Tertiary Outcomes) AIM 3: Evaluate the fidelity and acceptability of N/E. N/E's fidelity and acceptability will be evaluated using qualitative methods, including focus groups, activity logs, and staff field notes and meetings.

### Conditions

Conditions: Reproductive Behavior

Sexual Behavior

Keywords:

### Study Design

Study Type: Interventional

Primary Purpose: Prevention

Study Phase: N/A

Interventional Study Model: Sequential Assignment

Stepped Wedge Design

Number of Arms: 3

Masking: None (Open Label)

Allocation: Randomized

Enrollment: 1008 [Anticipated]

#### Arms and Interventions

#### Cluster 1

Cluster 1 is 1 school on the Fort Peck Reservation that will be randomized into the intervention in 2019. Cluster 1 will receive all four levels of the intervention including: 1) A school-based SRH curriculum called Native Stand, designed to address individual-level factors that lead to sexual risk behaviors; 2) a family-level curriculum called Native Voices, tailored to increase communication between adult family members and youth about SRH topics; 3) a cultural mentoring component at the community level that

Arms

### **Assigned Interventions**

Behavioral: We are here now: a multi-level, multi-component sexual and reproductive health intervention for American Indian youth

N/E will be implemented simultaneously over the 9-month school year. Components include: 1) Individual Level- Native Stand 2) Family Level - Native Voices; 3) Community Level - Cultural mentoring program; and 4) Systems Level. The fourth level of N/E mobilizes the existing Epi Team to enhance the coordination and implementation of SRH services at Fort Peck.

| Arms | Assigned Interventions |
|---|---|
| pairs Al youth with adults and elders to discuss traditional Al beliefs and practices about SRH; and 4) a mobilizing strategy to activate a multi-sectoral network of youth-servicing organizations at the systems level in Fort Peck to coordinate SRH services for Al youth. | |
| Cluster 2 Cluster 2 includes 2 schools on the Fort Peck Reservation that will be randomized in the intervention in 2019-2020. Cluster 2 will receive all four levels of the intervention including: 1) A school-based SRH curriculum called Native Stand, designed to address individual-level factors that lead to sexual risk behaviors; 2) a family-level curriculum called Native Voices, tailored to increase communication between adult family members and youth about SRH topics; 3) a cultural mentoring component at the community level that pairs Al youth with adults and elders to discuss traditional Al beliefs and practices about SRH; and 4) a mobilizing strategy to activate a multisectoral network of youth-servicing organizations at the systems level in Fort Peck to coordinate SRH services for Al youth. | Behavioral: We are here now: a multi-level, multi-component sexual and reproductive health intervention for American Indian youth N/E will be implemented simultaneously over the 9-month school year. Components include: 1) Individual Level- Native Stand 2) Family Level - Native Voices; 3) Community Level - Cultural mentoring program; and 4) Systems Level. The fourth level of N/E mobilizes the existing Epi Team to enhance the coordination and implementation of SRH services at Fort Peck. |
| Cluster 3 Cluster 3 are the remaining 2 schools on the Fort Peck reservation that will be randomized into the intervention in 2020-2021. Cluster 3 will receive all four levels of the intervention including: 1) A school- based SRH curriculum called Native Stand, designed to address individual-level factors that lead to sexual risk behaviors; 2) a family-level curriculum called Native Voices, tailored to increase communication between adult family members and youth about SRH topics; 3) a cultural mentoring component at the community level that pairs Al youth with adults and elders to discuss traditional Al beliefs and practices about SRH; and 4) a mobilizing strategy to activate a multi-sectoral network of youth-servicing organizations at the systems level in Fort Peck to coordinate SRH | Behavioral: We are here now: a multi-level, multi-component sexual and reproductive health intervention for American Indian youth N/E will be implemented simultaneously over the 9-month school year. Components include: 1) Individual Level- Native Stand 2) Family Level - Native Voices; 3) Community Level - Cultural mentoring program; and 4) Systems Level. The fourth level of N/E mobilizes the existing Epi Team to enhance the coordination and implementation of SRH services at Fort Peck. |

### **Outcome Measures**

### **Primary Outcome Measure:**

services for Al youth.

Change in condom use during sexual intercourse at 3 months, 9 months and 12 months
 Change in condom use during sexual intercourse will be measured as proportion of condom use during sexual
 intercourse will be measured using 2 items (number of times condom used relative to number of times had sexual
 intercourse).

[Time Frame: 3 months, 9 months and 12 months]

### Secondary Outcome Measure:

2. Change in delayed onset of sexual intercourse at 3 months, 9 months and 12 months

Changes in delayed onset of sexual intercourse will be measured intercourse with 2 items (ever had sexual intercourse and age at first sexual intercourse)

[Time Frame: 3 months, 9 months and 12 months]

3. Change in decreased number of sex partners at 3 months, 9 months and 12 months

Change in decreased number of sex partners will be measured by 2 items ( lifetime of sex partners and the number of sex partners in the past month)

[Time Frame: 3 months, 9 months and 12 months]

4. Change in frequency of sexual intercourse at 3 months, 9 months and 12 months Change in frequency of sexual intercourse will be measured with 1 time (frequency of sexual intercourse in the past month)

[Time Frame: 3 months, 9 months and 12 months]

Change in number of pregnancies at 3 months, 9 months and 12 months
 Change in number of pregnancies will be measure with 1 item (number of pregnancies)

[Time Frame: 3 months, 9 months and 12 months]

6. Change in increased use of birth control during sexual intercourse at 3 months, 9 months and 12 months
Change in the increased use of birth control during sexual intercourse will be measured with 3 items (type of birth control used and number of times birth control was sued during sexual intercourse)

[Time Frame: 3 months, 9 months and 12 months]

7. Change in decreased alcohol/drug use concurrently sexual intercourse at 3 months, 9 months and 12 months Change in decreased alcohol/drugs used concurrently with sexual intercourse will be measured with 1 item (substance use with sexual intercourse)

[Time Frame: 3 months, 9 months and 12 months]

### Other Pre-specified Outcome Measures:

8. Change in increased parenUlegal guardian-child communication about sexual and reproductive health topics at 3 months, 9 months and 12 months

Change in increased parenUlegal-child communication about sexual and reproductive health topics will be measured using a 24 item Likert scale, higher score = higher communication

[Time Frame: 3 months, 9 months and 12 months]

9. Change in increased usage of sexual and reproductive health services at 3 months, 9 months and 12 months
Change in increased usage of sexual and reproductive health services will be measured with 9 items (frequency, type
and follow up of sexual and reproductive health services used)

[Time Frame: 3 months, 9 months and 12 months]

### Eligibility

Minimum Age: 15 Years

Maximum Age: 18 Years

Sex: All

Gender Based: No Accepts Healthy Volunteers: No

Criteria: Inclusion Criteria:

- 15 to 18 years old
- a registered member of a federally recognized tribe or an associate tribal member
- a resident of Fort Peck with a parenUlegal guardian. Exclusion criteria are minimal due to the CAB's value of inclusion in the intervention.
- For inclusion in the systems-level component of the intervention, only those staff members who sit on the Epi Team as representatives of their respective agencies are eligible.

### **Exclusion Criteria:**

- · not meeting the aforementioned inclusion criteria
- having a medically identified physical or cognitive impairment that would impede
  their understanding of and participation in the educational content and activities of
  Native Stand, Native Voices, and the cultural mentoring program.

### Contacts/Locations

Central Contact Person: Elizabeth Rink, PhD

Telephone: 406-994-3833

Email: elizabeth.rink@montana.edu

Central Contact Backup: Genevieve Cox, PhD

Telephone: 406-994-4622

Email: genevieve.cox@motnana.edu

Study Officials:

Locations: United States, Montana Montana State University

Bozeman, Montana, United States, 59715

Contact: Elizabeth Rink, PhD 406-994-3833 elizabeth.rink@montana.edu

Contact: Genevieve Cox, PhD 406-994-4622 genevieve.cox@montana.edu Sub-Investigator: Paula Brien-Firemoon

Fort PeckCommunity College

Poplar, Montana, United States, 59255

Contact: Paula Brien-FireMoon, MA 406-768-7653 PFiremoon@fpcc.edu

### **IPDSharing**

Plan to Share IPD: No

There is no plan to have an IPD sharing plan at this point in time.

### References

Citations:

Links:

Available !PD/Information:

U.S. National Library of Medicine | U.S. National Institutes of Health | U.S. Department of Health & Human Services

RPPR FINAL

### A COVER PAGE

| Project Title: We are here now - a multi-level, multi-component | t sexual and reproductive health intervention for American Indian youth |
|---|---|
| <b>Grant Number:</b> 5R01MD012761-02 | Project/Grant Period: 04/01/2018 - 11/30/2022 |
| Reporting Period: 04/01/2018 - 11/30/2018 | Requested Budget Period: 12/01/2018 -11/30/2019 |
| Report Term Frequency: Annual | Date Submitted: 10/03/2018 |
| Program Director/Principal Investigator Information: | Recipient Organization: |
| ELIZABETH LYNNE RINK, PHO BA 0TH Phone number: 406-994-3833 Email: elizabeth.rink@montana.edu | MONTANA STATE UNIVERSITY - BOZEMAN MONTANA STATE UNIVERSITY-BOZEMAN 309 Montana Hall BOZEMAN, MT 597170000 DUNS: 625447982 EIN: 1816010045A1 RECIPIENT ID: |
| Change of Contact PD/PI: No | |
| Administrative Official: TRACI MIYAKAWA MONTANA STATE UNIV (BOZEMAN) BOZEMAN, MT 59717 BOZEMAN, MT 59717 Phone number: 406-994-2381 Email: tracim@montana.edu | Signing Official: TRACI MIYAKAWA MONTANA STATE UNIV (BOZEMAN) BOZEMAN, MT 59717 BOZEMAN, MT 59717 Phone number: 406-994-2381 Email: tracim@montana.edu |
| Human Subjects: Yes HS Exempt: No Exemption Number: Phase III Clinical Trial: No | Vertebrate Animals: No |
| hESC:No | Inventions/Patents: No |

RPPR Page 1

### 8.1 WHAT ARE THE MAJOR GOALS OF THE PROJECT?

Our study, Nen OnkUmbi/EdaHiYedo ("We Are Here Now," or N/E), builds on an 11-year collaborative research relationship between the Assiniboine and Sioux Tribes of the Fort Peck Reservation and Montana State University (MSU) researchers to prevent STIs, HIV, HCV, and teen pregnancy among AI youth.

N/E is a community-based participatory research (CBPR) multi-level, multi-component sexual and reproductive health (SRH) intervention, constructed on Ecological Systems Theory. N/E is based on Fort Peck tribal members' desire to implement a holistic SRH intervention for Al youth. N/E includes: 1) A school-based SRH curriculum called Native Stand, designed to address individual-level factors that lead to sexual risk behaviors; 2) a family-level curriculum called Native Voices, tailored to increase communication between adult family members and youth about SRH topics; 3) a cultural mentoring component at the community level that pairs Al youth with adults and elders to discuss traditional Al beliefs and practices about SRH; and 4) a mobilizing strategy to activate a multi-sectoral network of youth-servicing organizations at the systems level in Fort Peck to coordinate SRH services for Al youth. The overarching aim of this proposal is to refine, tailor, and finalize the components of N/E and evaluate its efficacy. We will use a cluster-randomized stepped-wedge design (SWD), in which 5 schools that Al youth from Fort Peck attend are the clusters to be randomized into the intervention 1 at a time, with all schools eventually being randomized to the intervention. The 5 schools are located in separate communities, mitigating the potential for cross-contamination. N/E is a 5-year study involving 456 15- to 18-year-old Al youth.

Our specific aims are:

AIM 1: Refine, tailor, and finalize the components of N/E. Our community advisory board and the Fort Peck-based and MSU-based research team will design culturally appropriate adaptations for N/E's 4 levels during the first year of the study, based on the analysis of our recently completed qualitative and quantitative research (focus groups, interviews, and surveys), as well as discussions with elders and community stakeholders.

AIM 2: Test the efficacy of N/E for 15- to 18-year-old AI youth. Our hypotheses are:

H1: Al youth who participate in N/E will demonstrate increased condom use at 3, 9, and 12 months. (12 months will be used in the Primary Outcome analysis; 3 and 9 months will be used in the Secondary Outcomes analysis.)

H2: Al youth who participate in N/E will demonstrate increased use of other birth control at 3, 9, and 12 months. They also will demonstrate a decrease in sexual risk behaviors as measured by reduced number of sex partners, delayed onset of sexual intercourse, and decreased substance use during sex, at 3, 9, and 12 months. (Secondary Outcomes)

H3: N/E parents/legal guardians and youth will demonstrate significantly increased communication about topics related to SRH at 3, 9, and 12 months. All youth who participate in the cultural mentoring program will demonstrate significantly increased understanding of cultural values related to traditional All beliefs regarding SRH at 3, 9, and 12 months. And All youth who participate in N/E will report significantly increased use of SRH services at 3, 9, and 12 months as a result of improved coordination among education, health care, and social service agencies on the Fort Peck Reservation. (Tertiary Outcomes)

AIM 3: Evaluate the fidelity and acceptability of NIE. N/E's fidelity and acceptability will be evaluated using qualitative methods, including focus groups, activity logs, and staff field notes and meetings.

H4: N/E will result in a viable and sustainable multi-level, multi-component SRH intervention for Al youth.

Our short-term goal is to integrate N/E into the existing Fort Peck infrastructure to ensure local sustainability. Our long-term goal is to produce a toolkit, including curriculum manuals, an SRH cultural mentoring program, and specific systems-level actions suitable for replication in other tribal communities. The public health impact is the prevention of STIs, HIV, HCV, and teen pregnancies in Al youth resulting in reduced sexual and reproductive health disparities and improved health in Al families and communities.

### 8.1.a Have the major goals changed since the initial competing award or previous report?

No

#### 8.2 WHAT WAS ACCOMPLISHED UNDER THESE GOALS?

File uploaded: R01MD012761\_ YearOneRPPR\_Accomplishments\_101518.pdf

### 8.3 COMPETITIVE REVISIONS/ADMINISTRATIVE SUPPLEMENTS

For this reporting period, is there one or more Revision/Supplement associated with this award for which reporting is required?

Νo

### 8.4 WHAT OPPORTUNITIES FOR TRAINING AND PROFESSIONAL DEVELOPMENT HAS THE PROJECT PROVIDED?

File uploaded: R01MD012761\_YearOneRPPR\_ Training&ProfessionalDevelopment\_Rink\_101518.pdf

### 8.5 HOW HAVE THE RESULTS BEEN DISSEMINATED TO COMMUNITIES OF INTEREST?

Dissemination of the notice of award for NE was made through Fort Peck Tribal Council meetings, meetings with Fort Peck Community-

RPPR Page 2

**RPPR FINAL** 

College faculty, staff and students, and was published on the Montana State University webpage as well as in the Bozeman Chronicle. In addition, Dr. Rink was selected to give a Provost Distinguished Lecture at the Museum of the Rockies (9/17/18) to the academic and public community. As part of her Distinguished Lecture Dr. Rink presented on the process of developing NE in which she presented to the Although this dissemination of NE is not about the results from the study, it does provide information to the Fort Peck tribal community and the larger Montana State University and Montanans about the study.

### B.6 WHAT DO YOU PLAN TO DO DURING THE NEXT REPORTING PERIOD TO ACCOMPLISH THE GOALS?

The following will be completed during the next reporting cycle (12/01/18 to 11/30/19):

- \* Implement baseline data collection in the 5 schools at Fort Peck between 3/01/19 to 6/01/19.
- \* Begin implementation of Aim 2 to test the efficacy of NIE for 15- to 18-year-old Al youth. Implementation of NE will begin in 9/2019 in one school at Fort Peck. The first school to receive NE in 9/2019 has yet to be determined because, as outlined in our proposal and in keeping with our study's Stepped Wedge Design, we must collect baseline data first and then randomize the schools into the
- · Implement systems level component of NE.
- \* Manage data software REDCap.
  \* Convene DMSP committee and 2 hold meetings.
- \* Hold 4 community advisory board meetings and meet with community advisory board members individually as needed.

**RPPR** Page 3 The following accomplishments have been completed during reporting period (4/01/18 -11/30/18) related to the study's specific aims (goals):

<u>AIM 1</u>. Refine, tailor, and finalize the components of NIE. Our community advisory board and the Fort Peckbased and MSU-based research team will design culturally appropriate adaptations for NIE's 4 levels during the first year of the study, based on the analysis of our recently completed qualitative and quantitative research (focus groups, interviews, and surveys), as well as discussions with elders and community stakeholders.

- 3 community advisory board meetings have been held to refine, tailor and finalize the components of NIE, including Native Stand, Native Voices, the Cultural Mentoring Program, and the System's Level adaptations.
- 4 meetings have been held specifically with Paula Firemoon, Ramey GrowingThunder and Elizabeth Rink to discuss the integration of the Cultural Mentoring Program with Native Stand and Native Voices.
- 2 meetings have been held with members of the Fort Peck Epi Team to discuss the adaptation of reproductive health services for 15-18 year old tribal youth.
- 2 discussions have been held with elders to talk about NIE.
- Subawards have been established with Fort Peck Community College, the Fort Peck Tribes Language and Culture Department, and Northern Arizona University.
- 3 meetings (2 conference calls and 1 in-person) with Dr. Julie Baldwin at Northern Arizona University who is Dr. Rink's senior research mentor on the study, to discuss tailoring of *NIE*.
- 3 meetings with Adriann Ricker, consultant to discuss adaptation of systems level component of *NIE* including working with the schools to revise their sexual and productive health education policies and meetings with the Fort Peck Epi team to tailor their services for 15 18 year old tribal youth.
- Hiring of personnel with Fort Peck Community College has begun.
- · Hiring of personnel and mentors with the Fort Peck Tribes Language and Cultural Program has begun.
- · Hired research program manager to replace Elizabeth Bird.
- Initiation of ClinicalTrials.gov forms for approval has begun.

**AIM 2:** Test the efficacy of *NIE* for 15- to 18-year-old Al youth.

- Data collection instruments have been finalized by the community advisory board, Fort Peck based research team and the Montana State University (MSU) based research team.
- Participation in 2 REDCap trainings to establish data management systems of NIE.
- Data management systems, REDCap, has been used to create the data management components of the study including the development of the data entry systems for the youth and parent surveys.
- Institutional Review Board applications have been submitted to the Fort Peck IRS and the MSU IRS for review and approval.
- Study has been registered with ClincialTrials.gov (NCT # 03694418)
- Discussions with school administrators and teachers in each of the 5 schools involved in N/E have begun to prepare for the baselines data collection from March 1, 2019 to June 1, 2019.

<u>AIM 3</u>: Evaluate the fidelity and acceptability of NIE. NIE's fidelity and acceptability will be evaluated using qualitative methods, including focus groups, activity logs, and staff field notes and meetings.

- Aim 3 has not been implemented during this reporting period because the intervention has not started yet. However, per AIM 1 and AIM 2, the tailoring of N/E has been complemented, data collection instruments have been complemented and the research protocols for N/E are being reviewed and approved by the Fort Peck IRS and the MSU IRS.
- 2 conference calls have been held with Rachel Hallum-Montes, the study's evaluation consultant, to discuss and plan for the evaluation of the fidelity and acceptability of *NIE*.

R01 Mnn1?7R1 YA::irOnARPPR Ar.r.nmnli hmP.nt Pl· Fli7::ihP.th I vnnP. Rink


1

Training and Professional Development completed during this reporting period (4/01/18 - 11/30/18) including the following:

- Attendance at 2 REDCap trainings.
- 3 meetings with Julie Baldwin, Dr. Rink's senior research mentor.
- Participation in 1 seminar on reproduction and sexuality with underserved populations.
- Dr. Rink mentored 1 undergraduate student intern as part of a summer internship program from June 2018 to August 2018.
- Research Program Manager (new hire) attended one week NIH training on NIH grants management and NIH.gov systems, protocols, policies and procedures in San Francisco in October 2018.
- Attendance at 1 seminar through the Center for American Indian and Rural Health Equity on quantitative data analysis with small populations.


RPPR FINAL

### C.PRODUCTS

### **C.1 PUBLICATIONS**

Are there publications or manuscripts accepted for publication In a journal or other publication (e.g., book, one-time publication, monograph) during the reporting period resulting directly from this award?

No

### C.2 WEBSITE(S) OR OTHER INTERNET SITE(S)

Nothing to report

#### **C.3 TECHNOLOGIES OR TECHNIQUES**



### C.4 INVENTIONS, PATENT APPLICATIONS, AND/OR LICENSES

Have Inventions, patent applications and/or licenses resulted from the award during the reporting period? No

If yes, has this information been previously provided to the PHS or to the official responsible for patent matters at the grantee organization?

### C.5 OTHER PRODUCTS AND RESOURCE SHARING

Nothing to report

| Survey Instruments | Survey instruments for youth and parent data collection |
|---|---|
| Protocols | Institutional Review Board Protocols for the MSU and Fort Peck IRBs |
| Data or Databases | REDCap |
| Evaluation Instruments | Evaluation tracking materials for systems level component of intervention |
| Educational aids or curricula | Adaptation of Native Voices for Assiniboine & Sioux Tribes |

#### **D.PARTICIPANTS**

# D.1 WHAT INDIVIDUALS HAVE WORKED ON THE PROJECT?

| | | | | jaren ereken.<br>Tarihir | oneele. | la. | | Greione (<br>Joseph | ounity. | |
|---|---|---|---|---|---|---|---|---|---|---|
| ELRINK | Υ | Rink,<br>Elizabeth<br>Lynne | OTH,BA,P I | PD/PI | 0.0 | 3.5 | 0.0 | · | | NA |
| GENEVIEVE.CO | <b>y</b> | Genevieve, Co | PhD<br>x | Research<br>Program<br>Manager | 1 3.0 | 0.0 | 0.0 | | | NA |
| JBALDWIN | у | Baldwin, Julie <b>I</b><br>Ann | PhD | Co-<br>Investigator | <u>lo.o</u> | 0.0 | 1.0 | | | NA |
| RGROWINGTH | у | GrowingThun I<br>der, Ramey | MA | Co- UNDER<br>Investigator | <u>11.0</u> | 0.0 | 0.0 | | | NA |
| PBRIEN-<br>FIREMOON | у | Brien-<br>Firemoon,<br>Paula | JMA | Co-<br>Investigator | 13.0 | 0.0 | 0.0 | | | NA |

Glossary of acronyms:

S/K - Senior/Key

DOB - Date of Birth

Cal - Person Months (Calendar) Aca - Person Months (Academic)

Sum - Person Months (Summer)

Foreign Org - Foreign Organization Affiliation

SS - Supplement Support RE - Reentry Supplement DI - Diversity Supplement

OT - Other

NA - Not Applicable

#### **D.2 PERSONNEL UPDATES**

### D.2.a Level of Effort

Will there be, in the next budget period, either (1) a reduction of 25% or more in the level of effort from what was approved by the agency for the PD/PI(s) or other senior/key personnel designated in the Notice of Award, or (2) a reduction in the level of effort below the minimum amount of effort required by the Notice of Award?

No

#### D.2.b New Senior/Key Personnel

Are there, or will there be, new senior/key personnel?

Yes

File uploaded: Cox\_BioSketch.pdf

D.2.c Changes In Other Support

Has there been a change In the active other support of senior/key personnel since the last reporting period?

Nο

D.2.d New Other Significant Contributors

Are there, or will there be, new other significant contributors?

No

D.2.e Multi-PI (MPI) Leadership Plan

 $\lor Viii$  there **be a** change in the MPI Leadership Plan for the next budget period?

NA

OMB No. 0925-0001 and 0925-0002 (Rev. 09/17 Approved Through 03/31/2020)

#### **BIOGRAPHICAL SKETCH**

NAME: Cox, Genevieve Ramsey

eRA COMMONS USER NAME: Genevieve.Cox

POSITION TITLE: Research Program Manager

**EDUCATION/TRAINING** 

| INSTITUTION AND LOCATION | DEGREE<br>(if<br>applicable) | Completion<br>Date<br>MM/YYYY | FIELD OF STUDY |
|---|---|---|---|
| University of New Hampshire | Ph.D. | 06/2012 | Sociology |
| West Virginia University | M.A. | 08/2005 | Applied Social<br>Research |
| Ohio University | B.A. | 06/2002 | English and Theater |

#### A. Personal Statement

As a community, cultural, and environmental sociologist, I am committed to better understanding how the intersection of identities and issues such as race, class, and gender should be considered in tandem with geography and context when trying to determine the ways that knowledge, attitudes, perceptions, and values inform problems of public health or community development. I completed my Ph.D. as a Community, Health, and Environment fellow and I have a broad range of experience working with community-based research. I have been involved in all stages of research projects from program management to data collection to analysis to program evaluation of applied health care interventions to the writing of findings in both scholarly publications and research briefs. I have training in quantitative, qualitative, and mixed methodology research design and analysis. My master's thesis and article entitled "Poor Women with Sexually Transmitted Infections: Providers' Perspectives on Diagnoses," looked at the role that stigma plays as a barrier to health care for low-income women with sexually transmitted infections so my applied research interests are directly related to the intervention of this study.

As an Assistant Professor at a community college for three years after graduate school focused on teaching, I kept active in the research world by being a member of the Regional Institutional Review Board at the University of Southern Maine. I then helped steer a nonprofit organization as it's Program Director. My wide-ranging training and experience has helped inculcate a dedication to working with vulnerable and underserved populations. I carry this dedication with me in the community-based participatory research projects I am a part of.

### **B.** Positions and Honors

2005-2006 Program Manager, National Visitor Use Monitoring Study of the Pacific Northwest. USDA Forest Service and Pennsylvania State University, Portland, Oregon

2010-2013 Instructor and Lecturer, Department of Sociology, University of New Hampshire, Durham, NH 2008-2013 Research Assistant, Carsey School of Public Policy, University of New Hampshire, Durham, NH

2013-2016 Assistant Professor of Sociology, Department of Social Sciences, Southern Maine Community College, South Portland, ME

2013-2016 Institutional Review Board Member, University of Southern Maine, Portland, ME

2016-2017 Program Evaluator, Partnerships for Health, Augusta, ME

2017-2018 Program Director, Renewal in the Wilderness, Portland, ME

2018-current Research Program Manager, Center for American Indian and Rural Health Equity, Montana State University, Bozeman, MT

#### **Honors:**

2007-2011 Community, Health, and Environment Fellowship, Departments of Sociology and Psychology, University of New Hampshire

2005 Velma K. Miller Award, Outstanding Graduate Student in Women's Studies, West Virginia University

#### C. Contributions to Science

# **Mentoring Future Scientists:**

As a former college professor focused on teaching, my main contributions to science have been in working to mentor future scientists. In my past classes (which have totaled upwards of 50 classes taught), we have had a focus on current social problems through the scientific lens of evidence-based research. This works to expand the student's knowledge base beyond the personal and anecdotal to understanding larger structural patterns and historical influence. I am extremely proud to have been a part of so many students' understanding of the importance of the scientific method and evidence-based research beyond their own personal experience, especially at the community college level.

#### **Community Context:**

Much of my past written work has to do with utilizing the community context to better understand behaviors, attitudes, and outcomes within communities. My doctoral dissertation was entitled, "Culture, Place, and Identity in a Mobile Community" and focused on ways values and place identity combine to create a community cultural identity that participants often adhere to. Related articles, briefs, and research presentations:

- Cox, Genevieve R., Corinna Jenkins Tucker, Erin Sharp, Karen Van Gundy, and Cesar Rebellon. 2014. "Practical Considerations: Community Context in a Declining Rural Economy and Emerging Adults' Educational and Occupational Aspirations." *Emerging Adulthood.* 2 (3): 173-183.
- Cox, Genevieve R. and Corinna Jenkins Tucker. 2011. "No place like home: Place and community identity among North Country youth." New England Issue Brief No. 24. January, 2011. The Carsey Institute, University of New Hampshire: Durham, NH.
- March 23, 2013. "Place Identity and Artistic Visual Integration: Burning Man Participants in Portland, OR." Presentation at the Annual Meeting of the Eastern Sociological Association. Boston, MA.
- February, 2012. Genevieve Cox. "Urban Mobile Artists: Why Place Still Matters for Burners in Portland, Oregon." Presentation at the Annual Meeting of the Eastern Sociological Association. New York, NY.
- November, 2011. Erin Sharp, Genevieve Cox, Cesar Rebellion, Corinna Jenkins Tucker, and Karen Van Gundy. "The Power of Rural Youth: Findings from the Coos Youth Study." Presentation at the New Hampshire Annual Celebration of National Rural Health Day. Meredith, NH.

#### Familial Relationships:

My research has also looked at ways that familial context interacts with outcomes for adolescents in terms of violence within the family and how larger economic forces affect relationships within the family.

- Tucker, Corinna Jenkins, Genevieve R. Cox, Erin Sharp, Karen Van Gundy, Cesar Rebellon, and Nena Stracuzzi. 2013. "Sibling Proactive and Reactive Aggression in Adolescence." *Journal of Family Violence*. 28(3):299-310.
- Tucker, Corinna Jenkins and Genevieve R. Cox. 2011. "Coos teens' view of their family economic stress tied to quality of relationships at home." New England Issue Brief No. 28. October, 2011. The Carsey Institute, University of New Hampshire: Durham, NH.

# **Socioeconomic Status and Sexually Transmitted Infection:**

My master's thesis and subsequent manuscript focus on ways that stigma affects the experience of STI diagnosis between a provider and a patient.

Cox, Genevieve R. 2011. "Poor Women with Sexually Transmitted Infections: Providers' Perspectives on Diagnoses." *Online Journal of Rural Nursing and Health Care.* 11(2).

#### E. IMPACT

E.1 WHAT IS THE IMPACT ON THE DEVELOPMENT OF HUMAN RESOURCES?

Not Applicable

 ${\tt E.2WHATISTHE\,IMPACT\,ONPHYSICAL, INSTITUTIONAL, OR\,INFORMATION\,RESOURCES\,THAT\,FORM\,INFRASTRUCTURE?}$ 

NOTHING TO REPORT

E.3 WHAT IS THE IMPACT ON TECHNOLOGY TRANSFER?

Not Applicable

E.4 WHAT DOLLAR AMOUNT OF THE AWARD'S BUDGET IS BEING SPENT IN FOREIGN COUNTRY(IES)?

NOTHING TO REPORT

#### F. CHANGES

#### F.1 CHANGES IN APPROACH AND REASONS FOR CHANGE

Not Applicable

#### F.2 ACTUAL OR ANTICIPATED CHALLENGES OR DELAYS AND ACTIONS OR PLANS TO RESOLVE THEM

The challenges and delays encountered during this reporting period (4/01/18 to 11/30/18) and related actions/plans to resolve them are listed below.

- \* Elizabeth Bird resigned from her position in the beginning of the reporting period and new search had to be conducted to replace her. The search took several months longer than anticipated and was completed in August 2018. Currently there is a new hire who is working as the Research Program Manager for the study. The new hire began work on September 4, 2018.
- \* Two prominent elders died at Fort Peck, one in June 2018 and the other in July 2018. Both deaths were unexpected and were felt by all Fort Peck Tribal members. As a result several weeks were taken up with grieving and ceremonies to honor the passing of the two elders. There is of course no way to plan for these types of sorrowful events in tribal communities. Because of the role that the Fort Peck Tribal College and the Fort Peck Tribes Language and Culture Program have in the community study personnel were attentive to honoring the 2 deaths which delayed study activities.
- \* In the original proposal (that was truncated in the NOA by 4 months) the end of Year 1 baseline data collection was to be completed. The base line data collection was planned with the 5 schools in the study during the proposal submission process. Thus we could not change the base line data collection plans for Spring 2019 as schools have complicated academic schedules. Base line data collection will take place during Year 2 in Spring 2019 as initially planned as part of Year 1.
- \* All human subjects requirements were to be completed during Year 1 in the original proposal. The truncation of Year 1 in the NOA by 4 months has delayed this process. At present all the research protocols have been approved by the study's community advisory board; and Fort Peck IRB and MSU IRB are reviewing the research protocols for approval. It is anticipated that all human subjects requirements will be finalized by December 1, 2018 at the latest.
- \* Because of the time taken to recruit and hire a new research program manager and the death of 2 elders at Fort Peck, sub awards to Fort Peck Community College, the Fort Peck Tribes Language and Culture Program and Northern Arizona University, were late in getting executed.

# F.3 SIGNIFICANT CHANGES TO HUMAN SUBJECTS, VERTEBRATE ANIMALS, BIOHAZARDS, AND/OR SELECT AGENTS

#### F.3.a Human Subjects

No Change

#### F.3.b Vertebrate Animals

No Change

#### F.3.c Blohazards

No Change

#### F.3.d Select Agents

No Change

#### G. SPECIAL REPORTING REQUIREMENTS

# G.1 SPECIAL NOTICE OF AWARD TERMS AND FUNDING OPPORTUNITIES ANNOUNCEMENT REPORTING REQUIREMENTS

File(s) uploaded: FPIRB\_FWA\_2018.pdf

#### G.2 RESPONSIBLE CONDUCT OF RESEARCH

Not Applicable

#### G.3 MENTOR'S REPORT OR SPONSOR COMMENTS

Not Applicable

# **G.4 HUMAN SUBJECTS**

G.4.a Does the project involve human subjects?

Yes

Is the research exempt from Federal regulations?

No

Does this project involve a clinical trial?

Yes

If yes, is this an NIH-defined Phase III Clinical Trial?

No

#### G.4.b Inclusion Enrollment Data

Report Attached: 'We are here now' - a multi-level, multi-component sexual and reproductive health intervention for American Indian youth

#### G.4.c ClinIcalTrials.gov

Does this project include one or more applicable clinical trials that must be registered in ClinicalTrials.gov under FDAAA?

Yes

If yes, provide the ClinicalTrials.gov identifier, NCT number (e.g., NCT00654321) for those trials: NCT03694418

# G.5 HUMAN SUBJECTS EDUCATION REQUIREMENT

Are there personnel on this project who are newly involved in the design or conduct of human subjects research?

No

# G.6 HUMAN EMBRYONIC STEM CELLS (HESCS)

Does this project involve human embryonic stem cells (only hESC lines listed as approved in the NIH Registry may be used in NIH funded research)?

No

# **G.7 VERTEBRATE ANIMALS**

Does this project Involve vertebrate animals?

No

#### **G.8 PROJECT/PERFORMANCE SITES**

| | (a) | Soften Maria Carlo | Colores<br>Colores<br>Colores Colore |
|---|---|---|---|
| <b>Primary:</b> MONTANA<br>STATE UNIVERSITY -<br>BOZEMAN | 625447982 | MT-001 | P.O. Box 173540<br>318 Herrick Hall<br>BOZEMAN MT 597173540 |
| Fort Peck Community<br>College | 102366432 | MT-001 | PO Box 398<br>Poplar MT 592559398 |
| Fort Peck Assiniboine & Sioux Tribes Language & Culture Dept | 106578164 | MT-001 | PO Box 1027<br>Poplar MT 592551027 |

#### **G.9 FOREIGN COMPONENT**

No foreign component

#### **G.10 ESTIMATED UNOBLIGATED BALANCE**

G.10.a Is it anticipated that an estimated unobligated balance (including prior year carryover) will be greater than 25% of the current year's total approved budget?

Yes

Estimated unobligated balance: 666930

#### G.10.b Provide an explanation for unobligated balance:

The estimate unobligated balance will be greater that 25% because: 1) Year 1 was truncated by 4 months; 2) there was a new hire that had to be recruited and hired; 3) the subawards were delayed in getting executed because of the time allocated to getting the new hire and the death of 2 elders at Fort Peck during the Summer of 2018.

#### G.10.c If authorized to carry over the balance, provide a general description of how it is anticipated that the funds will be spent

The carryover funds will be used to complete the following:

- \* Hold monthly team meetings and quarterly CAB meetings. When necessary, we will meet with CAB members individually.
- \* Continue monthly trips to Fort Peck.
- \* Recruit, hire, and train staff in Native Stand and Native Voices; identify the cultural mentors; purchase all necessary materials and supplies.
- \* Collect baseline data from March 1, 2019 to June 1, 2019 as originally planned in Year 1.
- \* Upon completion of the baseline data collection randmonize the 5 schools for participation in the intervention.
- \* Analyze baseline data collection in collaboration with the CAB.
- \* Implement evaluation of the systems level intervention with the Fort Peck Epi Team.
- \* Start the implement of the full intervention in 1 school beginning September 1, 2019.
- \* Establish DSM Committee and hold 2 meetings.
- \* Establish contracts with study consultants.

#### **G.11 PROGRAM INCOME**

Is program Income anticipated during the next budget period?

No

#### **G.12 F&A COSTS**

Is there a change In performance sites that will affect F&A costs?

No

G.1 (FPIRB\_FWA\_2018.pdf)

FWA#: FWA00019355 OMB No. 0990-0278

Institution: Fort PeckCommunity College Approved for use through July 31, 2020

Expires: **06/20/2023** 

# Federalwide Assurance (FWA)

#### for the Protection of Human Subjects

#### L Institution Filing Assurance

Legal Name: Fort Peck Community College

City: Poplar State/Province: MT Country: USA

#### Institutional Com.u,onents

List below all components over which the Institution has legal authority that operate under a different name. Also list with an asterisk(\*) any alternate names under which the Institution operates.

NOTE: The Signatory Official signing this Assurance must be legally authorized to represent the Institution providing this Assurance and all components listed below.

Name of Component or Stat

Alternate Names Used City (or Country if Outside U.S.)

Fort Peck Community College !RB 1/1 Poplar MT A

# 3. Statement of Principles

This Institution assures that all of its activities related to human subjects research, regardless of the source of support, will be guided by the following statement of principles governing the institution in the discharge of its responsibilities for protecting the rights and welfare of human subjects of research conducted at or sponsored by the institution. (indicate below)

The Belmont Report
The Declaration of Helsinki

#### 4, Applicability

#### G. l (FPIRB FW A 2018.pdf)

- (a) This Assurance applies whenever this Institution becomes engaged in human subjects research conducted or supported by any U.S. federal department or agency that has adopted the U.S. Federal Policy for the Protection of Human Subjects (also known as the Common Rule), unless the research is otherwise exempt from the requirements of the Common Rule or the department or agency conducting or supporting the research determines that the research shall be conducted under a separate assurance.
- (b) Optional: This Institution elects to apply the following to all of its human subjects research regardless of the source of support, except for research that is covered by a separate assurance:

The Common Rule and subparts B, C, and D of the HHS regulations at 45 CFR part 46

# 5, Assurance of Compliance with the Terms of the Federalwide Assurance

(a) This Institution assures that whenever it engages in research to which this Assurance applies, it will comply with the Terms of the Federalwide Assurance (contained in a separate document on the Office for Human Research Protections (OHRP) website).

# 6, Designation of Institutional Review Boards (IRBs)

This Institution assures that it will rely upon only IRBs registered with OHRP for review of research to which this FWA applies. This institution (a) designates the following internal IRB(s) for review of research under this Assurance; or (b) does not have an internal IRB and designates the following external IRB for review of all research to which this FWA applies or, if multiple external IRBs are relied upon, the following external IRB that reviews the largest percentage of research to which this fWA applies.

NOTE: Institutions designating internal IRBs do not need to designate any of the external IRBs upon which it relies.

HHSIRB

Registration
Number Name of IRB as Registered with HHS

Is the IRB Internal or External to the Institution?

# 1, Human Protecti!)ns Administrator (e.g., Human Subjects Administrator or Human Subjects Contact Person)

First Name: Joy Middle Initial: Last Name: Toavs

Degrees or Suffix: BA Institutional Title: Administrative Officer

Institution: Fort Peck Community College

Telephone: 406 768-5555 FAX: 406 768-3026 E-Mail: jtoavs@fpcc.edu

Address: P.O. Box 398

605 Indian Avenue

City: Poplar State/Province: MT Country: USA

#### Signatory Official (i.e., Official Legally Authorized to Represent the Institution)

I have read and agree to the Terms of the Federalwide Assurance.

I recognize that providing research investigators, /RB members and staff, and other relevant personnel with appropriate initial and continuing education and training about human subject protections will help ensure that the requirements of this Assurance are satisfied.

Acting officially **in** an authorized capacity on behalf of this Institution and with an understanding of the Institution's responsibilities under this Assurance, I assure protections for human subjects as specified above. The IRB(s) that this institution relies upon will comply with the Terms of the Federalwide Assurance when reviewing research covered by this Assurance and possess appropriate knowledge of the local context in which this Institution's research will be conducted.

All information provided with this Assurance is up-to-date and accurate. I am aware that false statements could be cause for invalidating this Assurance and may lead to other administrative or legal action.

Signature: Wayne Two Bulls MS Ed.

Date: 06/20/2018

First Name: Wayne Middle Initial: Last Name: Two Bulls

Degrees or Suffix: MS Ed. Institutional Title: Vice President of Academics

Institution: Fort Peck Community College

Telephone: 406 768-6300 FAX: 406 768-6301 E-Mail: WTwoBulls@fpcc.edu

Address: P.O. Box 398

605 Indian Avenue

City: Poplar State/Province: MT Country: USA

#### 2, FWA AQProval

The Federal wide Assurance for the Protection of Human Subjects for Institutions Within the United States submitted to **HHS** by the above Institution is hereby approved.

Assurance Number: FWA00019355 Expiration Date: 06/20/2023
Signature of HHS Approving Official: Gail Holloway Date: 06/20/2018

According to the Paperwork Reduction Act of 1995, no persons are required to respond to a collection of information unless it displays a valid OMB control number. The valid OMB control number for this information collection is 0990-0278. The time required to complete this information collection is estimated to average 30 minutes per response, including the time to review instructions, gather the data needed, and complete and review the information collection. If you have comments concerning the accuracy of the time estimate(s) or suggestions for improving this form, please write to: U.S. Department of Health & Human Services, OS/OCIO/PRA, 200 Independence Ave., S.W., Suite 336-E, Washington D.C. 20201, Attention: PRA Reports Clearance

# Inclusion Enrollment Report

Inclusion Data Record (IDR) #:200138 Using an Existing Dataset or Resource: No

Delayed Onset Study ?: No Clinical Trial: Yes

Enrollment Location: Domestic NIH Defined Phase III Clinical Trial: No

Study Title: 'We are here now' - a multi-level, multi-component sexual and reproductive health intervention for American Indian youth

# **Planned Enrollment**

| | Ethnic Gateaories | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Racial Categories | Not Hispanic or Latino | | | Hispanic or Latino | | | Unknown/Not<br>Reported Ethnicity | | | Total |
| | Female | Male | Unknown/<br>Not Reported | Female | Male | Unknown/<br>Not Reported | Female | Male | Unknown/<br>Not Reported | |
| American Indian/Alaska Native | 500 | 500 | | 0 | 0 | | | | | 1000 |
| Asian | 0 | 0 | | 0 | 0 | | | | | 0 |
| Native Hawaiian or<br>Other Pacific Islander | 0 | 0 | | 0 | 0 | | | | | 0 |
| Black or African American | 0 | 0 | | 0 | 0 | | | | | 0 |
| While | 4 | 4 | | 0 | 0 | | | | | 8 |
| More than One Race | 0 | 0 | | 0 | 0 | | | | | 0 |
| Unknown or Not Reported | | | | | | | | | | |
| Total | 504 | 504 | | 0 | 0 | | | | | 1008 |

# **Cumulative Enrollment**

**NOTE:** No cumulative enrollment data exists. Although prompted to do so, the PD/PI did not enter information. No data can be displayed.

# Nen OnkUmbi/EdaHiYedo ("We Are Here Now") Informed Consent to Participate in Human Subjects Research with Montana State University in Partnership with Fort Peck Community College

# What is this project about?

We Are Here Now is an intervention project with Fort Peck Community College and Montana State University. The purpose of this intervention is to teach youth at Fort Peck important things they need to know about sex so that they can stay healthy and not get a sexually transmitted disease, HIV, or Hepatitis C, and so that they can make healthy decisions about having children, getting pregnant, or getting someone pregnant. We Are Here Now also teaches Assiniboine and Sioux youth about their culture and traditional beliefs and practices about what it means to be a young Native person who will soon be an adult.

# Why me?

You have been selected to participate in *We Are Here Now* because you are a young person at Fort Peck. You may choose to participate or not participate at any time.

# What happens to me if I decide to participate?

If you decide to be in *We Are Here Now,* you will participate in a survey that will take 50 to 60 minutes. You will be asked to complete this survey three more times during the next year so that we can keep track of any changes you may have in your beliefs and behaviors as a result of participating in *We Are Here Now.* You will be asked several questions about different topics related to sex, having children, and sexually transmitted diseases in order to learn about what you think about having children and what you know about sexually transmitted diseases. You will also be asked questions about your sexual behavior and experiences with drugs and alcohol. You will also be asked questions about your feelings and emotions and your traditional culture. It is important that you know that all of your responses on this survey are anonymous. This means that no one will know that it is you who answered these questions. Your responses will be kept track of in the computer that you are taking the survey on. Your name will be nowhere in the computer or on the survey. If you agree to participate in this survey, you will receive a \$10 gift card that you can use here at Fort Peck. Also by agreeing to participate in *We Are Here Now*, your parent/legal guardian is agreeing to participate in an educational program called *Native Voices*, and you are agreeing to be part of a cultural mentoring program with the Fort Peck Tribes' Language and Culture Department.

# What are the risks?

There may be minor risks to agreeing to participate in the survey. Some of the questions may make you feel uncomfortable, sad, or confused. You may choose to stop the survey at any time or decline to answer a particular question. The questions will be about your life experiences as they relate to sex, drug and alcohol use, having children, sexually transmitted diseases, your feelings and emotions, and your understanding of your traditional culture. None of the things that you say on the survey will be connected to your name.

#### What are the benefits?

The information gathered in this survey will help the intervention's research team and members of the Fort Peck community to understand what kind of impact your participation in *We Are Here Now* is having on your decisions to avoid getting a sexually transmitted disease and your decisions about having children when you feel you are ready. We would also like you to know that if you tell us about any abusive situation you are experiencing or have experienced, we will need to report that to the appropriate services here at Fort Peck so that you can receive assistance.

# Who gets access to information from this interview?

The research team has access to the data collected for this project. The *We Are Here Now* community advisory board will also have access to the data collected for this intervention. All responses on this survey will be anonymous. Neither the research team nor the community advisory board will know who you are and what your responses to the survey are.

<u>How am I informed about the results of the project, and when will they be released and presented</u> to someone else?

We will publish the intervention results and make presentations on the results from *We Are Here Now.* Your identity will never appear in a publication or in print or be discussed at a presentation. In addition, you will have the opportunity to learn about the intervention results by contacting members of the research team, attending community meetings where we share the results of the project, and through local (Fort Peck Reservation) media.

# Who is involved in We Are Here Now?

If you have any questions regarding this survey please contact:

# Paula FireMoon, Fort Peck Community College

Email: PFiremoon@fpcc,edu; Phone: 406.768.6300

# Elizabeth Rink, Montana State University

Email: elizabeth.rink@montana.edu; Phone: 406.994.3833

# **CONSENT STATEMENT**

# If the research <u>participant</u> is a minor:

If you are 18 years or younger and you agree to participate in this survey, please read, complete, and sign the statement below. By signing this consent form you are giving your verbal and written consent to complete this survey.

| Minor: I have read the above and under | stand the discomfort, inconvenience, and risks associated with this |
|---|---|
| survey. | stand the discomfort, inconvenience, and risks associated with this |
| | , <b>agree</b> to participate in this survey. |
| Name of Minor | |
| Minor Participant Signature: | Date: |
| Parent/Legal Guardian agreement for | minor: |
| If as a parent or guardian you <b>do want</b> y<br>the statement below. | our child to participate in this survey, please read, complete, and sign |
| Parent/Legal Guardian for Minor: I havrisks associated with this survey. | ve read the above and understand the discomfort, inconvenience, and |
| I,<br>Name of Parent/Guardian | , do agree to have my child participate in this survey. |
| Parent/Guardian Signature: | Date: |
| Survey Administrator Signature: | Date |

#### Introduction

This survey will ask you questions about yourself. Many of the questions are about topics related to sex, alcohol and drugs, how you talk to your parents about sex, and your life experiences. Please remember that all of your answers to the questions are anonymous. This means that no one will know that it was you who answered these questions. No one will know your name and your answers to the questions. Only the answers to the questions will be recorded, not your name.

Thank you for taking the time to complete this survey.

| SECTION 1: DEMOGRPA | HICS | |
|---|---|---|
| 1.1 What is your gender? | Male | Female |
| 1.2 How old are you? | | (age in years) |
| 1.3 What town do you live | in? | |
| Frazer Oswego Wolf Point Poplar Brockton Fort Kipp Other | | - |
| .41 What grade are you in? | | |
| gth<br>10th | | |

# **SECTION 2: CULTURAL IDENTITY** (terliary outcome variable)

The next set of questions are related to your culture and what it means for you to be an American Indian.

- 2.1 How much do you now live by or follow an American Indian way of life?
  - a. Not at all
  - b. A little

11th 12th

- c. Some
- d. A lot
- 2.2 How much do you now live by or follow a White or Anglo way of life?
  - a. Not at all
  - b. A little
  - c. Some
  - d. A lot
- 2.3 How important is it to you to follow religious or spiritual beliefs which are based on traditional Indian beliefs?
  - a. Not at all important
  - b. Not very important

| <ul><li>c. Somewhat important</li><li>d. Very important</li></ul> | |
|---|---|
| 2.4 How important is it to you to follow religious or s Catholic, Baptist, Mormon, etc.? | piritual beliefs that are based on Christian beliefs such as |
| <ul><li>a. Not at all important</li><li>b. Not very important</li><li>c. Somewhat important</li><li>d. Very important</li></ul> | |
| 2.7. How proud are you to be an American Indian? | |
| <ul><li>a. Not at all proud</li><li>b. Not very proud</li><li>c. Somewhat proud</li><li>d. Very proud</li><li>e. I do not consider myself to be an American</li></ul> | n Indian. |
| 2.8 What kinds of activities have you participated in | over the past year? |
| ☐ Gathering traditional foods | ☐ Singing and drumming |
| ☐ Beading | ☐ Traditional ceremonies |
| ☐ Hand/stick games | ☐ Sweats |
| ☐ Hunting | ☐ Kinship History |
| ☐ Using sacred medicine | ☐ Going to Pow Wows |
| ☐ Dancing at Pow Wows | ☐ Learning what it means to be a |
| ☐ Traditional beliefs about sex | man (if male)/woman(if female) |
| $\square$ Learning about what it means to be | |
| an adult | |
| ☐ Sundance/Medicine lodge | |
| ☐ Other (please describe): | |
| SECTION 3: COMMUNICATION ABOUT SEX WIT variable) | TH PARENTS/LEGAL GUARDIAN (tertiary outcome |
| Now you are going to be asked questions about wh your parents/legal guardian about. | at kinds of topics related to sex you do or do not talk with |
| 3.1. Have you talked with your parent/legal guardia | n about each of the following topics in the past year? |
| a. What qualities are important in choosing of | |
| <ul><li>b. What qualities to look for in a boyfriend/gir</li><li>partner</li></ul> | rifriend/life |
| c. How boys' bodies change physically as th | |
| <ul> <li>d. How girls' bodies change physically as the</li> <li>e. How women get pregnant and have babie</li> </ul> | |
| f. Symptoms of sexually transmitted infection | |
| g. Reasons why people like to have sex | |

| h. How well birth control can prevent pregnancy |
|--------------------------------------------------------------------------|
| i. How to choose a method of birth control |
| j. How to say no if someone wants to have sex and you don't want to |
| k. How well condoms can prevent sexually transmitted infections (STIs) |
| I. Menstruation (having menstrual periods) |
| m. The importance of not pressuring other people to have sex |
| n. How you will make decisions about whether or not to have sex |
| o. Consequences of getting pregnant/getting someone preqnant |
| p. How to use a condom |
| q. Reasons why you should not have sex |
| r. Masturbation |
| s. What it feels like to have sex |
| t. Homosexuality/people being qay |
| u. Wet dreams fmeasured for boys onlyl |
| v. What to do if a partner doesn't want to use a condom |
| w. How people can prevent getting sexually transmitted infections (STIs) |
| x. How you will know if you are in love |

# SECTION 4: ACCESS TO REPRODUCTIVE HEALTH SERVICES(terliary outcome variable)

This next set of questions is about where you go to get services like getting a pregnancy test, sexually transmitted disease test, or birth control.

- 4.1 Have you ever been to Indian Health Service or Fort Peck Tribal Health for things like condoms, birth control, a pregnancy test or a sexually transmitted disease test?
  - a. yes
  - b. no
- 4.2 If you need to get condoms, birth control, a pregnancy test, or a sexually transmitted disease test, where would you go? (Mark all that apply)
  - a. Indian Health Services
  - b. Fort Peck Tribal Health
  - c. Roosevelt County Health Department
  - d. Somewhere off the reservation
  - e. The Hospital
  - f. A private doctor
  - g. Local stores
  - h. School nurse
  - i. Teachers or counselors in your school
  - j. Elder
  - k. Other
- 4.3 If you had to put your response on a scale, how uncomfortable or comfortable would you say you feel when a health care provider talks with you about birth control and STDs? Would you say you are:
  - a. Very uncomfortable
  - b. Slightly uncomfortable
  - c. Neither uncomfortable or comfortable

| d. Slightly comfortable e. Very comfortable |
|---|
| 4.4 In general, how satisfied or dissatisfied would you say you are with the birth control and STD information<br>and services you have received from health care providers in the past? |
| <ul> <li>a. Very dissatisfied</li> <li>b. Somewhat dissatisfied</li> <li>c. Neither satisfied nor dissatisfied</li> <li>d. Somewhat satisfied</li> <li>e. Very satisfied</li> </ul> |
| 4.5 How likely is it that you will seek birth control or STD services from a health care provider in the next year? |
| <ul> <li>a. Not at all likely</li> <li>b. A little likely</li> <li>c. Moderately likely</li> <li>d. Very likely</li> <li>e. Extremely likely</li> </ul> |
| Section 5: Sexual Behavior (primary, secondary, tertiary outcome variables) |
| The next questions ask you about your sexual behavior. |
| 5.1 Have you ever had sexual intercourse? Yes No |
| If you have <u>never</u> had sexual intercourse, skip to Section 6. |
| 5.2 How old were you when you had sexual intercourse for the first time? |
| <ul> <li>a. I have never had sexual intercourse</li> <li>b. 11 years old or younger</li> <li>c. 12 years old</li> <li>d. 13 years old</li> <li>e. 14 years old</li> <li>f. 15 years old</li> <li>g. 16 years old</li> <li>h. 17 years old or older</li> </ul> |
| 5.3 During your life, with how many people have you had sexual intercourse? |
| <ul> <li>a. 1 person</li> <li>b. 2 people</li> <li>c. 3 people</li> <li>d. 4 people</li> <li>e. 5 people</li> <li>f. 6 or more people</li> </ul> |
| 5.4 During the <u>past month</u> , how many people have you had sex with? [# of people] |
| 5.5 During the past month, how many TIMES have you had sex?times |
| 5.6 Of the times you had sex over the <u>past month</u> , how many TIMES was a condom used?times |

| 5.7 Of the times you had sex over the <u>past month</u> , how many TIMES did you use birth control other than a condom, like birth control pills or having a deprova shot?times |
|---|
| ⊕er the past month, did you drink alcohol or take any kind of drug and have sex? Yes No |
| 5.9 Did you drink alcohol or use drugs before you had sexual intercourse the <i>last</i> time? |
| <ul><li>a. I have never had sexual intercourse</li><li>b. Yes</li><li>c. No</li></ul> |
| 5.10 The last time you had sexual intercourse, what one method did you or the person you had sex with use to prevent pregnancy? (Select only one response.) |
| <ul> <li>a. No method was used to prevent pregnancy</li> <li>b. Birth control pills</li> <li>c. Condoms</li> <li>d. An IUD (such as Mirena or ParaGard) or implant (such as Implanon or Nexplanon)</li> <li>e. A shot (such as Depo-Provera), patch (such as OrthoEvra), or birth control ring (such as NuvaRing)</li> <li>f. Withdrawal or some other method</li> <li>g. Not sure</li> </ul> |
| 5.11 How many times have you been pregnant or gotten someone pregnant? |
| <ul><li>a. 0 times</li><li>b. 1 time</li><li>c. 2 or more times</li><li>d. Not sure</li></ul> |
| 5.12 Have you ever been tested for HIV, the virus that causes AIDS? |
| a. Yes<br>b. No<br>c. Not sure |
| 5.13 Have you ever been tested for other sexually transmitted diseases (STDs), such as genital herpes, chlamydia, syphilis, or genital warts? |
| a. Yes<br>b. No<br>c. Not sure |
| 5.14Have you ever been told by a doctor or nurse that you had the HIV infection or any other sexually transmitted disease (STD)? |
| a. Yes<br>b. No<br>c. Not sure |
| If yes, did you receive follow-up care? Yes No Not sure |
| 5.15 Have you ever been tested for HCV (Hepatitis C)? |
| a. Yes<br>b. No |

- c. Not sure
- 5.16 Have you ever been told by a doctor or nurse that you had Hepatitis C?
  - a. Yes
  - b. No
  - c. Not sure

If ves, did you receive follow-up care? Yes No Not sure

# Section 6: Substance Use **Questions** (secondary outcome variables)

These next questions are about alcohol and drug use.

6.1 How old were you when you tried any of the following for the first time?

| Alcohol | I have<br>never | 8 years old or | 9 or<br>10 | 11 or<br>12 | 13 or<br>14 | 15 or<br>16 | 17 years old or older |
|---|---|---|---|---|---|---|---|
| | tried | younger | years<br>old | years<br>old | years<br>old | years<br>old | |
| Marijuana<br>(grass, pot,<br>weed, or reefer) | I have<br>never<br>tried | 8 years<br>old or<br>younger | 9 or<br>10<br>years<br>old | 11 or<br>12<br>years<br>old | 13 or<br>14<br>years<br>old | 15 or<br>16<br>years<br>old | 17 years old or older |
| Meth (speed,<br>crystal, crank, or<br>ice) | I have<br>never<br>tried | 8 years<br>old or<br>younger | 9 or<br>10<br>years<br>old | 11 or<br>12<br>years<br>old | 13 or<br>14<br>years<br>old | 15 or<br>16<br>years<br>old | 17 years old or older |
| Cocaine<br>(powder, crack,<br>or freebase) | I have<br>never<br>tried | 8 years<br>old or<br>younger | 9 or<br>10<br>years<br>old | 11 or<br>12<br>years<br>old | 13 or<br>14<br>years<br>old | 15 or<br>16<br>years<br>old | 17 years old or older |
| Ecstasy<br>(MOMA) | I have<br>never<br>tried | 8 years<br>old or<br>younger | 9 or<br>10<br>years<br>old | 11 or<br>12<br>years<br>old | 13 or<br>14<br>years<br>old | 15 or<br>16<br>years<br>old | 17 years old or older |
| Heroin (smack, junk, or diesel) | I have<br>never<br>tried | 8 years<br>old or<br>younger | 9 or<br>10<br>years<br>old | 11 or<br>12<br>years<br>old | 13 or<br>14<br>years<br>old | 15 or<br>16<br>years<br>old | 17 years old or older |
| Steroids (pills or<br>shots without a<br>doctor's<br>prescription) | I have<br>never<br>tried | 8 years<br>old or<br>younger | 9 or<br>10<br>years<br>old | 11 or<br>12<br>years<br>old | 13 or<br>14<br>years<br>old | 15 or<br>16<br>years<br>old | 17 years old or older |
| Inhalants (sniff glue, breathe the contents of aerosol spray cans, or inhale any paints or sprays to get hiQh) | I have<br>never<br>tried | 8 years<br>old or<br>younger | 9 or<br>10<br>years<br>old | 11 or<br>12<br>years<br>old | 13 or<br>14<br>years<br>old | 15 or<br>16<br>years<br>old | 17 years old or older |

6.2 During your life, how many times have you used any of the following:

| Alcohol | 0 times | 1-2<br>times | 3-9<br>times | 10-19<br>times | 20-39<br>times | 40-99<br>times | 100 or<br>more<br>times |
|---|---|---|---|---|---|---|---|
| Marijuana<br>(grass, pot,<br>weed, or<br>reefer) | 0 times | 1-2<br>times | 3-9<br>times | 10-19<br>times | 20-39<br>times | 40-99<br>times | 100 or<br>more<br>times |
| Meth (speed, crystal, crank, or ice) | 0 times | 1-2<br>times | 3-9<br>times | 10-19<br>times | 20-39<br>times | 40-99<br>times | 100 or<br>more<br>times |
| Cocaine<br>(powder,<br>crack, or<br>freebase) | 0 times | 1-2<br>times | 3-9<br>times | 10-19<br>times | 20-39<br>times | 40-99<br>times | 100 or<br>more<br>times |
| Ecstasy<br>(MOMA) | 0 times | 1-2<br>times | 3-9<br>times | 10-19<br>times | 20-39<br>times | 40-99<br>times | 100 or<br>more<br>times |
| Heroin<br>(smack,<br>junk, or<br>diesel) | 0 times | 1-2<br>times | 3-9<br>times | 10-19<br>times | 20-39<br>times | 40-99<br>times | 100 or<br>more<br>times |
| Steroids (pills or shots without a doctor's prescription) | 0 times | 1-2<br>times | 3-9<br>times | 10-19<br>times | 20-39<br>times | 40-99<br>times | 100 or<br>more<br>times |
| Inhalants<br>(sniff glue,<br>breathe the<br>contents of | 0 times | 1-2<br>times | 3-9<br>times | 10-19<br>times | 20-39<br>times | 40-99<br>times | 100 or<br>more<br>times |
| aerosol<br>spray cans,<br>or inhale<br>any paints | | | | | | | |
| or sprays to qet hiqh) | | | | | | | |

# 6.3 During the past 30 days, how many times did you use any of the following:

| Alcohol | 0 times | 1 time | 2 times | 3 to 5 times | 6 to 9 times | 10to 19<br>times | 20 or more times |
|---|---|---|---|---|---|---|---|
| Marijuana<br>(grass, pot,<br>weed, or reefer) | 0 times | 1 time | 2 times | 3 to 5 times | 6 to 9<br>times | 10 to 19<br>times | 20 or more times |
| Meth (speed,<br>crystal, crank,<br>or ice) | 0 times | 1 time | 2 times | 3 to 5 times | 6 to 9<br>times | 10 to 19<br>times | 20 or more times |
| Cocaine<br>(powder, crack,<br>or freebase) | 0 times | 1 time | 2 times | 3 to 5 times | 6 to 9<br>times | 10to 19<br>times | 20 or more<br>times |
| Ecstasy<br>(MOMA) | 0 times | 1 time | 2 times | 3 to 5 times | 6 to 9 times | 10 to 19<br>times | 20 or more times |

| Heroin (smack, iunk, or diesel) | 0 times | 1 time | 2 times | 3 to 5 times | 6 to 9<br>times | 10 to 19<br>times | 20 or more times |
|---|---|---|---|---|---|---|---|
| Steroids (pills or<br>shots without a<br>doctor's<br>prescription) | 0 times | 1 time | 2 times | 3 to 5 times | 6 to 9<br>times | 10 to 19<br>times | 20 or more times |
| Inhalants (sniff glue, breathe the contents of aerosol spray cans, or inhale any paints or sprays to get hiqh) | 0 times | 1 time | 2 times | 3 to 5 times | 6 to 9<br>times | 10 to 19 times | 20 or more<br>times |

- 6.4 During the past 30 days, on how many days did you have 5 or more drinks of alcohol in a row-that is, within a couple of hours?
  - a. 0 days
  - b. 1 day
  - c. 2 days
  - d. 3 to 5 days
  - e. 6 to 9 days
  - f. 10 to 19 days
  - g. 20 or more days
- 6.5 During your life, how many times have you used a needle to inject any illegal drug into your body?
  - a. 0 times
  - b. 1 time
  - c. 2 or more times

# **SECTION** 7: **BELIEFS ABOUT PREGNANCY** (Other Variables)

These questions are about your beliefs about pregnancy.

- 7.1. How old do you think a woman should be when she has her first child?
  - a. YEARS OLD
  - b. I don't know.
- 7.2. How old do you think a man should be when he has his first child?
  - a. YEARS OLD
  - b. I don't know.
- 7.3. If you or your partner/boyfriend/girlfriend had a child in the next year, please tell us how <u>having a child</u> would affect you. (Even if you don't have a partner right now, tell us what you think you would do if this happened.)
  - a. It would interfere with my relationship with my partner.
    - i. Disagree
    - ii. Neither agree nor disagree
    - iii. Agree

- b. It would take away my freedom.
  - i. Disagree
  - ii. Neither agree nor disagree
  - iii. Agree
- c. It would interfere with my plans.
  - i. Disagree
  - ii. Neither agree nor disagree
  - iii. Agree
- d. It would be a real problem.
  - i. Disagree
  - ii. Neither agree nor disagree
  - iii. Agree
- e. It would fit in with my plans.
  - i. Disagree
  - ii. Neither agree nor disagree
  - iii. Agree
- f. My family would be upset or disappointed.
  - i. Disagree
  - ii. Neither agree nor disagree
  - iii. Agree
- g. My family would kick me out.
  - i. Disagree
  - ii. Neither agree nor disagree
  - iii. Agree
- h. It would give my life direction.
  - i. Disagree
  - ii. Neither agree nor disagree
  - iii. Agree
- i. It would make it difficult to get or keep a job.
  - i. Disagree
  - ii. Neither agree nor disagree
  - iii. Agree
- j. I would consider it a great gift.
  - i. Disagree
  - ii. Neither agree nor disagree
  - iii. Agree
- k. It would encourage me to keep my job or look for a better job.
  - i. Disagree
  - ii. Neither agree nor disagree
  - iii. Agree
- I. My family would support me.
  - i. Disagree
  - ii. Neither agree nor disagree
  - iii. Agree
- m. It would make it difficult to stay in school.

- i. Disagree
- ii. Neither agree nor disagree
- iii. Agree
- 7.4. If you or your partner got pregnant within the next year or are currently expecting a child, how likely do you think it is that you would do any of the following things? (Even if you don't have a partner right now, tell us what you think you would do if this happened.)

#### I WOULD ...

- a. Raise the baby.
  - i. Not at all likely
  - ii. Not very likely
  - iii. Somewhat likely
  - iv. Very likely
- b. Get married or stay married.
  - i. Not at all likely
  - ii. Not very likely
  - iii. Somewhat likely
  - iv. Very likely
- c. Put the baby up for adoption.
  - i. Not at all likely
  - ii. Not very likely
  - iii. Somewhat likely
  - iv. Very likely
- d. Give the child to a relative to raise.
  - i. Not at all likely
  - ii. Not very likely
  - iii. Somewhat likely
  - iv. Very likely

# SECTION 8: BELIEFS ABOUT BIRTH CONTROL METHODS, STIS, & HCV (Other Variables)

These next questions are about your beliefs about birth control and sexually transmitted diseases.

- 8.1 I believe that ...
  - a. Used correctly, most birth control methods will lower the chances a woman will get pregnant.
    - i. Disagree
    - ii. Neither Disagree nor Agree
    - iii. Agree
  - b. Talking about birth control methods will make your partner uncomfortable.
    - i. Disagree
    - ii. Neither Disagree nor Agree
    - iii. Agree
  - c. Using some birth control methods can be dangerous to a woman's health.
    - i. Disagree
    - ii. Neither Disagree nor Agree
    - iii. Agree
  - d. Talking about birth control methods with your partner will bring the two of you a lot closer.

- i. Disagree
- ii. Neither Disagree nor Agree
- iii. Agree
- e. It is hard for Indian women to accept using birth control methods because at times in the past the federal government forced it on them.
  - i. Disagree
  - ii. Neither Disagree nor Agree
  - iii. Agree
- f. Some birth control methods are too difficult to use correctly.
  - i. Disagree
  - ii. Neither Disagree nor Agree
  - iii. Agree
- g. Most of my friends and same-age relatives who have sexual intercourse use some type of birth control method.
  - i. Disagree
  - ii. Neither Disagree nor Agree
  - iii. Agree
- h. My friends and same-age relatives encourage me to use some type of birth control method every time I have sexual intercourse.
  - i. Disagree
  - ii. Neither Disagree nor Agree
  - iii. Agree
- 8.2. I believe that ...
  - a. My parents and most of my older relatives have talked with me about abstinence (not having sexual intercourse) as a method of birth control.
    - i. Disagree
    - ii. Neither Disagree nor Agree
    - iii. Agree
  - b. My parents and most of my older relatives have talked with me about the importance of using some type of birth control method.
    - i. Disagree
    - ii. Neither Disagree nor Agree
    - iii. Agree
  - c. I will insist on using a condom with a new sexual partner, even if my partner doesn't want to.
    - i. Disagree
    - ii. Neither Disagree nor Agree
    - iii. Agree
  - d. If I were going to have sex in the next year, I would use condoms.
    - i. Disagree
    - ii. Neither Disagree nor Agree
    - iii. Agree
  - e. I would avoid using condoms if at all possible.
    - i. Disagree
    - ii. Neither Disagree nor Agree
    - iii. Agree

- f. Using condoms makes sex feel unnatural.
  i. Disagree
  ii. Neither Disagree nor Agree
  iii. Agree
- g. You feel closer to your partner when you don't use condoms.
  - i. Disagree
  - ii. Neither Disagree nor Agree
  - iii. Agree
- h. If I decided to have sexual intercourse with someone, I'm quite certain I could get my partner to agree to use condoms.
  - i. Disagree
  - ii. Neither Disagree nor Agree
  - iii. Agree
- i. If my partner wanted to use a condom, we could use one correctly.
  - i. Disagree
  - ii. Neither Disagree nor Agree
  - iii. Agree
- j. I would never talk to a sex partner about using condoms.
  - i. Disagree
  - ii. Neither Disagree nor Agree
  - iii. Agree
- 8.3 The next few questions are about Hepatitis C (HCV). Answer True or False.

| a. HCV has no long-term effects on your healthTrue | False |
|-----------------------------------------------------------------|-------|
| b. It is possible to be vaccinated against HCVTrue | False |
| c. People who have injected drugs are not at risk for HCVTrue | False |
| d. HCV can be transmitted by tattooing and body piercingTrue | False |
| e. All people who have HCV can be curedTrue | False |
| f. HCV can be transmitted by sharing razors or toothbrushesTrue | False |
| g. A person can get HCV by sharing a needle and syringe | |
| with someone when injecting drugsTrue | False |
| h. A woman can get HCV through having sex with a manTrue | False |
| i. A person can get HCV from mosquitosTrue | False |
| j. Someone who looks very healthy can pass on HCVTrue | False |

# **SECTION 9: CONTRACEPTIVE & CONDOM USE SELF-EFFICACY** (Other variables)

We are now going to ask you some questions about what is important to you when selecting a birth control method to use when you have sex.

- 9.1 Indicate how important or unimportant these things about birth control are to you when selecting a birth control method to use to prevent pregnancy. Use this scale for your answers:
  - 1. Not important
  - 2. Slightly important
  - 3. Moderately important
  - 4. Very important
  - 5. Extremely important
  - a. Does not require me to touch my partners genitals
    - 1 2 3 4 5

| | b. Is no | | y to us | е. | |
|---|---|---|---|---|---|
| | 1 | 2 | 3 | 4 | 5 |
| | c. Does | | | | ed or stored. |
| | 1 | 2 | 3 | 4 | 5 |
| | | | | | eing a health care provider or getting a prescription |
| | 1 | 2 | 3 | 4 | 5 |
| | | | | | knowing about it. |
| | 1 | 2 | 3 | 4 | 5 |
| | | | | | en I have sex. |
| | 1 | 2 | 3 | 4 | 5 |
| | | ices yo | | | getting HIV. |
| | 1 | 2 | 3 | 4 | 5 |
| | h. Redu<br>1 | ices yo | | nces of<br>4 | getting an STD other than HIV. 5 |
| | i. Does | not ca | use sid<br>3 | e effect<br>4 | s like bleeding, cramps, weight gain, or changes in mood in [NAME]. 5 |
| | Does<br>1 | not ca | use pai<br>3 | n or irrit | tation.<br>5 |
| | اد ۱۸/:۱۱ س | ant dan | | م امینید | Negative for you or INAME1 |
| | 1 1 | 2 | 3 | 4 | oleasure for you or [NAME].<br>5 |
| | l le offe | activo i | n nrovo | nting pr | ognanov |
| | 1. 15 6116 | 2 | 3 | 4 | egnancy.<br>5 |
| | m. It is | inavna | neiva | | |
| | 1 | 2 | 3 | 4 | 5 |
| | n. It is e | easy to | use | | |
| | 1 | 2 | 3 | 4 | 5 |
| | o. It is a | a metho | od vou | can con | ntrol. |
| | 1 | 2 | 3 | 4 | 5 |
| | p. It is a | a metho | od your | partnei | r likes. |
| | 1 | 2 | 3 | 4 | 5 |
| 9.2 Ne | xt we are | e going | j to ask | some o | questions about how confident you are using a condom. Use this scale |
| | ır answe | | - | | |

for

j.

1 Not at all confident

2 Slightly confident
3 Moderately confident
4 Very confident
5 Extremely confident

| a. | | | | e you tha<br>ect you?<br>4 | t you could suggest using a condom even if you were afraid that your 5 |
|---|---|---|---|---|---|
| b. | | | | e you tha<br>condom<br>4 | t you could suggest using a condom even if you were unsure of how your s? |
| C. | | | | | t you could suggest using a condom even if you were afraid that your ou have had sex with another person before? |
| d. | | | | | it you could suggest using a condom even if you were afraid that your<br>ave an STD?<br>5 |
| e. | How<br>1 | confid<br>2 | lent do<br>3 | you feel<br>4 | in your ability to discuss using condoms with your partner? |
| f. | How<br>1 | confide<br>2 | ent do<br>3 | you feel<br>4 | in your ability to use a condom correctly? 5 |
| g. | | | | you feel | in your ability to put a condom on without breaking the sexual mood with |
| | your<br>1 | partne<br>2 | 3 | 4 | 5 |
| h. | How<br>1 | confid<br>2 | lent do | you feel<br>4 | in your ability to buy condoms without feeling embarrassed? |
| i. I | How 1 | confide<br>2 | ent are | you that | you could remember to carry a condom with you in case you need one? |
| j. l | How<br>1 | confide<br>2 | ent do<br>3 | you feel<br>4 | in your ability to use a condom with your partner even after drinking? |
| k. | How<br>1 | confid<br>2 | ent do<br>3 | you feel<br>4 | in your ability to use a condom with your partner even if you are high? |
| | How<br>excite | | ent do | you feel | in your ability to use a condom with your partner even if you are sexually |
| , | 1 | 2 | 3 | 4 | 5 |
| | G | ood jo | b! Yo | u are do | ing great so far! Please continue answering the questions. |
| | | | | | ow sure you are that you could say NO to sex, alcohol, drugs, etceven if nese things before. (Choose one answer for each question) |
| a. | a fev | w days<br>i. I De<br>ii. I Ca<br>iii. I Do<br>iv. I Ca | or les<br>finitely<br>in Say<br>on't Kn<br>an't Sa | s?<br>Can Say<br>No<br>low | |
| | | | | Answer | |

- b. How sure are you that you would be able to say NO to having sex with someone you want to date again?
  - i. I Definitely Can Say No
  - ii. I Can Say No
  - iii. I Don't Know
  - iv. I Can't Say No
  - v. I Definitely Can't Say No
  - vi. Refuse to Answer
- c. How sure are you that you would be able to say NO to having sex with someone who you want to fall in love with you?
  - i. I Definitely Can Say No
  - ii. I Can Say No
  - iii. I Don't Know
  - iv. I Can't Say No
  - v. I Definitely Can't Say No
  - vi. Refuse to Answer
- d. How sure are you that you would be able to say NO to having sex with someone who is pressuring you to have sex?
  - i. I Definitely Can Say No
  - ii. I Can Say No
  - iii. I Don't Know
  - iv. I Can't Say No
  - v. I Definitely Can't Say No
  - vi. Refuse to Answer
- e. How sure are you that you would be able to say NO to having sex with someone after one or both of you have been drinking alcohol, smoking pot, and/or using drugs, etc.?
  - i. I Definitely Can Say No
  - ii. I Can Say No
  - iii. I Don't Know
  - iv. I Can't Say No
  - v. I Definitely Can't Say No
  - vi. Refuse to Answer
- f. How sure are you that you would be able to say NO to having sex with someone who refuses to wear a condom?
  - i. I Definitely Can Say No
  - ii. I Can Say No
  - iii. I Don't Know
  - iv. I Can't Say No
  - v. I Definitely Can't Say No
  - vi. Refuse to Answer
- g. How sure are you that you would be able to say NO to having sex with someone who you have had sex with before?
  - i. I Definitely Can Say No
  - ii. I Can Say No
  - iii. I Don't Know
  - iv. I Can't Say No
  - v. I Definitely Can't Say No
  - vi. Refuse to Answer

# **SECTION 10: HEALTHY RELATIONSHIPS CHARACTERISTICS** (other variables)

Think about a current close relationship (other than with a family member)-it could be a romantic relationship, a close friend, or another. (If you don't have a relationship like that right now, think about one you had in the past, or think about a relationship that you would like to have in the future.)

| 10.1 Are the following signs of a healthy relationship? (Choose one a. | nswer for each question) |
|---|---|

| 10.1 Are the foll | owing signs of a healthy relationship? (Choose one answer for each question) |
|---|---|
| i.<br>ii. | vartner acts jealous or possessive. Yes . No i. Don't Know |
| | v. Refuse to Answer |
| i.<br>ii.<br>iii | vartner criticizes or puts the other one down. Yes . No i. Don't Know v. Refuse to Answer |
| | f you threatens to hurt themselves or the other person if the relationship ever ends. |
| i.<br>ii.<br>iii | Yes . No i. Don't Know v. Refuse to Answer |
| i.<br>ii.<br>iii | nd your partner feel free to ask honestly for what you want.<br>Yes<br>. No<br>i. Don't Know<br>v. Refuse to Answer |
| i.<br>ii.<br>iii | partner tries to change or control you (what you do and where you go).<br>Yes<br>. No<br>i. Don't Know<br>v. Refuse to Answer |
| i.<br>ii<br>iii | nd your partner are both comfortable with how physical the relationship is (or isn't). Yes No i. Don't Know V. Refuse to Answer |
| i.<br>ii.<br>iii | ring out the best qualities in each other.<br>Yes<br>. No<br>i. Don't Know<br>v. Refuse to Answer |
| h. You b | oth feel close to each other (not just physically) and are willing to trust each other with personal |

stuff.

- i. Yes
- ii. No
- iii. Don't Know
- iv. Refuse to Answer
- i. You make decisions jointly, with input from each partner.
  - i. Yes
  - ii. No
  - iii. Don't Know
  - iv. Refuse to Answer
- j. Your partner thinks there are some situations in which it is OK for him or her to hit you.
  - i. Yes
  - ii. No
  - iii. Don't Know
  - iv. Refuse to Answer

# **SECTION 11: LIFE EVENTS** (other variables)

11.1 Life Events are the next set of questions. For each life event, answer "No" if the event did *not* happen to you in the *past year*. or "Yes" if the life event *did* happen to you in the 12.§.§!\_y\_ear.

| | No | Yes |
|---|---|---|
| 1. Has a family member called you names, insulted you, or shamed you on a regular basis? | 0 | 1 |
| 2. Was your partner very jealous of you a lot of the time? | 0 | 211 |
| 3. Was your partner stingy toward you a lot of the time? | 0 | 1 |
| 4. Have you lived with someone who spent a lot of money gambling? | 0 | 1 |
| 5. Has a member of your partner's family called you names, insulted you, or shamed you on a regular basis? | 0 | 1 |
| 6. Have you wanted to work but could not find a job or lost a job? | 0 | 1. |
| 7. Has your partner wanted to work but could not find a job or lost a job? | 0 | 1 |
| Have you worried about getting kicked out of school, or what your parents would say about your school performance? | 0 | 1 |
| Have you worried about doing poorly in sports? | 0 | 1 |
| 10. Were you or a close family member threatened or hurt by gang violence? | .0 | 232 <b>1</b> 340 |
| 11. Have people gossiped or spread rumors about you? | 0 | 1 |
| 12. Has someone important to you attempted suicide and survived? | 0 | 1.1 |
| 13. Has someone important to you committed suicide? | 0 | 1 |
| 14. Have you had a serious argument with a friend or friends? | 0 | Q. <b>1</b> 37 |
| 15. Have you broken up with your partner? | 0 | 1 |
| 16. Have you gotten in a car wreck in which someone was hurt or killed? | 0 | 1 |
| 17. Has a relative taken over the care of your child (or children)? | 0 | 1 |
| 18. Have you lost custody of your child (or children)? | 0 | 35 <b>1</b> 37 |
| 19. Were you unable to find good child care for your child (or children)? | 0 | 1 |
| 20. Has someone important to you died from causes other than suicide? | 0 | 1 |
| 21. Have you or someone important to you had an alcohol or drug problem? | 0 | 1 |
| 22. Have you or someone important to you gone to an alcohol or drug treatment program? | 0.1 | 1 |
| 23. Have you or someone important to you "fallen off the wagon"? | 0 | 11 |
| 24. Have you or someone important to you had a serious health 71 or injury or was hospitalized (not including alcohol or drug problems or relatment)? | 0 | 1 |
You are almost done with the survey. These are the last questions.

- 11.1 Please mark which best describes how you felt during the past week.
  - a. I felt that I could not shake off the blues even with help from my family or friends.
    - i. None of the time (0 days)
    - ii. Rarely or a little of the time (1-2 days)
    - iii. Some of the time (3-4 days)
    - iv. Most or all of the time (5-7 days)
  - b. I felt depressed.
    - i. None of the time (0 days)
    - ii. Rarely or a little of the time (1-2 days)
    - iii. Some of the time (3-4 days)
    - iv. Most or all of the time (5-7 days)
  - c. I thought my life had been a failure.
    - i. None of the time (0 days)
    - ii. Rarely or a little of the time (1-2 days)
    - iii. Some of the time (3-4 days)
    - iv. Most or all of the time (5-7 days)
  - d. I felt fearful.
    - i. None of the time (0 days)
    - ii. Rarely or a little of the time (1-2 days)
    - iii. Some of the time (3-4 days)
    - iv. Most or all of the time (5-7 days)
  - e. I felt lonely.
    - i. None of the time (0 days)
    - ii. Rarely or a little of the time (1-2 days)
    - iii. Some of the time (3-4 days)
    - iv. Most or all of the time (5-7 days)
  - f. I had crying spells.
    - i. None of the time (0 days)
    - ii. Rarely or a little of the time (1-2 days)
    - iii. Some of the time (3-4 days)
    - iv. Most or all of the time (5-7 days)
  - g. I felt sad.
    - i. None of the time (0 days)
    - ii. Rarely or a little of the time (1-2 days)
    - iii. Some of the time (3-4 days)
    - iv. Most or all of the time (5-7 days)
  - h. I felt crabby.
    - i. None of the time (0 days)
    - ii. Rarely or a little of the time (1-2 days)
    - iii. Some of the time (3-4 days)
    - iv. Most or all of the time (5-7 days)
  - i. I felt hopeless.
    - i. None of the time (0 days)
    - ii. Rarely or a little of the time (1-2 days)

- iii. Some of the time (3-4 days)
- iv. Most or all of the time (5-7 days)
- j. I felt like no one cared.
  - i. None of the time (0 days)
  - ii. Rarely or a little of the time (1-2 days)
  - iii. Some of the time (3-4 days)
  - iv. Most or all of the time (5-7 days)
- k. I felt discouraged.
  - i. None of the time (0 days)
  - ii. Rarely or a little of the time (1-2 days)
  - iii. Some of the time (3-4 days)
  - iv. Most or all of the time (5-7 days)
- 11.2. During the past week ....
  - a. Have you often worried that you have made a fool of yourself in front of other people?
    - i. No
    - ii. Yes
  - b. Have you often worried that you have made a mistake or done something the wrong way?
    - i. No
    - ii. Yes
  - c. Have you been almost always worried about something?
    - i. No
    - ii. Yes
  - d. Have you been very worried about whether other people like you?
    - i. No
    - ii. Yes
  - e. Have you often gotten worried or nervous?
    - i. No
    - ii. Yes

YOU ARE FINISHED WITH THE SURVEY! THANK YOU VERY MUCH FOR TAKING THE TIME TO COMPLETE THE SURVEY. PLEASE REMEMBER THAT NONE OF YOUR RESPONSES WILL BE ASSOCIATED WITH YOUR NAME. IF YOU HAVE ANY QUESTIONS ABOUT THIS SURVEY PLEASE ASK US.

# Nen OnkUmbi/EdaHiYedo {"We Are Here Now") Informed Consent to Participate in Human Subjects Research with Montana State University in Partnership with Fort Peck Community College

#### What is this project about?

We Are Here Now is an intervention project with Fort Peck Community College and Montana State University. Nen OnkUmbi/EdaHiYedo {"We are Here Now," or NIE) derives from the Assiniboine (Nen OnkUmbt) and Sioux (EdaHiYedo) names for their traditional coming-of-age ceremonies. The purpose of this program is to teach youth at Fort Peck important things they need to know about sex so that they can stay healthy and not get a sexually transmitted disease, HIV, or Hepatitis C, and so that they can make healthy decisions about having children, getting pregnant, or getting someone pregnant. We Are Here Now also includes tribal elders and leaders teaching Assiniboine and Sioux youth about their culture and traditional beliefs and practices about what it means to be a young Native person who will soon be an adult. In addition to working with youth, We Are Here Now also is offering education to parents/legal guardians about how to speak with their children about sensitive topics related to sex.

#### Why me?

You and your child have been invited to participate in *We Are Here Now* and to help gather information about the program and its effects. Your participation in this intervention is entirely voluntary. You can choose not to participate at any time. You and your child may withdraw from the intervention at any time without negative consequences. Your participation in *We Are Here Now* is your choice.

#### What happens to me if I decide to participate?

If you agree to participate in *We Are Here Now*, you will be with other guardians or parents of young people who are participating in *We Are Here Now*, and you will learn about how to talk with your child about sex. *We Are Here Now* is a project that educates youth and their guardians/parents about sexual and reproductive health. As a participant in *We Are Here Now*, you will be talking with other guardians/parents about healthy sexual behaviors and about how to talk with your children about sex. You will be asked to complete a survey specifically for guardians/parents about how you talk to your child about sex and what kinds of things about sex you speak with them about. You will receive an incentive of \$20 for this first survey, and then \$10 each time you attend the four *Native Voices* sessions (at 2 of these sessions you will again fill out the survey). Finally, you will receive a \$25 incentive for completing the final survey after the end of the program.

#### What are the risks?

Some of the questions may make you feel a bit uncomfortable. For example, we will ask you about what kinds of sexual topics you talk about with your child.

#### What are the benefits?

Through this program you will learn about ways to speak effectively with your child about sex and topics related to sexual health. The information gathered in this survey will help the intervention's research team and members of the Fort Peck community to understand what kind of impact your participation in *We Are Here Now* is having on your decisions to talk with your child about sensitive topics related to sex.

#### Who gets access to information from this interview?

All responses on this survey will be anonymous. Only one person, Paula FireMoon, will know that you participated, because she will keep this signed consent form in a locked file cabinet in her locked office. Neither she nor the rest of the research team, nor the community advisory board, will know what your individual responses to the survey are. The research team will have access to the anonymous data collected for this project. The *We Are Here Now* community advisory board will also have access to the anonymous data collected for this intervention.

## <u>How am I informed about the results of the project. and when will they</u> be released and presented to someone else?

We will publish the intervention results and make presentations on the results from *We Are Here Now.* Your identity will never appear in a publication or in print or be discussed at a presentation. In addition, you will have the opportunity to learn about the intervention results by contacting members of the research team, by attending community meetings where we share the results of the project, and through local (Fort Peck Reservation) media.

#### Who is involved in We Are Here Now?

If you have any questions regarding this survey please contact:

#### Paula FireMoon, Fort Peck Community College

Email: PFiremoon@fpcc,edu; Phone: 406.768.6300

#### Elizabeth Rink, Montana State University

Email: elizabeth.rink@montana.edu; Phone: 406.994.3833

#### **CONSENT STATEMENT**

| Parent/Legal Guardian for Minor: I hav inconvenience, and risks associated with | e read the above and understand the discomfort, this survey. |
|---|---|
| I,<br>Name of Parent/Guardian | , do agree to participate in this survey. |
| Parent/Guardian Signature: | Date: |
| SuNey Administrator Signature: | Date |

### "NenUnkUmbi/EdaHiYedo" (We Are Here Now)

#### **PARENT SURVEY**

We want to learn more about how you discuss sex with your child and what kinds of topics you discuss. We will be asking you a series of questions about how you talk to your child about sex and how you experience this communication. We thank you for your time.

#### **SECTION 1: DEMOGRAPHICS**

| We would like to start by asking you some questions abou | t yoursel | f. | |
|---|---|---|---|
| 1. How old are you? | | | |
| 2. What is the highest grade you have completed? | | | |
| 3. What is your occupation? | | | |
| 4. What is your martial status? Please circle one. | | | |
| a. married b. single c. living with a boyfrie | end/girlfri | end | |
| SECTION 2: COMMUN/CATION WITH CHILD | | | |
| Next we are going to ask some questions about how you for child about sex and what kinds of things about sex you specified. | | - | |
| How would you rate your ability to communicate with you a. Difficult b. Somewhat Difficult c. Neither Difficult or Easy d. Somewhat Easy e. Easy | ur child i | n gen | ieral? |
| 2. How would you rate your ability to communicate with you a. Difficult b. Somewhat Difficult c. Neither Difficult or Easy d. Somewhat Easy e. Easy | ur child a | about | sex? |
| I would like to talk more often with my child about sex at a. Yes b. No | nd sexua | lity. | |
| 4. Have you ever talked with your child about each of the f | ollowing | topics | 5? |
| | YES | NO | I DON'T KNOW |
| a. What qualities are important in choosinQ close friends | | | |
| <b>b.</b> What qualities to look for in a boyfriend/girlfriend/life partner | | | |

| c. How to ask someone out on a date | 1 | Ì |
|---------------------------------------------------------------------|---|---|
| d. How boys' bodies change physically as they grow up | | |
| e. How qirls' bodies change physically as they grow up | | |
| f. How women get pregnant and have babies | | |
| g. Symptoms of sexually transmitted infections (STIs) | | |
| h. Reasons why people like to have sex | | |
| i. How well birth control can prevent pregnancy | | |
| j, How to choose a method of birth control | | |
| k. How to say no if someone wants to have sex and you | | |
| don't want to | | |
| I. How well condoms can prevent sexually transmitted | | |
| infections (STIs) | | |
| m. Menstruation (having menstrual periods) | | |
| <b>n.</b> The importance of not pressuring other people to have | | |
| sex | | |
| How your child will make decisions about whether or not to have sex | | |
| p. Consequences of getting pregnant/getting someone | | |
| pregnant | | |
| q. How to use a condom | | |
| r. Reasons why your child should not have sex at this time | | |
| s. Masturbation | | |
| t. What it feels like to have sex | | |
| u. Homosexuality/people being gay | | |
| v. Wet dreams [measured for parents of boys only] | | |
| w. What to do if a partner doesn't want to use a condom | | |
| x. How people can prevent getting sexually transmitted | | |
| infections (STIs) | | |
| V. How your child will know if he/she is in love | | |

<u>CLOSING STATEMENT</u>
Thank you so much! That is all of our questions. As I said in the beginning, everything you told me today will remain private. Your name will not be on any information.

#### Nen OnkUmbi/EdaHiYedo (We Are Here Now)

## Systems-Level Intervention Component BARRIERS & FACILITATORS DISCUSSION GUIDE

We Are Here Now is a 5-year intervention project with Fort Peck Community College and Montana State University. Nen OnkUmbi/EdaHiYedo ("We are Here Now," or NIE) derives from the Assiniboine (NenUnkUmbi) and Sioux (EdaHiYedo) names for their traditional coming-of-age ceremonies. The overall goal of We Are Here Now is to reduce STIs, HIV, HCV, and teen pregnancy among American Indian (Al) youth living on the Fort Peck Reservation. There are four levels of We Are Here Now. a school-based curriculum called Native Stand; a parent curriculum called Native Voices; a cultural mentoring program with the Fort Peck Tribes' Language and Culture Department; and a systems-level component that involves increasing access to sexual and reproductive health (SRH) services for Al youth here at Fort Peck. As part of the systems-level component of We Are Here Now, we are working with the members of the Epi Team to identify and track the barriers and facilitators to provision of SRH services for Al youth here at Fort Peck. We would like to discuss with you what is and is not being provided to Al youth in your agencies and discuss possible solutions and steps to enhancing what and how SRH services are provided to Al youth. Our discussion today is based on the 8 service domains relative to improving SRH services of adolescents as outlined by the Centers for Disease Control and Prevention's (CDC) Contraceptive and Reproductive Health Services for Teens: Evidence-based Clinical Best Practices. We will use the results from our annual discussions to develop a monitoring plan tracking log to track our efforts to increase access to and utilization of SRH services for Al youth over the 5 years of We Are Here Now. As we have discussed, we will audio-tape the annual discussions, so please try to talk one person at a time. We would like everyone to be able to express their viewpoints without being interrupted. Do you have any questions for me before we begin the discussion? [Answer questions, if any] OK, let's get started.

#### **SERVICE DOMAIN #1: CONTRACEPTIVE ACCESS**

Discuss the extent to which your agency <u>does or does not</u> provide the services listed below. Please address what the barriers are to providing these services and/or what the factors are that facilitate the provision of these services.

- Offers same-day appointments
- Offers after-school-hours appointments
- Offers appointments during the weekend
- Takes/updates sexual health history at every visit
- Offers a wide-range of contraception (via prescription and/or dispensed onsite)
- Offers hormonal contraception or IUD at every visit to the clinical provider regardless
  of reason for visit (e.g., urgent, preventive, school health, sports physical,
  pregnancy testing, emergency contraception, sexually transmitted disease [STD]
  testing, HIV testing) to ensure that there are no missed opportunities

 Prescribes hormonal contraception without prerequisite exams or STI testing (i.e., without first requiring any of the following: Pap smear, pelvic examination, breast examination, or STD testing)

## SERVICE DOMAIN #2: QUICK START PROVISION OF HORMONAL CONTRACEPTION/IUD

Discuss the extent to which your agency <u>does or does not</u> provide the services listed below. Please address what the barriers are to providing these services and/or what the factors are that facilitate the provision of these services.

- Initiates hormonal contraception using the Quick Start method<sup>1</sup>
- Initiates hormonal contraception after the client has had a negative pregnancy test using Quick Start method
- Initiates hormonal contraception using the Quick Start method when an adolescent client is provided with emergency contraception where a pregnancy test is negative
- · Offers Quick Start insertion of IUD

#### SERVICE DOMAIN #3: EMERGENCY CONTRACEPTION

Discuss the extent to which your agency <u>does or does not</u> provide the services listed below. Please address what the barriers are to providing these services and/or what the factors are that facilitate the provision of these services.

- Ensures emergency contraception is available to females
- Provides emergency contraception to females for future use
- Provides emergency contraception to males for future use

#### **SERVICE DOMAIN #4: CERVICAL CANCER SCREENING**

Discuss the extent to which your agency <u>does or does not</u> provide the service listed below. Please address what the barriers are to providing these services and/or what the factors are that facilitate the provision of these services.

 Adheres to current cervical cancer screening (Pap Smear) guidelines (i.e., initiate pap screening at age 21)

#### SERY\_ICE DOMAI\_t-.1 #5: STI/HIV TESTING AND TREATMENT

Discuss the extent to which your agency <u>does or does not</u> provide the services listed below. Please address what the barriers are to providing these services and/or what the factors are that facilitate the provision of these services.

 Provides Chlamydia screening at least annually, or based on diagnostic criteria, consistent with USPSTF and CDC recommendations

- Offers Chlamydia screening for females using a urine or vaginal swab specimen
- Offers Chlamydia screening for males using a urine specimen
- · Offers Gonorrhea screening for both females and males
- Offers HIV rapid testing for females and males as per CDC recommendations
- Offers expedited, patient-delivered partner therapy as an option for the treatment of uncomplicated chlamydia! infection

Additional question for HCV testing: Discuss the extent to which your agency <u>does or does not</u> provide HCV testing and treatment. In your discussion, address what the barriers are to providing HCV testing and treatment and/or what the factors are that facilitate the provision of HCV testing and treatment.

#### SERVICE DOMAIN #6: COST, CONFIDENTIALITY, CONSENT

Discuss the extent to which your agency <u>does or does not</u> provide the services listed below. Please address what the barriers are to providing these services and/or what the factors are that facilitate the provision of these services.

- Provides low-cost or no-cost contraceptive and reproductive health care services
- Provides confidential contraceptive and reproductive health care to adolescents without need for parental or caregiver consent (in accordance with state policy)

#### SERVICE DOMAIN #7: HEALTH CENTER/AGENCY INFRASTRUCTURE

Discuss the extent to which your agency <u>does or does not</u> provide the services listed below. Please address what the barriers are to providing these services and/or what the factors are that facilitate the provision of these services.

- Participates in the federal 3408 drug discount purchasing program
- Uses electronic medical records (e.g., eClinical Works, Centricity, Epic, NextGen)
- Has systems in place to facilitate billing third party payers for contraceptive and reproductive health care services provided

#### SERVICE DOMAIN #8: HEALTH CENTER/AGENCY ENVIRONMENT

Discuss the extent to which your agency <u>does or does not</u> provide the services listed below. Please address what the barriers are to providing these services and/or what the factors are that facilitate the provision of these services.

- Has a counseling area that provides both visual and auditory privacy
- Has an examination room that provides visual and auditory privacy
- Has teen-focused magazines in the waiting room or examination areas
- Displays information on issues related to adolescent sexual and reproductive health

(e.g., confidentiality, cost, what services are available to adolescents)

• Has brief evidence-based or evidence-informed video or other interventions designed for adolescents

**THANK YOU!** That is it for our discussion today. Are there any questions? Or does anyone have anything more you would like to add?

#### NenUnkUmbi/EdaHiYedo (We are Here Now): COORDINATION & IMPLEMENTING MONITORING PLAN TRACKING LOG

| AGENCY NAME: | AGENCY CONTACT NAME: |
|-------------------------------|----------------------|
| AGENCY CONTACT INFORMATION: | |
| DATE TRACKING LOG FILLED OUT: | |

#### **OVERVIEW AND INSTRUCTIONS**

The purpose of this assessment is to help your health center identify current services, as well as opportunities for improving the quality of services for adolescent patients. Information collected through this assessment will be used to trach health center progress in improving adolescent access to contraceptive and reproductive health services within Fort Peck.

This assessment should be completed every 3 months. Please meet with members of your multidisciplinary health care team to complete this assessment. This team-based approach to completing the assessment is important to ensure the information collected is accurate, and also to ensure that relevant team members are aware of the data being collected, and able to work together to identify opportunities for improving the quality of services offered to adolescents.

#### SERVICE DOMAIt-,1 #1: CONTRA\_CEPTIVE ACC\_ESS

| Evidence Based Clinical Practice | <br>vice Provid<br>eck only on | Barriers/Facilitators Description | Action Steps<br>Required | Completion<br>Timeline | Responsible<br>Party |
|---|---|---|---|---|---|
| Offers same-day appointments | | | | | |
| Offers after-school hours appointments. | | | | | |
| Offers weekend appointments. | | | | | |
| Takes/updates sexual health history at every visit | | | | | |
| Offers a wide-range of contraception | | | | | |
| Offers hormonal contraception or IUD at every visit to the clinical provider regardless of reason for visit | | | | | |
| Prescribes hormonal contraception without prerequisite exams or STI testing | | | | | |

#### SERVICE DOMAIN #2: qUJCK START PROVISION of HORMONAL CONTRACEPTION/IUO

| Evidence Based Clinical Practice | (ch | vice Provid<br>eck only o | n ) | Barriers/Facilitators Description | Action Steps<br>Required | Completion<br>Timeline | Responsible<br>Party |
|---|---|---|---|---|---|---|---|
| Initiates hormonal contraception using the Quick Start method | Alwavs | Sometimes | Never | | | | |
| Initiates hormonal contraception after the client has had negative pregnancy test using Quick Start method | | | | | | | |
| Initiates hormonal contraception using the Quick Start method when an adolescent client is provided with emergency contraception where a pregnancy test in negative | | | | | | | |
| Offers Quick Start Insertion of IUD | | | | | | | |

#### SERVICE DOMAIN #3: EMERGENCY CONTRACEPTION

| Evidence Based Clinical Practice | Service Provided (check only one) | | | Barriers/Facilitators Description | Action Steps<br>Required | Completion<br>Timeline | Responsible<br>Party |
|---|---|---|---|---|---|---|---|
| | Alwavs | Sometimes | Never | | | | - |
| Ensures emergency contraception is available | | | | | | | |
| Provides emergency contraception to females for future use | | | | | | | |
| Provides emergency contraception to males for future use | | | | | | | |

### SERVICE DOMAIN #4: CERVICAJ.. CANCER SCREE; ING

| Evidence Based Clinical Practice | Service Provided (check only one\ Atways Sometimes Never | | | Barriers/Facilitators Description | Action Steps<br>Required | Completion<br>Timeline | Responsible<br>Party |
|---|---|---|---|---|---|---|---|
| Adheres to current cervical cancer screening (Pap Smear) guidelines (i.e., intiate pap screening at age 21) | Always | Gomeanies | Nevel | | | | |

### SERVICE DOMAIN #5: <u>STI/I-IIV/HCV</u> TESTING AND <u>TREATM\_ENT</u>

| Evidence Based Clinical Practice | <br>rvice Provi<br>neck only o | Barriers/Facilitators Description | Action Steps<br>Required | Completion<br>Timeline | Responsible<br>Party |
|---|---|---|---|---|---|
| Provides Chlamydia screening at least annually, or based on diagnostic criteria, consistent with USPSTF and CDC recommendations | | | | | |
| Offers Chlamydia screening for females using a urine or vaginal swab specimen | | | | | |
| Offers Chlamydia screening for males using a urine specimen | | | | | |
| Offers Gonorrhea screening for both females and males | | | | | |
| Offers HIV rapid testing for females and males as per CDC recommendations | | | | | |
| Offers expedited, patient-delivered partner therapy as an option for the treatment of uncomplicated chlamydia! infection | | | | | |
| Offers HCV testing and treatment | | | | | |

### SERVICE DOMAIN #6: COST. CONFIDENTIALITY, CONSENT

| Evidence Based Clinical Practice | Service Provided (check only one) Aways Sometimes Never | | | Barriers/Facilitators Description | Action Steps<br>Required | Completion<br>Timeline | Responsible<br>Party |
|---|---|---|---|---|---|---|---|
| Provides low-cost or no-cost contraceptive and reproductive health care services | , and to | Sundamo | 110101 | | | | |
| Provides confidential contraceptive and reproductive health care to adolescents without need for parental or caregiver consent (in accordance with state policy) | | | | | | | |

### SERVICE DOMAIN #7: HEALTHCARE/AG\_f:NCY INFRASTRUCTURE

| Evidence Based Clinical Practice | Service Provided (check only one\ | | ne\ | Barriers/Facilitators Description | Action Steps<br>Required | Completion<br>Timeline | Responsible<br>Party |
|---|---|---|---|---|---|---|---|
| Participates in the federal 340B drug discount purchasing program | Alwavs | Sometimes | Never | | | | |
| Uses electronic medical records | | | | | | | |
| Has systems in place to facilitate billing third party payers for contraceptive and reproductive health care services provided | | | | | | | |

### SERVICE DOMAIN #8:\_HEAL<u>TI-LCENTER/AGENCY</u> ENVIRONMENT

| Evidence Based Clinical Practice | rvice Provineck only o | Barriers/Facilitators Description | Action Steps<br>Required | Completion<br>Timeline | Responsible<br>Party |
|---|---|---|---|---|---|
| Has a counseling area that provides both visual and auditory privacy | | | | | |
| Has an examination room that provides visual and auditory privacy | | | | | |
| Has teen-focused magazines in the waiting room or examination areas | | | | | |
| Displays information on issues related to adolescent sexual and reproductive health (e.g., confidentiality, cost, what services area available to adolescents) | | | | | |
| Has brief evidence-based or evidence-<br>informed video or other interventions<br>designed for adolescents | | | | | |

#### SERVICE DOMAN #SA: HEALTII CEI'IITER STAFF TRAINING

Please indicate the number and percentage of <u>ALL health center staff</u> (e.g., all clinical and non-clinical staff that have direct contact with adolescent clients) that have received training in the following areas in the **past two years**.

| In the past two years, staff received trainina on | Number of staff | % of staff | Barriers/Facilitators Description | Action Steps<br>Reauired | Completion<br>Timeline | Responsible<br>Partv |
|---|---|---|---|---|---|---|
| Stages of adolescent development | | | | | | |
| State-specific minors' rights to consent and confidentiality laws or provisions | | | | | | |
| Cultural competency, including relevant | | | | | | |
| Native beliefs and cultural traditions | | | | | | |
| Continuous quality improvement (CQI) | | | | | | |
| Youth-friendly services | | | | | | |
| Strategies for serving non-English speaking populations (inc interoreter) | | | | | | |
| Addressing the needs of lesbian, gay, bisexual, transgender, and queer (LGBTQ) youth | | | | | | |

Please indicate the number and percentage of <u>clinical staff</u> (e.g., MDs, advance practice clinicians, nurse-extenders) that have been trained in the following areas in the past two years.

| In the past two years, clinical staff received trainina on | Number of staff | % of staff | Barriers/Facilitators Description | Action Steps<br>Reauired | Completion<br>Timeline | Responsible<br>Party |
|---|---|---|---|---|---|---|
| Contraceptive Services for Adolescents | | | | | | |
| Use of the Quick Start method for initiation of hormonal contraception | | | | | | |
| Use of Quick Start method for initiation of IUD | | | | | | |
| IUDs for Adolescents | | | | | | |
| Hormonal Implants | | | | | | |
| Emergency Contraception | | | | | | |
| Pap Smear Guidelines | | | | | | |
| Breast exam guidelines | | | | | | |
| Conducting a sexual health assessment/history for adolescents | | | | | | |
| STI testing for adolescents | | | | | | |
| HIV testing for adolescents | | | | | | |
| Male sexual and reproductive health services | | | | | | |
| Continuous quality improvement (CQI) | | | | | | |
| Youth-friendly services | | | | | | |
| Cultural competency, including relevant Native beliefs and cultural traditions | | | | | | |

#### SERVICE DOMAN #9: ADOLESCENT PATIENT DEMOGRAPHICS

NOTE: The following data may be collected via billing records, EMRs, and other methods. We are open to suggestions for other data collection methods based on your familiarity with your health center partners and your ability to collect data from your partners. It is recommended that you collect these data every 3 months.

Please note that by "visits" we mean any visit where an adolescent is seen by a health care team member - not only visits designated as reproductive/sexual health visits.

Please note that by "adolescent visits where contraceptive, reproductive, or sexual health services are provided" we mean any health center visit where contraceptive, reproductive, or sexual health services are provided to the adolescent patient, regardless of the primary reason for the visit.

| For the <u>past 3 months</u> . | # adolescents seen (unduplicated) | #adolescent vis | eadolescent visits at which contracepuve<br>eproductive, or sexual health services are the<br>provided |
|---|---|---|---|
| FEMALE PATIENTS 12-14 years | | | |
| 15-18 years | | | THE TOTAL STATE OF THE STATE OF |
| 12-14 years<br>15-18 years | | | |

| For the past 3 months | # adolescents tested for HTV | # positive results | # negative resums |
|---|---|---|---|
| FEMALE PATIENTS | | | 12 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 |
| 12-14 years | | | |
| 15-18 years | | | |
| MALEPATIENTS | | | |
| 12-14 years | | | |
| 15-18 years | | | |

| For the past 3 months | # adolescents tested for chlamydia | # positive results | # negative results | 7.00 |
|---|---|---|---|---|
| FEMALE PATIENTS | | | | |
| 12-14 years | | | | |
| 15-18 years | | | | |
| MALE PATIENTS | | | | |
| 12-14 years | | | | |
| 15-18 years | | | | |

| For the past 3 months | # adolescents | tested for gonorrhea | # positive results | # negative results |
|---|---|---|---|---|
| FEMALE PATIENTS | | | | <u> </u> |
| 12-14 years | | | | |
| 15-18 years | | | | |
| MALE PATIENTS | | | | |
| 12-14 years | | | | |
| 15-18 years | | | | <br> |

Please complete the below table regarding the provision of hormonal contraception and IUD for adolescents in the J:!ast 3 months.

| 4 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | -276-≥ <b>4</b> ш | duplicated adolescents p | etivided | | |
|---|---|---|---|---|---|
| | The pill | Injectable : | NO A | Contraceptive implants (e.g., | Emergency contracentical |
| | 0.000 | contraception (e.g.,<br>Depo Provera) | | Nexplanon) | |
| FEMALE PATIENTS | | <u>uepo: turstaj</u> | | | terit in the second |
| 12-14 years | | | | | |
| 15-18 years | | | | | |

Filled out once per quarter after each Community Advisory Board meeting.

| Barriers or Facilitators to<br>Intervention implementation<br>discussed: | Type of contextual factors discussed (i.e. Social context, Environmental context, Political context, or Bureaucratic context): | Suggestions or solutions discussed: |
|---|---|---|

## NenUnkUmbi/EdaHiYedo (We are Here Now)

## Whole Team meeting form

| Date of Meeting | |
|------------------------------------------------|-------------|
| Date form filled out (today's date): | |
| Filled out once every other month beginning Fe | bruary 2019 |

| Barriers or Facilitators to<br>Intervention<br>implementation<br>discussed: | Type of contextual factors discussed (i.e. Social context, Environmental context, Political context, or Bureaucratic context): | Suggestions or solutions discussed: | Action and responsible party: | Adherence to Community- Based Participatory Research Principles? |
|---|---|---|---|---|

| NenUnkUmbi/EdaHiYedo (We are Here Now) |
|---------------------------------------------------------------------|
| Fidelity Reach Log and Field Notes: |
| Date form filled out (today's date): |
| Filled out each day any component of the Intervention is delivered. |

mod out oddin ddy diny ddinpondin o'i ard intervoliaen ioddin e

## **Intervention Delivery**

| Intervention Component Name (i.e. Native Stand, Native Voices, Cultural Mentoring, or Systems): | Date of<br>Intervention<br>delivery or<br>meeting: | Length of<br>time of<br>Intervention<br>delivery: | If Native Stand, Native<br>Voices, or Cultural<br>Mentoring, specific<br>modules delivered: | Barriers to Intervention delivery: | Facilitators to Intervention delivery: |
|---|---|---|---|---|---|

## **Field Notes:**

Below to be filled out by the School Coordinator after any component of the Intervention is delivered.

| Intervention Component Name (i.e. Native Stand, Native Voices, Cultural Mentoring, or Systems): | Environmental (weather, travel, etc.) barriers or facilitators to Intervention Delivery? | Social (basketball, mood of the group or general community etc.) barriers or facilitators to Intervention delivery? | Political or bureaucratic barriers or facilitators to Intervention delivery? | Suggestions or solutions? |
|---|---|---|---|---|

# MONTANA STATE UNIVERSITY

#### INSTITUTIONAL REVIEW BOARD

#### For the Protection of Human Subjects FWA 00000165

2155 Analysis Drive c/o Microbiology & Immunology Montana State University Bozeman, MT 59718 Telephone: 406-994-4706 FAX: 406-994-4303 E-mail: chervi@montana.edu Chair: Mark Quinn 406-994-4707 mquinn@montana.edu Administrator: Cheryl Johnson

Cheryl Johnson 406-994-4706 cherylj@montana.edu

## MEMORANDUM

TO:

Elizabeth Rink

FROM:

Mark Ouinn Wark June Cy

Chair, Institutional Review Board for the Protection of Human Subjects

DATE:

November 6, 2020

SUBJECT:

"Nen Ünk?umbi/Edahiyedo ("We Are Here Now") - a Multi-level, Multi-component

sexual and Reproductive Health Intervention for American Indian Youth - Pilot

Study" [ER020518]

Thank you for submitting the follow-up report on the above research project. Reapproval of this project for an additional year will be reflected on the agenda of the next Institutional Review Board meeting. In the meantime, work on the project may continue. At the end of this approval period you will receive another follow-up form which will be used to evaluate this proposal for renewal. If the project extends beyond five years, you will need to submit a new application. Please keep track of the number of subjects who participate in the study and of any unexpected or adverse consequences of the research. If there are any adverse consequences, please report them to the committee within 3 calendar days. If there are serious adverse consequences, please suspend the research until the situation has been reviewed by the Institutional Review Board.

Any changes in the human subjects' aspects of the research should be approved by the committee before they are implemented.

It is the investigator's responsibility to inform subjects about the risks and benefits of the research. Although the subject's signing of the consent form, documents this process, you, as the investigator should be sure that the subject understands it. Please remember that subjects should receive a copy of the consent form and that you should keep a signed copy for your records.

In one year, you will be sent a questionnaire asking for information about the progress of the research. The information that you provide will be used to determine whether the committee will give continuing approval for another year. After initial approval, if the research is still in progress beyond a 5-year period, a completely new application will be required.



#### Fort Peck Tribal Institutional Review Board For the Protection of Human Subjects

FWA00019355

hair: Robert McAnally 406-768-8377

bmcassin@gmail.com

Fort Peck Community College Box 398 Poplar, MT 59255 406-768-6300 Administrator: (Acting)

Paula FireMoon 406-768-6300 pfiremoon@fpcc.edu



## MEMORANDUM

TO:

Elizabeth Rink, PhD, MSW

FROM:

Robert McAnally, J.D. Shut J midway

Chairman, Institutional Review Board for the Protection of Human Subjects

DATE:

November 1, 2023

RE:

IRB Approval for the following: 1) Continued Data Analysis, 2) Continued Work with Community Advisory Board, 3) Design & Completion of "We Are Here Now" Tool Kit, 4) Implementation of Pilot Study that includes a Revised High School Survey, New Teacher Survey, and Revised Informed Consent Forms for Students and Parents,

and New Informed Consent Forms for Teachers.

The Institutional Review Board has reviewed the above referenced requests and have officially granted approval on November 1, 2023.

#### As a reminder:

Please keep track of the number of subjects who participate in the study and of any unexpected or adverse consequences of the research. If there are any adverse consequences, please report them to the committee as soon as possible. If there are serious adverse consequences, please suspend research until the situation has been reviewed by the Institutional Review Board.

It is the investigator's responsibility to inform subjects about the risks and benefits of the research. Although the subjects' signing of the consent form, documents this process, you, as the investigator should be sure that the subject understands it. Please remember that subjects should receive a copy of the consent form and that you should keep a signed copy for your records.

Any future changes in the human subjects' aspects of the research will need approval by the Institutional Review Board before implementation.

The Fort Peck IRB requests that when you have a manuscript, thesis, or presentation prepared for public consumption, that you provide a copy to the Fort Peck IRB for prior approval. The IRB needs an opportunity to review the document pre-publication and may make recommendations to ensure the document appropriately respects the members of the Fort Peck Assiniboine and Sioux Tribes.